CLINICAL TRIAL: NCT02531633
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Sirukumab in the Treatment of Patients With Giant Cell Arteritis
Brief Title: Efficacy and Safety Study of Sirukumab in Patients With Giant Cell Arteritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: GSK decision to return rights to sirukumab to Janssen and discontinue sirukumab development in giant cell arteritis.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201677
Record Dates: First submitted 2015-07-06; First posted 2015-08-24 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis, Sirukumab, Prednisone
MeSH Terms: conditions — Giant Cell Arteritis | interventions — sirukumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part A: Sirukumab, Dose 1+prednisone (6-month taper) (Experimental): Subjects will receive blinded sirukumab 100 mg subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-month oral prednisone taper regimen.
  Interventions: Drug: Sirukumab; Drug: Prednisone; Drug: Placebo to match prednisone
- Part A: Sirukumab, Dose 1+prednisone (3-month taper) (Experimental): Subjects will receive blinded sirukumab 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month oral prednisone taper regimen.
  Interventions: Drug: Sirukumab; Drug: Prednisone; Drug: Placebo to match prednisone
- Part A: Sirukumab, Dose 2+prednisone (6-month taper) (Experimental): Subjects will receive blinded sirukumab 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month oral prednisone taper regimen.
  Interventions: Drug: Sirukumab; Drug: Prednisone; Drug: Placebo to match prednisone
- Part A:Placebo to match sirutkumab+prednisone (6-month taper) (Placebo Comparator): Subjects will receive blinded placebo to match sirutkumab q2w for 52 weeks plus a pre-specified maximum of 6-month oral prednisone taper regimen.
  Interventions: Drug: Placebo to match sirukumab; Drug: Prednisone; Drug: Placebo to match prednisone
- Part A:Placebo to match sirukumab+prednisone (12-month taper) (Placebo Comparator): Subjects will receive blinded placebo to match sirutkumab q2w for 52 weeks plus a pre-specified maximum of 12-month oral prednisone taper regimen.
  Interventions: Drug: Placebo to match sirukumab; Drug: Prednisone; Drug: Placebo to match prednisone
- Part B:Open-label sirukumab 100 mg SC (if applicable) (Experimental): Subjects completing Part A will receive open label 100 mg SC q2w for a maximum of 52 weeks based on remission status and disease activity at the primary 52-week endpoint or prednisone tapering status of subject during Part A. Methotrexate will be provided to subjects, alone or in addition to sirukumab treatment during Part B, based on the discretion of the investigator.
  Interventions: Drug: Sirukumab

INTERVENTIONS:
Drug: Sirukumab — Sirukumab will be provided as 1 millilitre (mL) Pre-filled Syringe (PFS), containing 100 mg/mL or 50 mg/mL of sirukuma, fitted with a spring-powered, disposable autoinjector device for single use SC administration of liquid biologic drug.
  Arms: Part A: Sirukumab, Dose 1+prednisone (3-month taper); Part A: Sirukumab, Dose 1+prednisone (6-month taper); Part A: Sirukumab, Dose 2+prednisone (6-month taper); Part B:Open-label sirukumab 100 mg SC (if applicable)
Drug: Placebo to match sirukumab — Placebo to match sirukumab will be provided as 1.0 mL PFS fitted with a spring-powered, disposable autoinjector device for single use SC administration of liquid biologic drug.
  Arms: Part A:Placebo to match sirukumab+prednisone (12-month taper); Part A:Placebo to match sirutkumab+prednisone (6-month taper)
Drug: Prednisone — Prednisone will be provided as tablets with dosage level up to-60 mg/day. The prednisone dose for all subjects will be determined by the Investigator and starting doses will be within 20-60 mg prednisone at Baseline (Randomization).
  Arms: Part A: Sirukumab, Dose 1+prednisone (3-month taper); Part A: Sirukumab, Dose 1+prednisone (6-month taper); Part A: Sirukumab, Dose 2+prednisone (6-month taper); Part A:Placebo to match sirukumab+prednisone (12-month taper); Part A:Placebo to match sirutkumab+prednisone (6-month taper)
Drug: Placebo to match prednisone — Placebo to match prednisone will be provided as tablets.
  Arms: Part A: Sirukumab, Dose 1+prednisone (3-month taper); Part A: Sirukumab, Dose 1+prednisone (6-month taper); Part A: Sirukumab, Dose 2+prednisone (6-month taper); Part A:Placebo to match sirukumab+prednisone (12-month taper); Part A:Placebo to match sirutkumab+prednisone (6-month taper)

SUMMARY:
Sirukumab is a fully human anti-interleukin-6 (IL-6) immunoglobulin G1-kappa with a high affinity and specificity for binding to the human IL-6 molecule that may have therapeutic benefit in the treatment of giant cell arteritis (GCA) by interruption of multiple pathogenic pathways. Sirukumab inhibits IL-6-mediated signal transducer and activator of transcription 3 (STAT3) phosphorylation, resulting in the inhibition of the biological effect of IL-6. This study will evaluate the efficacy and safety of sirukumab to characterize the benefit-to-risk profile of sirukumab in the treatment of active GCA. The study will be conducted in 2 distinct parts (Part A and Part B) and consists of the following phases: Screening phase, Part A: 52-week double-blind treatment phase, Part B: 104-week extension phase with the option to receive open-label sirukumab based on disease status and a 16-week follow-up phase if applicable.

Approximately 204 subjects with a diagnosis of GCA and active disease within 6 weeks of baseline will be randomized into Part A, the 52-week double-blind treatment phase, to receive one of two doses of sirukumab or placebo, each in addition to a pre-specified prednisone taper. The efficacy and safety of sirukumab in sustaining remission will be assessed at Week 52. Subjects completing Part A of the study will be eligible to enter Part B, the 104-week extension phase, designed to investigate the long-term maintenance of remission and safety following cessation of sirukumab treatment and to assess long-term corticosteroid use. Subjects with active GCA at the end of Part A or those with new onset of GCA flare during the first 52 weeks of Part B will be eligible to receive open-label sirukumab. Subjects will need to have follow-up safety evaluations for at least 16 weeks after receiving the last dose of study drug, applicable only for those who are withdrawn prematurely from the study or whose open-label sirukumab treatment in Part B completes after Week 88.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA defined by the following Revised GCA Diagnosis Criteria:

Age >=50 years. History of ESR >=50 millimeter/hour (mm/hour) or CRP >=2.45 milligram/deciliter(mg/dL).

Presence of at least one of the following: Unequivocal cranial symptoms of GCA; Unequivocal symptoms of polymyalgia rheumatic (PMR).

Presence of at least one of the following: Temporal artery biopsy revealing features of GCA; Evidence of large-vessel vasculitis by angiography or cross-sectional imaging.

* Active GCA within 6 weeks of Randomization (Baseline) where active disease is defined by an ESR >=30 mm/hr or CRP >=1 mg/dL AND the presence of at least one of the following:

Unequivocal cranial symptoms of GCA; Unequivocal symptoms of PMR; Other features judged by the clinician investigator to be consistent with GCA or PMR flares.

* At screening, receiving or able to receive prednisone 20-60 mg/day for the treatment of active GCA.
* Clinically stable GCA disease at baseline such that the subject is able to safely participate in the blinded prednisone taper regimen in the opinion of the investigator.
* Practicing acceptable methods of birth control if a female of child-bearing potential.
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

* Are pregnant or breastfeeding.
* Recent (within the past 12 weeks) or planned major surgery that would impact on study procedures or assessments.
* Organ transplantation recipients (except corneas within 3 months prior to baseline visit).
* Had prior treatment with any of the following:

Systemic immunosuppressives) within 4 weeks of baseline; Biologic agents targeted at reducing tumor necrosis factor-alpha (TNF-alpha) within 2-8 weeks of baseline, depending on the agent; Any prior use of tocilizumab or other anti-IL-6 agents; B-cell depleting agents (eg, rituximab) within 12 months prior to baseline or longer if B cell counts have not returned to normal range or baseline levels; Cytotoxic drugs such as cyclophosphamide, chlorambucil, nitrogen mustard, or other alkylating agents within 4 weeks of baseline; Abatacept within 8 weeks of baseline; Tofacitinib within 4 weeks of baseline; Methotrexate use within 2 weeks of baseline.

Methylprednisolone > 100 mg/day intravenous (IV) (or equivalent) within 8 weeks of baseline.

* History of severe allergic reactions to monoclonal antibodies, human proteins, or excipients.
* Evidence of serious concomitant disease, which in the opinion of the investigator makes them unsuitable for participation in the study.
* Major ischemic event, unrelated to GCA, within 12 weeks of screening.
* Marked baseline prolongation of corrected QT (QTc) interval >= 450 milliseconds (msec) (QTc by Bazett's formula [QTcB ]or QTc by Fridericia's formula [QTcF] ), history of Torsade de Pointes, family history of long QT syndrome, history of second or third degree heart block.
* Current liver disease that could interfere with the trial
* History of or current active diverticulitis, inflammatory bowel disease, or other symptomatic gastrointestinal tract condition that might predispose to bowel perforation.
* History of known demyelinating diseases such as multiple sclerosis or optic neuritis.
* Active infections, or history of recurrent infections or have required management of acute or chronic infections, as follows:

Currently on any suppressive therapy for a chronic infection, history or suspicion of chronic infection, hospitalization for treatment of infection within 60 days of the baseline visit, or use of parenteral (IV) or intra-muscular [IM]) antimicrobials within 60 days of baseline or oral antimicrobials within 30 days of baseline

* Primary or secondary immunodeficiency or any other autoimmune disease.
* Human immunodeficiency virus (HIV) infection, hepatitis C or hepatitis B infection
* Live virus or bacterial vaccination within 3 months before the first administration of study drug

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- United States (12):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Vancouver, Washington
- Australia (6):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Malvern East, Victoria
  - GSK Investigational Site, Victoria Park, Western Australia
- Belgium (2):
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- France (3):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
- Germany (10):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Bad Abbach
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Kirchheim unter Teck
  - GSK Investigational Site, München
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
- Italy (3):
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano
- Netherlands (3):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Nijmegen
- New Zealand (2):
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Timaru
- GSK Investigational Site, Krakow, Poland
- Spain (4):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, San Cristóbal de La Laguna
- United Kingdom (8):
  - GSK Investigational Site, Westcliff-on-Sea, Essex
  - GSK Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - GSK Investigational Site, Bury St Edmunds, Suffolk
  - GSK Investigational Site, Sheffield, Yorkshire
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Reading

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Schmidt WA, Dasgupta B, Luqmani R, Unizony SH, Blockmans D, Lai Z, Kurrasch RH, Lazic I, Brown K, Rao R. A Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Sirukumab in the Treatment of Giant Cell Arteritis. Rheumatol Ther. 2020 Dec;7(4):793-810. doi: 10.1007/s40744-020-00227-2. Epub 2020 Aug 25. PMID 32844378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of sirukumab in treatment of participants with Giant Cell Arteritis (GCA). A total of 161 participants were enrolled.
Pre-assignment Details: This study was conducted in 2 distinct parts (Part A and Part B), Part A was a 52-week double-blind treatment phase and Part B was a 104-week long-term extension phase with the option to receive open-label sirukumab (SIR) (up to a 52-week duration of open-label treatment). This study was terminated early by sponsor.
Groups:
- Part A:SIR 100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen
- Part A:SIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen
- Part A:SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- Part A:Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- Part A:Placebo SC q2w+12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen
- Part B:SIR 100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen in Part A
- Part B:SIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen in Part A
- Part B:SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A
- Part B:Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A
- Part B:Placebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen in Part A
Period: Part A (52 Weeks)
Arm/Group | Part A:SIR 100 mg SC q2w+6 Month Prednisone | Part A:SIR 100 mg SC q2w+3 Month Prednisone | Part A:SIR 50 mg SC q4w+6 Month Prednisone | Part A:Placebo SC q2w + 6 Month Prednisone | Part A:Placebo SC q2w+12 Month Prednisone | Part B:SIR 100 mg SC q2w+6 Month Prednisone | Part B:SIR 100 mg SC q2w+3 Month Prednisone | Part B:SIR 50 mg SC q4w+6 Month Prednisone | Part B:Placebo SC q2w + 6 Month Prednisone | Part B:Placebo SC q2w + 12 Month Prednisone
Started | 42 | 39 | 26 | 27 | 27 | 0 | 0 | 0 | 0 | 0
Completed Part A and Didn't Enter Part B (2 Participants completed Part A then withdrew. They are counted again in withdrawals) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Part A and entered Part B) | 8 | 5 | 4 | 5 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 34 | 34 | 22 | 22 | 23 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor request | 24 | 24 | 18 | 18 | 19 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (104 Weeks)
Arm/Group | Part A:SIR 100 mg SC q2w+6 Month Prednisone | Part A:SIR 100 mg SC q2w+3 Month Prednisone | Part A:SIR 50 mg SC q4w+6 Month Prednisone | Part A:Placebo SC q2w + 6 Month Prednisone | Part A:Placebo SC q2w+12 Month Prednisone | Part B:SIR 100 mg SC q2w+6 Month Prednisone | Part B:SIR 100 mg SC q2w+3 Month Prednisone | Part B:SIR 50 mg SC q4w+6 Month Prednisone | Part B:Placebo SC q2w + 6 Month Prednisone | Part B:Placebo SC q2w + 12 Month Prednisone
Started | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 4 | 5 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 4 | 5 | 4
Not completed — Sponsor request | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 3 | 5 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SIR100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen
- SIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen
- SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- Placebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen
- Total: Total of all reporting groups
Arm/Group | SIR100 mg SC q2w+6 Month Prednisone | SIR 100 mg SC q2w+3 Month Prednisone | SIR 50 mg SC q4w+6 Month Prednisone | Placebo SC q2w + 6 Month Prednisone | Placebo SC q2w + 12 Month Prednisone | Total
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (7.25) | 68.1 (6.72) | 67.5 (9.45) | 71.6 (7.10) | 70.7 (8.96) | 69.6 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 19 | 23 | 21 | 124
  Male | 11 | 9 | 7 | 4 | 6 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 1 | 0 | 0 | 0 | 1
  White: Arabic/North African Heritage | 1 | 1 | 0 | 0 | 0 | 2
  White/Caucasian/European Heritage | 41 | 37 | 25 | 26 | 27 | 156
  Mixed Race | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants in Sustained Remission at Week 52
Description: Sustained remission was defined as having achieved all of the following: 1) remission at Week 12, 2) absence of disease flare Week 12 through Week 52, 3) completion of the assigned prednisone taper, and 4) no requirement for rescue therapy through Week 52. Remission was defined as absence of clinical signs and symptoms of GCA and normalization of erythrocyte sedimentation rate (ESR) [<30 millimeters per hour] and C-reactive Protein (CRP) [<1 milligram/deciliter]) and flare was defined as recurrence of symptoms attributable to active GCA, with or without elevations in ESR and/or CRP. Data for number of participants in sustained remission at Week 52 is presented. Only those participants who completed Week 52 visit or withdrew before 10 Oct 2017 were included in the analysis.
Time Frame: Week 52
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants who received at least 1 dose of SC investigational product (IP).
Measure: Count of Participants; unit: Participants
Groups:
- PartA:SIR 100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen
- PartA:SIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen
- PartA:SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- PartA:Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- PartA:Placebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 17 | 13 | 9 | 9 | 7
Participants | 3 | 2 | 1 | 0 | 0

2. Secondary Outcome: Part B: Number of Participants Who Remained in Sustained Remission Without Requirement for Rescue Therapy or Treatment Change at Week 24
Description: Participants who remained in sustained remission without requirement for rescue therapy or treatment change at each scheduled visit of Part B were defined as participants having achieved all of the following criteria: 1. Participants in sustained remission at the Week 52 visit of Part A, 2. Absence of disease flare, 3. No requirement for rescue therapy at any time through Week 24 of Part B, 4. No requirement for treatment change at any time through Week 24 of Part B. Remission was defined as absence of clinical signs and symptoms of GCA and normalization of ESR [<30 millimeters per hour] and CRP [<1 milligram/deciliter]) and flare was defined as recurrence of symptoms attributable to active GCA, with or without elevations in ESR and/or CRP.
Time Frame: Week 24
Population: ITT-Part B Population included all randomized participants who received at least 1 dose of SC IP in Part A and entered Part B.
Measure: Count of Participants; unit: Participants
Groups:
- PartB:SIR 100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen in Part A
- PartB:SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | Part B:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | Part B:Placebo SC q2w + 6 Month Prednisone | Part B:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 0
Participants | NA — 5 participants in clinical remission entered Part B, all withdrew prior to week 24. Therefore, No data was available for week 24 for this population. | NA — 5 participants in clinical remission entered Part B, all withdrew prior to week 24. Therefore, No data was available for week 24 for this population. | NA — 5 participants in clinical remission entered Part B, all withdrew prior to week 24. Therefore, No data was available for week 24 for this population. |  |

3. Secondary Outcome: Part A: Cumulative Prednisone Dose Over Time
Description: Cumulative prednisone is the dose from the taper (both open-label and blinded) as well as from the corticosteroid rescue therapies. Cumulative dose at the specified Week was derived as the sum of all the doses from Baseline to the specified Week at each visit was calculated based on the number of participants who attended that visit. For the main analysis of cumulative prednisone dose over time. Data for Prednisone Dose- Study Drug and Prednisone Equivalent Concomitant Therapy for part A is presented. ITT population and the number of participants included at specific time points were based on the participants who attended a scheduled or unscheduled visit mapped to that time point and received a total prednisone dose greater than 0 mg.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Milligrams
  Week 2, n= 40,39,26,27,26: number analyzed (Participants) | 40 | 39 | 26 | 27 | 26
  Week 2, n= 40,39,26,27,26 | 439.575 (237.8990) | 464.923 (299.6445) | 424.577 (270.2183) | 432.815 (315.6851) | 430.846 (241.3540)
  Week 4,n=40,39,26,25,27: number analyzed (Participants) | 40 | 39 | 26 | 25 | 27
  Week 4,n=40,39,26,25,27 | 701.100 (370.9798) | 741.115 (436.4205) | 701.192 (439.7251) | 705.480 (601.9706) | 751.407 (431.3442)
  Week 8,n=37, 37,26,23,26: number analyzed (Participants) | 37 | 37 | 26 | 23 | 26
  Week 8,n=37, 37,26,23,26 | 1086.676 (600.7400) | 987.730 (559.4458) | 1014.731 (592.3515) | 1161.391 (1202.8504) | 1129.077 (546.8037)
  Week 12,n=34,32,24,22,24: number analyzed (Participants) | 34 | 32 | 24 | 22 | 24
  Week 12,n=34,32,24,22,24 | 1344.441 (779.6775) | 1063.773 (619.4002) | 1208.167 (650.6975) | 1379.409 (1255.4397) | 1462.917 (630.1717)
  Week 16,n=32,30,24,22,22: number analyzed (Participants) | 32 | 30 | 24 | 22 | 22
  Week 16,n=32,30,24,22,22 | 1545.602 (964.3264) | 1182.288 (718.6186) | 1348.750 (689.2484) | 1672.795 (1261.7121) | 1729.977 (701.3734)
  Week 20,n=29,27,21,24,19: number analyzed (Participants) | 29 | 27 | 21 | 24 | 19
  Week 20,n=29,27,21,24,19 | 1690.302 (1173.6005) | 1339.546 (888.5007) | 1475.786 (734.7667) | 1646.177 (701.5240) | 2041.632 (771.3504)
  Week 24,n=30,25,19,18,17: number analyzed (Participants) | 30 | 25 | 19 | 18 | 17
  Week 24,n=30,25,19,18,17 | 1878.458 (1333.1175) | 1495.015 (1055.9615) | 1626.342 (813.8284) | 1917.444 (861.6887) | 2299.471 (840.8758)
  Week 28,n=24,23,15,17,15: number analyzed (Participants) | 24 | 23 | 15 | 17 | 15
  Week 28,n=24,23,15,17,15 | 2000.813 (1594.5982) | 1575.549 (1170.7294) | 1797.533 (933.3753) | 2141.294 (1082.2754) | 2387.800 (741.1663)
  Week 32,n=19,21,13,15,18: number analyzed (Participants) | 19 | 21 | 13 | 15 | 18
  Week 32,n=19,21,13,15,18 | 2216.000 (1953.8211) | 1716.863 (1328.1426) | 1859.346 (858.5431) | 2531.417 (1327.9125) | 2404.500 (808.8642)
  Week 36,n=19,17,14,13,14: number analyzed (Participants) | 19 | 17 | 14 | 13 | 14
  Week 36,n=19,17,14,13,14 | 2321.711 (2090.2393) | 1803.919 (1536.5304) | 1705.214 (802.8858) | 2617.817 (1636.2516) | 2717.696 (897.0689)
  Week 40,n=18,15,11,13,12: number analyzed (Participants) | 18 | 15 | 11 | 13 | 12
  Week 40,n=18,15,11,13,12 | 2003.264 (1426.0271) | 2023.342 (1651.4092) | 1842.500 (904.4136) | 2960.144 (1736.2249) | 2963.865 (909.0195)
  Week 44,n=17,13,10,12,13: number analyzed (Participants) | 17 | 13 | 10 | 12 | 13
  Week 44,n=17,13,10,12,13 | 2051.603 (1588.9627) | 1481.115 (1381.3957) | 1980.733 (1444.8664) | 2783.542 (1776.0608) | 2954.760 (1022.5491)
  Week 48,n=10,16,9,8,11: number analyzed (Participants) | 10 | 16 | 9 | 8 | 11
  Week 48,n=10,16,9,8,11 | 1821.325 (1139.5986) | 1601.656 (1362.9717) | 1562.333 (828.5650) | 2859.208 (1882.7422) | 3167.898 (1195.4020)
  Week 52,n=11,10,6,7,6: number analyzed (Participants) | 11 | 10 | 6 | 7 | 6
  Week 52,n=11,10,6,7,6 | 2974.295 (2966.6259) | 2418.213 (2085.2345) | 2556.222 (1363.1832) | 3157.054 (1988.0610) | 3603.229 (1477.6777)

4. Secondary Outcome: Part B: Number of Participants in Sustained Remission Over Time
Description: Sustained remission was defined as having achieved all of the following: 1) remission at Week 12 (absence of signs and symptoms of GCA and normalization of ESR and CRP), 2) absence of disease flare Week 12 through Week 52 with or without elevations in ESR and/or CRP, 3) completion of the assigned prednisone taper, and 4) no requirement for rescue therapy through Week 52. Remission was defined as absence of clinical signs and symptoms of GCA and normalization of ESR [<30millimeters per hour] and CRP [<1milligram/deciliter]) and Flare was defined as recurrence of symptoms attributable to active GCA, with or without elevations in ESR and/or CRP. Data for number of participants in sustained remission over time for Part B is presented. Only participants who were in sustained remission at Week 52 of Part A, who Completed the Week X Visit of Part B or who Withdraw before 10th of October 2017 were included in the analysis.
Time Frame: Weeks 4, 8 and 12
Population: ITT-Part B Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Groups:
- PartB:SIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen in Part A
- PartB:Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A
- PartB:Placebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen in Part A
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 0
Participants
  Week 4,n=1,1,1,0,0: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0
  Week 4,n=1,1,1,0,0 | 1 | 1 | 1 |  |
  Week 8,n=1,0,1,0,0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0
  Week 8,n=1,0,1,0,0 | 1 |  | 1 |  |
  Week 12,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 12,n=1,0,0,0,0 | 1 |  |  |  |

5. Secondary Outcome: Part A: Time to First Disease Flare After Clinical Remission
Description: Clinical remission was defined as absence of clinical signs and symptoms of GCA, which was determined by a lack of flare for the participant. If a participant had a flare, they had one or more signs and symptoms, and therefore are not considered as being in clinical remission. Time to first disease flare (days) was calculated as (Date of First Flare - Date of Clinical Remission + 1 day). Data for Time to first disease flare after clinical remission for part A is presented.
Time Frame: Week 52
Population: ITT Population. Only participants who achieved clinical remission were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 40 | 39 | 26 | 27 | 27
Days | NA [NA to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [NA to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [176.0 to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [99.0 to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [183.0 to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52

6. Secondary Outcome: Part B: Time to First Disease Flare for Participants in Sustained Remission
Description: Clinical remission was defined as absence of clinical signs and symptoms of GCA. If a participant had a flare, they had one or more signs and symptoms, and therefore are not considered as being in clinical remission. Time to event (days) is defined as the duration in days from the date of the Week 52 visit of Part A to the start date of Event (Date of First Flare - Date of Week 52 visit of Part A + 1). Data for Time to first disease flare after clinical remission for part B is presented.
Time Frame: Week 52
Population: ITT-Part B Population. Only those participants with available data at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 0
Days | NA [NA to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [NA to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 | NA [NA to NA] — No. of participants achieving remission was not sufficient to calculate the median survival time from the Kaplan-Meier analysis, as less than half of subjects who achieved clinical remission in any dose arm had a flare at or before Week 52 |  |

7. Secondary Outcome: Part A: Number of Disease Flares Over Time
Description: This summarizes disease flares over time with no adjustment for exposure to study drugs, calculated by taking the last visit before a participant withdrew and then counting the number of participants with at least 1 flare up to that point and summing up the total number of flares experienced by each of these participants; participants who did not reach Week 2 were not included in this analysis. Data for number of disease flares per participant over time for part A were presented.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Number; unit: Disease flares
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Disease flares
  Week 2, n=38, 39,26,25,27: number analyzed (Participants) | 38 | 39 | 26 | 25 | 27
  Week 2, n=38, 39,26,25,27 | 1 | 2 | 2 | 0 | 2
  Week 4, n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  Week 4, n=37,37,25,23,27 | 3 | 4 | 3 | 0 | 2
  Week 8, n=34,32,24,23,23: number analyzed (Participants) | 34 | 32 | 24 | 23 | 23
  Week 8, n=34,32,24,23,23 | 2 | 6 | 3 | 1 | 5
  Week 12, n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  Week 12, n=32,29,24,22,22 | 4 | 9 | 4 | 4 | 4
  Week 16, n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16, n=28,26,22,19,19 | 4 | 9 | 5 | 9 | 4
  Week 20, n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20, n=26,23,19,18,16 | 4 | 9 | 6 | 10 | 3
  Week 24, n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  Week 24, n=23,21,16,17,16 | 6 | 9 | 8 | 11 | 5
  Week 28, n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  Week 28, n=19,18,12,14,14 | 5 | 8 | 8 | 11 | 5
  Week 32, n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32, n=19,15,10,12,13 | 5 | 8 | 5 | 10 | 6
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 3 | 8 | 5 | 10 | 6
  Week 40, n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40, n=15,11,9,10,10 | 2 | 7 | 5 | 8 | 5
  Week 44, n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44, n=11,11,6,8,9 | 1 | 8 | 3 | 6 | 7
  Week 48, n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48, n=9,8,5,8,5 | 1 | 4 | 1 | 7 | 3
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 1 | 2 | 1 | 7 | 4

8. Secondary Outcome: Part A: Number of Participants With at Least One Hospitalization for Disease Flare
Description: Number of participants with at least one hospitalization for disease flare at a given visit is the number of participants with at least one hospitalization for disease flare between first SC IP intake and the day of the given visit. Data for participants requiring at least one hospitalization for disease flare for part A is presented.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Participants
  Week 2, n=38, 39,26,25,27: number analyzed (Participants) | 38 | 39 | 26 | 25 | 27
  Week 2, n=38, 39,26,25,27 | 0 | 0 | 0 | 0 | 0
  Week 4, n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  Week 4, n=37,37,25,23,27 | 0 | 0 | 0 | 0 | 0
  Week 8, n=34,32,24,23,23: number analyzed (Participants) | 34 | 32 | 24 | 23 | 23
  Week 8, n=34,32,24,23,23 | 0 | 0 | 0 | 0 | 0
  Week 12, n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  Week 12, n=32,29,24,22,22 | 1 | 0 | 0 | 0 | 0
  Week 16, n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16, n=28,26,22,19,19 | 1 | 0 | 0 | 0 | 0
  Week 20, n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20, n=26,23,19,18,16 | 1 | 0 | 1 | 0 | 0
  Week 24, n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  Week 24, n=23,21,16,17,16 | 1 | 0 | 1 | 0 | 0
  Week 28, n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  Week 28, n=19,18,12,14,14 | 0 | 0 | 1 | 0 | 0
  Week 32, n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32, n=19,15,10,12,13 | 0 | 0 | 0 | 0 | 0
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 0 | 0 | 0 | 0 | 0
  Week 40, n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40, n=15,11,9,10,10 | 0 | 0 | 0 | 0 | 0
  Week 44, n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44, n=11,11,6,8,9 | 0 | 0 | 0 | 0 | 0
  Week 48, n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48, n=9,8,5,8,5 | 0 | 0 | 0 | 0 | 0
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part A: Number of Hospitalizations for Disease Flare Over Time
Description: Number of hospitalizations for disease flare at given visit is the number of hospitalizations for disease flare between first SC IP intake and the day of the of the given visit.. Data for number of hospitalizations for disease flare over time for part A was presented.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Number; unit: Number of Hospitalizations
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Number of Hospitalizations
  Week 2, n=38, 39,26,25,27: number analyzed (Participants) | 38 | 39 | 26 | 25 | 27
  Week 2, n=38, 39,26,25,27 | 0 | 0 | 0 | 0 | 0
  Week 4, n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  Week 4, n=37,37,25,23,27 | 0 | 0 | 0 | 0 | 0
  Week 8, n=34,32,24,23,23: number analyzed (Participants) | 34 | 32 | 24 | 23 | 23
  Week 8, n=34,32,24,23,23 | 0 | 0 | 0 | 0 | 0
  Week 12, n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  Week 12, n=32,29,24,22,22 | 2 | 0 | 0 | 0 | 0
  Week 16, n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16, n=28,26,22,19,19 | 2 | 0 | 0 | 0 | 0
  Week 20, n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20, n=26,23,19,18,16 | 2 | 0 | 1 | 0 | 0
  Week 24, n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  Week 24, n=23,21,16,17,16 | 2 | 0 | 1 | 0 | 0
  Week 28, n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  Week 28, n=19,18,12,14,14 | 0 | 0 | 1 | 0 | 0
  Week 32, n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32, n=19,15,10,12,13 | 0 | 0 | 0 | 0 | 0
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 0 | 0 | 0 | 0 | 0
  Week 40, n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40, n=15,11,9,10,10 | 0 | 0 | 0 | 0 | 0
  Week 44, n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44, n=11,11,6,8,9 | 0 | 0 | 0 | 0 | 0
  Week 48, n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48, n=9,8,5,8,5 | 0 | 0 | 0 | 0 | 0
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part A: Mean 36-item Short Form Health Survey Version 2 (SF-36 v2) Acute Score Over Time
Description: SF-36v2 acute health survey questionnaire consists of the following 8 multi-item scales: 1. Limitations in physical functioning due to health problems, 2. Limitations in usual role activities due to physical health problems, 3. Bodily pain, 4. General mental health (psychological distress and well-being), 5. Limitations in usual role activities due to personal or emotional problems, 6. Limitations in social functioning due to physical or mental health problems. 7. Vitality (energy and fatigue) and 8. General health perception. These 8 scales were scored from 0 to 100, 0 (worst score) to 100 (best score) where higher scores indicates better health. Data for Physical Component Summary (PCS), Mental Component Summary (MCS) scores was presented.
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  PCS,Baseline, n=42,38,25,23,27: number analyzed (Participants) | 42 | 38 | 25 | 23 | 27
  PCS,Baseline, n=42,38,25,23,27 | 49.258 (11.7655) | 43.271 (12.3169) | 42.919 (11.7298) | 49.240 (9.2759) | 45.470 (12.8498)
  PCS,Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  PCS,Week 12, n=31,28,24,22,22 | 51.519 (10.5352) | 43.128 (11.4559) | 43.655 (11.0324) | 48.552 (10.4184) | 47.007 (12.8749)
  PCS,Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  PCS,Week 24, n=23,20,15,17,16 | 50.023 (11.4731) | 45.677 (12.1192) | 45.097 (15.0552) | 46.911 (9.2901) | 44.280 (11.4740)
  PCS,Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  PCS,Week 36, n=15,13,10,12,13 | 51.989 (10.7521) | 47.069 (12.7103) | 46.005 (12.2496) | 48.336 (10.0154) | 44.946 (10.1921)
  PCS,Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  PCS,Week 52, n=9,5,5,5,4 | 50.269 (10.8743) | 53.690 (7.9049) | 53.608 (7.7721) | 52.026 (6.4892) | 53.143 (12.8351)
  MCS,Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  MCS,Week 12, n=31,28,24,22,22 | 43.955 (4.6164) | 45.264 (5.7982) | 46.393 (6.1792) | 43.746 (5.3179) | 43.182 (4.6707)
  MCS,Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  MCS,Week 24, n=23,20,15,17,16 | 44.538 (5.6952) | 45.954 (5.4884) | 44.877 (6.5210) | 45.372 (6.4561) | 45.526 (5.8924)
  MCS,Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  MCS,Week 36, n=15,13,10,12,13 | 45.258 (5.2429) | 45.540 (4.8330) | 44.550 (6.7199) | 42.959 (4.8484) | 46.755 (4.8284)
  MCS,Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  MCS,Week 52, n=9,5,5,5,4 | 44.810 (6.4757) | 45.008 (2.2373) | 42.004 (5.5695) | 42.258 (4.1002) | 42.125 (1.9020)

11. Secondary Outcome: Part A: Mean EuroQol - 5 Dimensions, 5 Levels (EQ-5D-5L) Index Score Over Time
Description: EuroQoL-5 Dimensions consist of 2 elements: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprised of following 5 dimensions: 1.Mobility, 2.Self-Care, 3.Usual Activities, 4.Pain/Discomfort and 5.Anxiety/Depression. Each of these 5 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The digits for each of 5 dimensions were combined in a 5-digit number describing the participant's health state: e.g. state 11111 indicates no problem on any of the 5 dimensions. Index score was derived from the 5 dimensions scores using UK tariff. The weights based from the UK population was used for conversion, regardless of the origin country of participant. The score ranged from -0.594 (worst score) to 1.000 (best score).
Time Frame: Baseline (Week 0) and Weeks 12, 24, 36, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,38,25,23,27: number analyzed (Participants) | 42 | 38 | 25 | 23 | 27
  Baseline, n=42,38,25,23,27 | 0.7918 (0.20589) | 0.6681 (0.31299) | 0.6912 (0.19348) | 0.7429 (0.22387) | 0.7554 (0.16610)
  Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, n=31,28,24,22,22 | 0.7866 (0.22042) | 0.7024 (0.22087) | 0.7452 (0.17942) | 0.7228 (0.16993) | 0.7069 (0.22289)
  Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, n=23,20,15,17,16 | 0.7485 (0.20310) | 0.7217 (0.21397) | 0.7135 (0.24006) | 0.7323 (0.10346) | 0.7301 (0.11498)
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 0.8011 (0.13468) | 0.7454 (0.22373) | 0.7774 (0.11809) | 0.6950 (0.15242) | 0.7506 (0.17536)
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 0.8210 (0.13502) | 0.7628 (0.15352) | 0.8092 (0.04275) | 0.7864 (0.05892) | 0.8068 (0.06050)

12. Secondary Outcome: Part A: Mean EQ-5D-5L Visual Analogue Scale (VAS) Over Time
Description: EQ-5D essentially consists of 2 elements: the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system comprised of the following 5 dimensions: 1.Mobility, 2.Self-Care, 3.Usual Activities, 4.Pain/Discomfort and 5.Anxiety/Depression. Each of these 5 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The digits for each of the 5 dimensions were combined in a 5-digit number describing the participant's health state: e.g. state 11111 indicates no problem on any of the 5 dimensions. The index score was derived from the 5 dimensions scores using UK tariff. The weights based from the UK population was used for the conversion, regardless of the origin country of participant. The score ranged from -0.594 (worst score) to 1 (best score). The EQ VAS records the respondent's self-rated health on a vertical line, VAS where the endpoints are 'Best imaginable health state' and 'Worst imaginable health state'.
Time Frame: Baseline (Week 0) and Weeks 12, 24, 36, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,38,25,23,27: number analyzed (Participants) | 42 | 38 | 25 | 23 | 27
  Baseline, n=42,38,25,23,27 | 67.0 (17.83) | 65.6 (21.43) | 57.0 (17.61) | 62.1 (23.81) | 65.1 (16.00)
  Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, n=31,28,24,22,22 | 74.3 (19.77) | 64.2 (22.89) | 68.4 (19.39) | 63.3 (22.61) | 65.5 (21.33)
  Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, n=23,20,15,17,16 | 74.6 (16.26) | 70.6 (24.05) | 65.1 (23.11) | 64.9 (19.03) | 61.5 (19.71)
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 79.5 (9.55) | 73.9 (24.55) | 66.9 (20.72) | 68.3 (18.66) | 61.6 (21.29)
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 79.9 (9.74) | 80.6 (16.50) | 78.4 (14.77) | 60.2 (26.33) | 70.0 (27.41)

13. Secondary Outcome: Part A: Mean Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-Fatigue) Scores Over Time
Description: The FACIT-Fatigue is a 13-item questionnaire formatted for self-administration that assesses participant reported fatigue and its impact upon daily activities and function over the past seven days. Participants were asked to answer each question using a 5-point Likert-type scale (4 = Not at all; 3 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 0 = Very Much) where 0 is a bad response and 4 is good response. Each of the 13 items of the FACIT-Fatigue Scale ranges from 0-4, with a range of possible total score from 0-52, 0 (Extreme fatigue) to 52 (No fatigue) where 0 being the worst possible score and 52 the best (i.e. less fatigue). Scores below 30 indicate severe fatigue. Each negatively-worded item response was recoded so that 0 is a bad response and 4 is good response. All responses were added with equal weight to obtain the total score. The total score was calculated as the sum of all the individual items after recoding some of the items.
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,38,25,23,27: number analyzed (Participants) | 42 | 38 | 25 | 23 | 27
  Baseline, n=42,38,25,23,27 | 38.7 (10.72) | 34.2 (12.25) | 31.1 (9.89) | 38.0 (8.37) | 34.1 (13.32)
  Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, n=31,28,24,22,22 | 40.2 (8.83) | 32.7 (11.25) | 34.3 (11.12) | 38.5 (9.82) | 35.5 (13.34)
  Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, n=23,20,15,17,16 | 38.1 (10.48) | 36.5 (13.22) | 31.2 (13.09) | 36.2 (6.15) | 36.0 (9.18)
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 41.4 (9.41) | 38.4 (9.95) | 36.9 (10.88) | 40.9 (6.49) | 37.5 (10.02)
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 42.1 (6.72) | 43.0 (6.48) | 40.4 (5.22) | 44.0 (5.48) | 41.0 (12.25)

14. Secondary Outcome: Part A: Mean Pain Numeric Rating Scale (NRS) Scores Over Time
Description: The assessment of pain severity was made using a single pain severity item on which participants were asked to rate the severity of their average pain on a 11-point numeric rating scale ranging from 0, "no pain" to 10, "the worst pain imaginable". Data for NRS scores over time for part A is reported.
Time Frame: Baseline (Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,38,25,23,27: number analyzed (Participants) | 42 | 38 | 25 | 23 | 27
  Baseline, n=42,38,25,23,27 | 1.8 (2.31) | 2.5 (2.97) | 3.1 (2.27) | 2.6 (2.09) | 2.6 (2.39)
  Week 2, n=38,38,25,21,27: number analyzed (Participants) | 38 | 38 | 25 | 21 | 27
  Week 2, n=38,38,25,21,27 | 1.3 (1.55) | 2.8 (3.08) | 2.8 (1.96) | 2.6 (2.13) | 2.6 (2.63)
  Week 4, n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4, n=36,37,24,22,27 | 1.7 (2.16) | 3.1 (3.13) | 3.3 (2.20) | 2.4 (2.28) | 1.8 (1.72)
  Week 8, n=34,30,24,21,23: number analyzed (Participants) | 34 | 30 | 24 | 21 | 23
  Week 8, n=34,30,24,21,23 | 1.8 (2.42) | 2.9 (2.73) | 3.0 (2.54) | 2.1 (1.96) | 3.3 (2.82)
  Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, n=31,28,24,22,22 | 1.7 (2.30) | 3.6 (3.05) | 3.3 (2.42) | 2.3 (2.50) | 2.0 (2.08)
  Week 16, n=27,25,22,19,19: number analyzed (Participants) | 27 | 25 | 22 | 19 | 19
  Week 16, n=27,25,22,19,19 | 1.4 (2.22) | 3.3 (2.84) | 3.0 (2.60) | 2.4 (2.06) | 2.7 (2.16)
  Week 20, n=26,23,19,18,15: number analyzed (Participants) | 26 | 23 | 19 | 18 | 15
  Week 20, n=26,23,19,18,15 | 1.7 (2.27) | 2.9 (2.70) | 3.6 (2.63) | 1.4 (1.54) | 2.7 (2.02)
  Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, n=23,20,15,17,16 | 2.4 (2.82) | 2.5 (2.42) | 3.3 (2.94) | 2.4 (1.84) | 3.5 (2.22)
  Week 28, n=18,17,11,13,14: number analyzed (Participants) | 18 | 17 | 11 | 13 | 14
  Week 28, n=18,17,11,13,14 | 2.6 (2.38) | 2.8 (3.03) | 3.6 (2.87) | 2.3 (2.14) | 2.9 (2.40)
  Week 32, n=19,14,9,12,12: number analyzed (Participants) | 19 | 14 | 9 | 12 | 12
  Week 32, n=19,14,9,12,12 | 2.1 (2.57) | 1.9 (2.67) | 2.9 (1.90) | 2.6 (2.15) | 3.1 (2.35)
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 1.6 (1.88) | 2.0 (2.55) | 2.9 (2.02) | 2.3 (2.42) | 1.9 (1.93)
  Week 40, n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40, n=15,11,9,10,10 | 2.0 (2.54) | 2.0 (2.57) | 3.1 (2.09) | 1.9 (1.91) | 2.6 (2.07)
  Week 44, n=11,11,6,8,8: number analyzed (Participants) | 11 | 11 | 6 | 8 | 8
  Week 44, n=11,11,6,8,8 | 2.1 (2.74) | 1.9 (2.47) | 2.2 (1.72) | 1.3 (0.71) | 3.0 (2.39)
  Week 48, n=9,8,5,7,5: number analyzed (Participants) | 9 | 8 | 5 | 7 | 5
  Week 48, n=9,8,5,7,5 | 1.9 (2.42) | 0.8 (1.04) | 2.6 (0.89) | 1.6 (1.27) | 4.0 (3.74)
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 1.3 (1.66) | 0.8 (0.84) | 2.8 (2.28) | 2.2 (0.84) | 1.0 (0.82)

15. Secondary Outcome: Part A: Mean Health Assessment Questionnaire - Disability Index (HAQDI) Score Over Time
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI) indicates the extent of participant's functional ability during the past week, and was assessed for subgroup of participants with symptoms of Polymyalgia Rheumatic (PMR). HAQ-DI included 20 questions in 8 categories of functioning - dressing and grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Each functional area contains at least two questions. For each question, there is a 4-level difficulty scale that is scored from 0 (minimum) to 3 (Maximum), representing "no difficulty" (0), "some difficulty" (1), "much difficulty" (2), and "unable to do" (3) where, lower score indicates less disability and higher scores indicates worse disability. Total score was calculated as average scores of 20 questions which can be interpreted in terms of 3 categories: from 0 to 1: mild difficulties to moderate disability, from 1 to 2: disability moderate to severe, from 2 to 3: severe to very severe disability.
Time Frame: Baseline (Week 0) and Weeks 12, 24, 36 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=19,14,13,9,12: number analyzed (Participants) | 19 | 14 | 13 | 9 | 12
  Baseline, n=19,14,13,9,12 | 0.6776 (0.65658) | 1.1250 (0.75479) | 0.9615 (0.84376) | 0.8889 (0.80875) | 0.8646 (0.62034)
  Week 12, n=12,8,12,9,9: number analyzed (Participants) | 12 | 8 | 12 | 9 | 9
  Week 12, n=12,8,12,9,9 | 0.3229 (0.41785) | 1.0938 (0.91063) | 0.7292 (0.87392) | 0.5694 (0.54526) | 0.9306 (0.66764)
  Week 24, n=10, 7,7,7,9: number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
  Week 24, n=10, 7,7,7,9 | 0.5875 (0.58940) | 0.8750 (0.78395) | 0.9821 (0.92823) | 0.9107 (0.83452) | 0.9583 (0.70986)
  Week 36, n=6,5,4,4,7: number analyzed (Participants) | 6 | 5 | 4 | 4 | 7
  Week 36, n=6,5,4,4,7 | 0.5208 (0.70007) | 0.8250 (0.80816) | 0.6250 (0.51031) | 0.5625 (0.58184) | 1.0000 (0.91287)
  Week 52, n=5,2,3,1,2: number analyzed (Participants) | 5 | 2 | 3 | 1 | 2
  Week 52, n=5,2,3,1,2 | 0.3000 (0.41079) | 0.3125 (0.44194) | 0.1667 (0.14434) | 0.0000 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 0.1875 (0.26517)

16. Secondary Outcome: Part A: Number of Participants With Patient Global Impression of Change (PGIC) Score Over Time
Description: Patient-reported response to treatment was assessed using the PGIC measure, a single item completed by participant to provide a clinically meaningful summary of an individual's response to treatment. The assessment provides an estimate of the magnitude of treatment response at different time points during the study. Responses include: Much Better, Better, Slightly Better, No Change, Slightly Worse, Worse, and Much Worse. The categorical data of participant rating of change is summarized by treatment group, visit and response category.
Time Frame: Weeks 12, 24 and 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Participants
  Week 12,Much Better, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,Much Better, n=31,28,24,22,22 | 11 | 7 | 2 | 5 | 5
  Week 12,Better, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,Better, n=31,28,24,22,22 | 11 | 10 | 11 | 4 | 11
  Week 12, Slightly Better, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, Slightly Better, n=31,28,24,22,22 | 3 | 5 | 4 | 8 | 3
  Week 12,No Change, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,No Change, n=31,28,24,22,22 | 3 | 3 | 4 | 0 | 3
  Week 12,Slightly Worse, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,Slightly Worse, n=31,28,24,22,22 | 1 | 1 | 2 | 4 | 0
  Week 12,Worse, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,Worse, n=31,28,24,22,22 | 2 | 2 | 1 | 1 | 0
  Week 12,Much Worse, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12,Much Worse, n=31,28,24,22,22 | 0 | 0 | 0 | 0 | 0
  Week 24,Much Better, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24,Much Better, n=23,20,15,17,16 | 11 | 6 | 6 | 5 | 6
  Week 24,Better, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24,Better, n=23,20,15,17,16 | 7 | 8 | 4 | 6 | 6
  Week 24, Slightly Better,n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, Slightly Better,n=23,20,15,17,16 | 2 | 2 | 0 | 4 | 1
  Week 24,No Change, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24,No Change, n=23,20,15,17,16 | 1 | 2 | 2 | 1 | 1
  Week 24,Slightly Worse, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24,Slightly Worse, n=23,20,15,17,16 | 2 | 1 | 2 | 1 | 1
  Week 24, Worse,n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, Worse,n=23,20,15,17,16 | 0 | 1 | 1 | 0 | 1
  Week 24, Much Worse,n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, Much Worse,n=23,20,15,17,16 | 0 | 0 | 0 | 0 | 0
  Week 52,Much Better, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Much Better, n=9,5,5,5,4 | 6 | 3 | 3 | 2 | 3
  Week 52,Better, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Better, n=9,5,5,5,4 | 2 | 2 | 1 | 2 | 0
  Week 52,Slightly Better, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Slightly Better, n=9,5,5,5,4 | 0 | 0 | 1 | 1 | 1
  Week 52,No Change, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,No Change, n=9,5,5,5,4 | 1 | 0 | 0 | 0 | 0
  Week 52,Slightly Worse, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Slightly Worse, n=9,5,5,5,4 | 0 | 0 | 0 | 0 | 0
  Week 52,Worse, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Worse, n=9,5,5,5,4 | 0 | 0 | 0 | 0 | 0
  Week 52,Much Worse, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,Much Worse, n=9,5,5,5,4 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part A: Mean Patient Global Assessment of Disease Activity (PtGA) Score Over Time
Description: The Patient's Global Assessments of Disease Activity was recorded on a Visual analog scale (VAS) of 10 centimeter (cm) ranging from 0 ("very well) to 10 ("very poor").
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,39,25,26,27: number analyzed (Participants) | 42 | 39 | 25 | 26 | 27
  Baseline, n=42,39,25,26,27 | 2.96 (2.148) | 3.72 (2.649) | 4.24 (2.049) | 3.60 (2.133) | 3.64 (2.732)
  Week 2, n=38,38,25,21,27: number analyzed (Participants) | 38 | 38 | 25 | 21 | 27
  Week 2, n=38,38,25,21,27 | 2.59 (1.923) | 3.51 (2.389) | 3.73 (1.911) | 3.45 (2.247) | 3.52 (2.177)
  Week 4, n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4, n=36,37,24,22,27 | 2.43 (2.138) | 3.75 (2.770) | 3.81 (1.737) | 3.01 (1.997) | 2.62 (1.762)
  Week 8, n=34,30,24,21,23: number analyzed (Participants) | 34 | 30 | 24 | 21 | 23
  Week 8, n=34,30,24,21,23 | 1.97 (2.076) | 3.87 (2.322) | 3.44 (1.763) | 2.85 (1.769) | 2.90 (2.230)
  Week 12, n=31,28,24,22,22: number analyzed (Participants) | 31 | 28 | 24 | 22 | 22
  Week 12, n=31,28,24,22,22 | 1.97 (1.567) | 3.80 (2.557) | 3.95 (2.200) | 3.20 (2.340) | 2.75 (2.056)
  Week 16, n=27,25,22,19,19: number analyzed (Participants) | 27 | 25 | 22 | 19 | 19
  Week 16, n=27,25,22,19,19 | 1.95 (2.237) | 3.82 (2.615) | 3.39 (2.523) | 2.86 (1.809) | 2.76 (1.777)
  Week 20, n=26,23,19,18,15: number analyzed (Participants) | 26 | 23 | 19 | 18 | 15
  Week 20, n=26,23,19,18,15 | 2.60 (2.089) | 3.20 (2.663) | 4.17 (2.334) | 2.45 (1.697) | 2.90 (1.869)
  Week 24, n=23,20,15,17,16: number analyzed (Participants) | 23 | 20 | 15 | 17 | 16
  Week 24, n=23,20,15,17,16 | 2.63 (2.140) | 2.33 (1.975) | 3.83 (2.447) | 2.85 (2.256) | 3.34 (1.791)
  Week 28, n=18,17,11,13,14: number analyzed (Participants) | 18 | 17 | 11 | 13 | 14
  Week 28, n=18,17,11,13,14 | 2.44 (2.094) | 3.09 (2.915) | 4.18 (2.169) | 2.68 (2.106) | 2.74 (1.791)
  Week 32, n=19,14,9,12,12: number analyzed (Participants) | 19 | 14 | 9 | 12 | 12
  Week 32, n=19,14,9,12,12 | 2.01 (1.781) | 2.22 (2.564) | 3.02 (1.199) | 2.43 (2.385) | 2.88 (2.541)
  Week 36, n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36, n=15,13,10,12,13 | 1.46 (1.253) | 2.66 (2.982) | 2.79 (2.013) | 2.68 (2.490) | 2.62 (1.990)
  Week 40, n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40, n=15,11,9,10,10 | 2.05 (1.809) | 2.35 (2.495) | 3.20 (2.329) | 2.24 (1.883) | 3.00 (2.658)
  Week 44, n=11,11,6,8,8: number analyzed (Participants) | 11 | 11 | 6 | 8 | 8
  Week 44, n=11,11,6,8,8 | 2.28 (2.872) | 2.19 (2.429) | 2.17 (1.824) | 2.18 (1.835) | 3.49 (2.322)
  Week 48, n=9,8,5,7,5: number analyzed (Participants) | 9 | 8 | 5 | 7 | 5
  Week 48, n=9,8,5,7,5 | 1.81 (1.934) | 1.03 (1.253) | 2.30 (1.515) | 1.86 (1.586) | 4.48 (3.545)
  Week 52, n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52, n=9,5,5,5,4 | 1.10 (0.857) | 0.46 (0.358) | 2.76 (2.668) | 2.44 (1.716) | 2.13 (2.651)

18. Secondary Outcome: Part A: Mean Physician Global Assessment of Disease Activity (PhGA) Score Over Time
Description: The Physician's Global Assessments of Disease Activity was recorded on a VAS of 10 cm ranging from 0 ("none") to 10 ("extremely active").
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Scores on scale
  Baseline, n=42,39,25,26,27: number analyzed (Participants) | 42 | 39 | 25 | 26 | 27
  Baseline, n=42,39,25,26,27 | 2.33 (2.101) | 2.95 (2.208) | 2.94 (2.374) | 3.05 (2.501) | 3.25 (2.823)
  Week 2, n=36,35,25,20,26: number analyzed (Participants) | 36 | 35 | 25 | 20 | 26
  Week 2, n=36,35,25,20,26 | 1.09 (1.373) | 1.52 (1.822) | 1.83 (1.558) | 1.85 (1.879) | 1.76 (2.094)
  Week 4, n=33,32,23,21,25: number analyzed (Participants) | 33 | 32 | 23 | 21 | 25
  Week 4, n=33,32,23,21,25 | 0.81 (1.191) | 1.44 (1.904) | 1.55 (1.236) | 0.92 (1.125) | 1.02 (1.090)
  Week 8, n=33,28,23,20,21: number analyzed (Participants) | 33 | 28 | 23 | 20 | 21
  Week 8, n=33,28,23,20,21 | 1.09 (1.508) | 1.30 (1.723) | 1.35 (1.229) | 0.79 (0.798) | 1.14 (1.226)
  Week 12, n=29,25,23,18,21: number analyzed (Participants) | 29 | 25 | 23 | 18 | 21
  Week 12, n=29,25,23,18,21 | 1.08 (1.486) | 1.81 (2.183) | 1.64 (1.908) | 1.28 (1.629) | 1.47 (2.151)
  Week 16, n=26,23,21,16,19: number analyzed (Participants) | 26 | 23 | 21 | 16 | 19
  Week 16, n=26,23,21,16,19 | 0.74 (0.895) | 1.54 (1.793) | 1.87 (2.078) | 1.39 (1.830) | 0.67 (0.779)
  Week 20, n=25,23,18,17,15: number analyzed (Participants) | 25 | 23 | 18 | 17 | 15
  Week 20, n=25,23,18,17,15 | 0.71 (1.189) | 1.42 (1.808) | 1.16 (1.628) | 0.83 (0.882) | 1.27 (1.622)
  Week 24, n=20,20,15,15,15: number analyzed (Participants) | 20 | 20 | 15 | 15 | 15
  Week 24, n=20,20,15,15,15 | 0.82 (1.089) | 0.68 (0.869) | 1.50 (1.690) | 1.48 (2.003) | 1.37 (1.551)
  Week 28, n=17,17,11,12,13: number analyzed (Participants) | 17 | 17 | 11 | 12 | 13
  Week 28, n=17,17,11,12,13 | 0.76 (1.068) | 1.43 (1.986) | 1.18 (2.116) | 0.88 (0.586) | 0.85 (1.440)
  Week 32, n=19,14,8,11,12: number analyzed (Participants) | 19 | 14 | 8 | 11 | 12
  Week 32, n=19,14,8,11,12 | 0.83 (1.320) | 0.67 (0.841) | 1.40 (1.516) | 1.26 (1.546) | 0.89 (1.672)
  Week 36, n=13,11,10,11,13: number analyzed (Participants) | 13 | 11 | 10 | 11 | 13
  Week 36, n=13,11,10,11,13 | 0.48 (0.660) | 1.12 (1.589) | 0.61 (0.792) | 0.56 (0.408) | 0.75 (0.906)
  Week 40, n=13,9,8,9,10: number analyzed (Participants) | 13 | 9 | 8 | 9 | 10
  Week 40, n=13,9,8,9,10 | 0.38 (0.395) | 0.77 (1.417) | 0.36 (0.283) | 0.52 (0.531) | 0.57 (0.566)
  Week 44, n=10,9,6,8,7: number analyzed (Participants) | 10 | 9 | 6 | 8 | 7
  Week 44, n=10,9,6,8,7 | 0.31 (0.228) | 1.07 (1.574) | 0.43 (0.547) | 0.58 (0.740) | 0.87 (1.404)
  Week 48, n=7,7,5,6,5: number analyzed (Participants) | 7 | 7 | 5 | 6 | 5
  Week 48, n=7,7,5,6,5 | 0.27 (0.446) | 0.31 (0.540) | 0.30 (0.316) | 0.78 (1.482) | 1.60 (2.164)
  Week 52, n=9,5,5,4,4: number analyzed (Participants) | 9 | 5 | 5 | 4 | 4
  Week 52, n=9,5,5,4,4 | 0.31 (0.434) | 0.10 (0.141) | 0.32 (0.311) | 1.35 (0.947) | 1.80 (3.082)

19. Secondary Outcome: Part A: Change From Baseline in Serum C Reactive Protein (CRP) Over Time
Description: Blood samples were collected for analysis of CRP. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for Change from Baseline in serum CRP over time for part A was reported. The Safety set comprised of all randomized participants who received at least 1 dose of SC IP.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Safety population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Milligrams per liter
  Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Week 2,n=38,39,26,24,26 | -5.07 (6.616) | -8.81 (22.954) | -5.15 (8.436) | 1.27 (13.155) | 1.07 (6.794)
  Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Week 4,n=37,38,25,23,27 | -4.39 (6.384) | -9.01 (23.327) | -4.09 (7.169) | 4.91 (10.503) | 0.76 (5.511)
  Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Week 8,n=34,31,24,22,23 | -4.98 (6.583) | -9.94 (25.685) | -4.19 (7.197) | 10.00 (14.652) | 7.86 (25.894)
  Week 12,n=32,28,24,21,21: number analyzed (Participants) | 32 | 28 | 24 | 21 | 21
  Week 12,n=32,28,24,21,21 | -5.08 (6.690) | -9.96 (26.849) | -4.22 (7.335) | 14.81 (18.082) | 4.04 (9.339)
  Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Week 16,n=28,26,22,19,18 | -4.35 (5.648) | -10.43 (27.765) | -4.48 (7.621) | 10.53 (17.303) | 6.99 (15.503)
  Week 20,n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20,n=26,23,19,18,16 | -4.50 (5.876) | -11.67 (29.422) | -4.78 (8.100) | 5.32 (14.506) | 2.35 (7.840)
  Week 24,n=23,20,16,17,16: number analyzed (Participants) | 23 | 20 | 16 | 17 | 16
  Week 24,n=23,20,16,17,16 | -4.38 (4.640) | -13.19 (31.269) | -5.14 (8.837) | 5.07 (13.815) | 6.54 (20.711)
  Week 28,n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  Week 28,n=19,18,12,14,14 | -5.28 (6.498) | -13.42 (33.182) | -6.33 (10.022) | 1.87 (10.926) | 0.22 (11.318)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -4.85 (7.259) | -14.47 (36.343) | -7.15 (10.875) | 2.61 (9.835) | 4.37 (16.277)
  Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Week 36,n=15,12,10,12,13 | -4.72 (4.473) | -16.28 (40.531) | -7.08 (10.874) | 5.73 (19.040) | 1.64 (10.418)
  Week 40,n=15,11,8,10,10: number analyzed (Participants) | 15 | 11 | 8 | 10 | 10
  Week 40,n=15,11,8,10,10 | -4.72 (4.374) | -17.67 (42.240) | -4.69 (8.510) | 6.27 (21.164) | 2.77 (13.101)
  Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44,n=11,11,6,8,9 | -5.35 (4.523) | -17.47 (42.350) | -1.90 (1.456) | 2.80 (20.439) | 5.13 (7.292)
  Week 48,n=9,7,5,8,5: number analyzed (Participants) | 9 | 7 | 5 | 8 | 5
  Week 48,n=9,7,5,8,5 | -5.91 (4.993) | -23.39 (52.962) | -2.20 (1.562) | 6.31 (20.952) | 8.10 (18.084)
  Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,n=9,5,5,5,4 | -6.00 (4.663) | -7.26 (9.461) | -2.20 (1.575) | 0.64 (9.453) | -1.65 (4.561)

20. Secondary Outcome: Part A: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) Over Time
Description: Blood samples were collected for analysis of ESR. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for Change from Baseline in ESR over time for part A was reported.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimeters per hour
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Millimeters per hour
  Week 2,n=37,39,26,24,26: number analyzed (Participants) | 37 | 39 | 26 | 24 | 26
  Week 2,n=37,39,26,24,26 | -13.05 (9.885) | -12.78 (15.560) | -14.62 (16.500) | -1.33 (9.323) | -9.96 (20.142)
  Week 4,n=36,38,25,22,27: number analyzed (Participants) | 36 | 38 | 25 | 22 | 27
  Week 4,n=36,38,25,22,27 | -12.83 (9.346) | -17.41 (15.867) | -14.13 (12.419) | 7.59 (15.308) | -5.30 (22.250)
  Week 8,n=33,31,24,22,23: number analyzed (Participants) | 33 | 31 | 24 | 22 | 23
  Week 8,n=33,31,24,22,23 | -14.21 (9.927) | -18.76 (17.727) | -15.05 (14.030) | 6.41 (12.105) | 1.78 (27.361)
  Week 12,n=32,28,24,22,22: number analyzed (Participants) | 32 | 28 | 24 | 22 | 22
  Week 12,n=32,28,24,22,22 | -14.97 (11.361) | -17.89 (17.846) | -14.30 (13.271) | 20.36 (18.017) | -2.55 (21.498)
  Week 16,n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16,n=28,26,22,19,19 | -12.50 (10.469) | -17.17 (17.693) | -15.37 (13.956) | 14.21 (25.189) | -2.53 (20.839)
  Week 20,n=26,23,18,18,16: number analyzed (Participants) | 26 | 23 | 18 | 18 | 16
  Week 20,n=26,23,18,18,16 | -13.19 (9.600) | -17.07 (18.498) | -14.33 (15.442) | 10.00 (22.141) | -5.81 (23.063)
  Week 24,n=23,19,16,17,16: number analyzed (Participants) | 23 | 19 | 16 | 17 | 16
  Week 24,n=23,19,16,17,16 | -13.63 (11.209) | -16.84 (15.378) | -14.89 (14.504) | 7.59 (21.567) | -3.06 (22.389)
  Week 28,n=19,18,11,14,14: number analyzed (Participants) | 19 | 18 | 11 | 14 | 14
  Week 28,n=19,18,11,14,14 | -15.26 (12.274) | -19.94 (20.069) | -16.84 (16.856) | 1.50 (15.854) | -1.71 (29.148)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -13.26 (17.486) | -19.80 (19.266) | -14.52 (13.630) | -2.42 (20.129) | -2.85 (29.493)
  Week 36,n=15,12,10,12, 13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Week 36,n=15,12,10,12, 13 | -14.47 (11.673) | -21.25 (20.855) | -14.42 (13.482) | 0.67 (19.009) | 0.92 (28.324)
  Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40,n=15,11,9,10,10 | -14.40 (12.070) | -22.27 (21.873) | -11.24 (13.277) | 9.80 (28.840) | -2.60 (27.818)
  Week 44,n=11,11,6,8,8: number analyzed (Participants) | 11 | 11 | 6 | 8 | 8
  Week 44,n=11,11,6,8,8 | -12.64 (10.347) | -22.18 (21.409) | -12.00 (13.520) | 4.88 (18.256) | 2.88 (21.860)
  Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48,n=9,8,5,8,5 | -15.33 (11.822) | -25.63 (24.372) | -14.00 (14.335) | 4.50 (24.308) | 8.60 (25.205)
  Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,n=9,5,5,5,4 | -14.78 (11.692) | -24.60 (17.700) | -12.80 (15.385) | -4.60 (10.431) | 1.25 (15.042)

21. Secondary Outcome: Part A: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs) and Corticosteroid Related AEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE. Number of participants with AEs, SAEs and corticosteroid related AEs have been reported.
Time Frame: Up to 52 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Participants
  Any AE | 41 | 36 | 25 | 26 | 24
  Any SAE | 8 | 6 | 6 | 5 | 6
  Any Corticosteroid related AE | 18 | 21 | 15 | 13 | 12

22. Secondary Outcome: Part A: Change From Baseline in : Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest at indicated time points. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0), Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Safety Population Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles)..
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Millimeters of mercury
  SBP,Week 2,n=37,39,26,24,27: number analyzed (Participants) | 37 | 39 | 26 | 24 | 27
  SBP,Week 2,n=37,39,26,24,27 | -0.9 (13.11) | 3.5 (13.97) | -2.1 (17.19) | 5.7 (12.67) | -0.9 (15.63)
  SBP,Week 4,n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  SBP,Week 4,n=37,37,25,23,27 | -0.9 (15.17) | 0.2 (15.99) | -4.7 (15.00) | -2.2 (14.60) | -3.4 (14.25)
  SBP,Week 8,n=34,32,24,22,23: number analyzed (Participants) | 34 | 32 | 24 | 22 | 23
  SBP,Week 8,n=34,32,24,22,23 | 0.3 (14.33) | -3.9 (17.17) | -3.5 (15.73) | -0.8 (18.94) | -8.3 (21.05)
  SBP,Week 12,n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  SBP,Week 12,n=32,29,24,22,22 | -2.3 (15.19) | -2.4 (17.15) | -6.2 (13.45) | 1.4 (12.97) | -6.1 (19.31)
  SBP,Week 16,n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  SBP,Week 16,n=28,26,22,19,19 | -6.0 (15.39) | -5.1 (18.28) | -3.0 (20.22) | 1.9 (17.51) | -6.4 (12.73)
  SBP,Week 20,n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  SBP,Week 20,n=26,23,19,18,16 | -6.7 (10.73) | -0.7 (14.09) | -3.4 (15.39) | -1.7 (17.16) | -9.4 (21.44)
  SBP,Week 24,n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  SBP,Week 24,n=23,21,16,17,16 | -5.2 (12.65) | -2.5 (15.46) | -5.6 (16.55) | -2.6 (18.75) | -8.6 (15.65)
  SBP,Week 28,n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  SBP,Week 28,n=19,18,12,14,14 | -8.8 (12.87) | -4.2 (20.49) | -0.1 (14.76) | 6.4 (19.31) | -2.6 (17.71)
  SBP,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  SBP,Week 32,n=19,15,10,12,13 | -10.7 (13.96) | -3.7 (15.03) | -7.4 (11.80) | 3.4 (14.99) | -8.8 (14.80)
  SBP,Week 36,n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  SBP,Week 36,n=15,13,10,12,13 | -6.2 (13.92) | -8.0 (15.80) | -6.8 (12.10) | -0.6 (20.46) | -2.5 (16.13)
  SBP,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  SBP,Week 40,n=15,11,9,10,10 | -11.9 (11.75) | 0.9 (13.14) | -4.8 (14.17) | 2.1 (19.31) | -7.4 (20.14)
  SBP,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  SBP,Week 44,n=11,11,6,8,9 | -12.7 (17.66) | -4.2 (19.22) | 2.7 (13.26) | 2.9 (15.99) | 1.8 (13.91)
  SBP,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  SBP,Week 48,n=9,8,5,8,5 | -13.6 (11.85) | -0.4 (9.44) | -3.6 (28.13) | 8.8 (14.15) | 4.8 (15.51)
  SBP,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  SBP,Week 52,n=9,5,5,5,4 | -8.1 (15.85) | 1.2 (14.46) | 2.2 (19.52) | 2.2 (18.46) | -3.8 (12.34)
  DBP,Week 2,n=37,39,26,24,27: number analyzed (Participants) | 37 | 39 | 26 | 24 | 27
  DBP,Week 2,n=37,39,26,24,27 | 0.3 (7.41) | 1.2 (10.05) | -2.3 (14.00) | 2.4 (9.85) | -2.2 (9.22)
  DBP,Week 4,n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  DBP,Week 4,n=37,37,25,23,27 | 1.8 (8.85) | 1.5 (10.24) | -4.1 (13.22) | 0.1 (11.66) | -3.0 (10.22)
  DBP,Week 8,n=34,32,24,22,23: number analyzed (Participants) | 34 | 32 | 24 | 22 | 23
  DBP,Week 8,n=34,32,24,22,23 | 2.1 (8.47) | -1.3 (7.62) | -4.0 (12.26) | 2.6 (11.27) | -5.6 (11.83)
  DBP,Week 12,n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  DBP,Week 12,n=32,29,24,22,22 | 1.0 (9.60) | 2.0 (12.35) | -4.7 (12.14) | 1.3 (10.58) | -2.5 (11.16)
  DBP,Week 16,n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  DBP,Week 16,n=28,26,22,19,19 | 0.2 (7.48) | -2.5 (11.58) | -3.1 (12.80) | -1.3 (10.64) | -3.4 (7.97)
  DBP,Week 20,n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  DBP,Week 20,n=26,23,19,18,16 | -0.9 (7.66) | 1.4 (12.47) | -3.2 (16.21) | -2.0 (9.06) | -2.1 (10.98)
  DBP,Week 24,n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  DBP,Week 24,n=23,21,16,17,16 | 1.3 (8.72) | -0.6 (12.85) | -2.7 (11.77) | -3.3 (10.21) | -3.1 (9.27)
  DBP,Week 28,n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  DBP,Week 28,n=19,18,12,14,14 | -3.1 (9.39) | -2.2 (10.05) | -4.3 (15.80) | 0.1 (13.87) | -1.9 (10.37)
  DBP,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  DBP,Week 32,n=19,15,10,12,13 | -4.2 (7.50) | -2.3 (12.92) | -6.9 (25.47) | -1.2 (11.17) | -5.8 (9.09)
  DBP,Week 36,n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  DBP,Week 36,n=15,13,10,12,13 | -0.6 (8.92) | -5.1 (9.89) | -5.6 (17.02) | -1.2 (13.31) | -2.7 (13.05)
  DBP,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  DBP,Week 40,n=15,11,9,10,10 | -6.9 (12.41) | 2.6 (11.88) | -8.0 (21.60) | -2.0 (14.07) | -6.1 (11.97)
  DBP,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  DBP,Week 44,n=11,11,6,8,9 | -2.7 (12.10) | -6.5 (14.56) | -2.5 (23.89) | -1.5 (8.28) | 1.3 (11.36)
  DBP,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  DBP,Week 48,n=9,8,5,8,5 | -5.6 (11.79) | -2.3 (11.42) | -2.0 (16.00) | -3.4 (12.75) | 0.6 (8.47)
  DBP,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  DBP,Week 52,n=9,5,5,5,4 | 0.2 (12.55) | 1.8 (10.23) | 2.2 (3.35) | 1.4 (11.89) | 0.5 (5.92)

23. Secondary Outcome: Part A: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest at Baseline and up to 52 weeks. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Beats per minute
  Week 2, ,n=37,39,25,24,27: number analyzed (Participants) | 37 | 39 | 25 | 24 | 27
  Week 2, ,n=37,39,25,24,27 | -1.9 (8.07) | -2.1 (8.93) | 1.8 (10.40) | -0.4 (12.34) | -1.6 (9.79)
  Week 4,n=37,37,25,22,27: number analyzed (Participants) | 37 | 37 | 25 | 22 | 27
  Week 4,n=37,37,25,22,27 | 0.2 (8.82) | -1.4 (8.94) | -2.4 (9.42) | 2.2 (13.39) | -1.9 (10.33)
  Week 8,n=34,32,24,22,23: number analyzed (Participants) | 34 | 32 | 24 | 22 | 23
  Week 8,n=34,32,24,22,23 | -1.1 (10.23) | -3.2 (11.42) | -3.1 (8.80) | 4.3 (12.36) | 0.5 (11.06)
  Week 12,n=32,29,23,22,22: number analyzed (Participants) | 32 | 29 | 23 | 22 | 22
  Week 12,n=32,29,23,22,22 | -3.8 (8.50) | -1.2 (13.62) | -0.8 (8.35) | 4.5 (14.54) | -2.7 (10.95)
  Week 16,n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16,n=28,26,22,19,19 | -3.4 (10.79) | 0.3 (9.06) | -5.3 (10.32) | 0.3 (15.04) | -2.2 (10.76)
  Week 20,n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20,n=26,23,19,18,16 | -3.0 (9.75) | 0.2 (11.35) | -0.7 (12.62) | 1.0 (13.76) | -4.0 (12.54)
  Week 24,n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  Week 24,n=23,21,16,17,16 | -2.1 (9.29) | -3.5 (11.18) | 0.7 (14.13) | 0.1 (12.76) | 2.7 (8.27)
  Week 28,n=19,18,12,14,14: number analyzed (Participants) | 19 | 18 | 12 | 14 | 14
  Week 28,n=19,18,12,14,14 | -1.4 (10.33) | -1.2 (9.21) | -3.5 (13.26) | 0.1 (13.24) | 0.5 (10.60)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -1.3 (8.20) | -4.7 (8.50) | -2.2 (10.78) | -0.8 (16.10) | -0.6 (12.58)
  Week 36,n=15,13,10,12,13: number analyzed (Participants) | 15 | 13 | 10 | 12 | 13
  Week 36,n=15,13,10,12,13 | -5.9 (9.79) | -5.1 (9.06) | -4.5 (9.12) | -0.5 (12.22) | -3.2 (9.83)
  Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40,n=15,11,9,10,10 | -3.9 (5.64) | -3.0 (11.93) | -3.4 (10.57) | 3.3 (12.83) | -3.8 (14.09)
  Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44,n=11,11,6,8,9 | -7.1 (8.01) | -3.4 (15.86) | -8.3 (13.41) | 4.3 (15.34) | -3.4 (8.57)
  Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48,n=9,8,5,8,5 | -8.2 (7.36) | -9.3 (8.76) | -7.2 (10.47) | -1.9 (11.47) | 0.0 (16.72)
  Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,n=9,5,5,5,4 | -5.0 (12.97) | -11.0 (3.74) | -4.0 (15.89) | 6.8 (6.34) | -5.3 (12.04)

24. Secondary Outcome: Part A: Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest at Baseline and up to 52 weeks. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Celsius
  Week 2, ,n=37,39,26,24,27: number analyzed (Participants) | 37 | 39 | 26 | 24 | 27
  Week 2, ,n=37,39,26,24,27 | -0.11 (0.269) | -0.04 (0.336) | 0.03 (0.433) | -0.16 (0.421) | 0.10 (0.449)
  Week 4,n=37,37,25,23,27: number analyzed (Participants) | 37 | 37 | 25 | 23 | 27
  Week 4,n=37,37,25,23,27 | -0.12 (0.345) | 0.01 (0.407) | 0.04 (0.399) | -0.10 (0.387) | 0.11 (0.340)
  Week 8,n=34,32,23,22,23: number analyzed (Participants) | 34 | 32 | 23 | 22 | 23
  Week 8,n=34,32,23,22,23 | -0.04 (0.400) | -0.09 (0.432) | -0.07 (0.553) | 0.04 (0.579) | 0.19 (0.425)
  Week 12,n=32,29,24,22,22: number analyzed (Participants) | 32 | 29 | 24 | 22 | 22
  Week 12,n=32,29,24,22,22 | -0.08 (0.461) | -0.11 (0.367) | 0.01 (0.444) | -0.15 (0.494) | 0.09 (0.450)
  Week 16,n=28,26,22,19,19: number analyzed (Participants) | 28 | 26 | 22 | 19 | 19
  Week 16,n=28,26,22,19,19 | -0.08 (0.313) | -0.05 (0.392) | 0.04 (0.316) | -0.21 (0.664) | 0.09 (0.317)
  Week 20,n=26,23,19,18,16: number analyzed (Participants) | 26 | 23 | 19 | 18 | 16
  Week 20,n=26,23,19,18,16 | 0.03 (0.428) | -0.05 (0.483) | -0.12 (0.651) | -0.07 (0.355) | 0.05 (0.395)
  Week 24,n=23,21,16,17,16: number analyzed (Participants) | 23 | 21 | 16 | 17 | 16
  Week 24,n=23,21,16,17,16 | 0.03 (0.389) | -0.11 (0.255) | -0.11 (0.558) | -0.26 (0.476) | 0.04 (0.441)
  Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Week 28,n=19,18,12,13,14 | 0.03 (0.444) | -0.07 (0.517) | -0.09 (0.683) | -0.16 (0.479) | -0.06 (0.282)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -0.01 (0.515) | -0.07 (0.349) | 0.28 (0.418) | -0.13 (0.367) | 0.01 (0.364)
  Week 36,n=15,13,9,12,13: number analyzed (Participants) | 15 | 13 | 9 | 12 | 13
  Week 36,n=15,13,9,12,13 | -0.09 (0.406) | -0.11 (0.569) | -0.10 (0.391) | -0.09 (0.390) | -0.08 (0.367)
  Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Week 40,n=15,11,9,10,10 | 0.08 (0.426) | -0.03 (0.454) | 0.18 (0.438) | -0.05 (0.334) | -0.05 (0.306)
  Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Week 44,n=11,11,6,8,9 | -0.14 (0.347) | -0.06 (0.391) | -0.03 (0.314) | 0.00 (0.438) | -0.08 (0.396)
  Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Week 48,n=9,8,5,8,5 | -0.22 (0.233) | -0.05 (0.510) | -0.14 (0.498) | -0.01 (0.280) | -0.08 (0.559)
  Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Week 52,n=9,5,5,5,4 | -0.08 (0.291) | -0.32 (0.286) | 0.14 (0.230) | 0.02 (0.409) | -0.08 (0.814)

25. Secondary Outcome: Part A: Change From Baseline in Hematology Parameters- Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets
Description: Blood samples were collected to analyze the hematology parameters including Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets. Change from Baseline is presented for these parameters. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Giga cells per liter
  Eosinophils,Week 2,n=37,36,24,23,25: number analyzed (Participants) | 37 | 36 | 24 | 23 | 25
  Eosinophils,Week 2,n=37,36,24,23,25 | 0.019 (0.0543) | 0.001 (0.0690) | 0.010 (0.0433) | 0.015 (0.0557) | 0.062 (0.2084)
  Eosinophils,Week 4,n=36,37,24,22,26: number analyzed (Participants) | 36 | 37 | 24 | 22 | 26
  Eosinophils,Week 4,n=36,37,24,22,26 | 0.043 (0.0934) | 0.035 (0.1238) | 0.012 (0.0719) | 0.023 (0.0617) | 0.030 (0.1164)
  Eosinophils,Week 8,n=34,29,22,22,21: number analyzed (Participants) | 34 | 29 | 22 | 22 | 21
  Eosinophils,Week 8,n=34,29,22,22,21 | 0.056 (0.0959) | 0.102 (0.1634) | 0.054 (0.1036) | 0.048 (0.1498) | 0.010 (0.0591)
  Eosinophils,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Eosinophils,Week 12,n=31,28,23,22,22 | 0.077 (0.1128) | 0.155 (0.1971) | 0.090 (0.0860) | 0.090 (0.1684) | 0.030 (0.0548)
  Eosinophils,Week 16,n=27,26,20,19,19: number analyzed (Participants) | 27 | 26 | 20 | 19 | 19
  Eosinophils,Week 16,n=27,26,20,19,19 | 0.097 (0.1307) | 0.162 (0.2170) | 0.117 (0.1772) | 0.067 (0.1148) | 0.067 (0.1746)
  Eosinophils,Week 20,n=25,22,18,17,16: number analyzed (Participants) | 25 | 22 | 18 | 17 | 16
  Eosinophils,Week 20,n=25,22,18,17,16 | 0.166 (0.2073) | 0.114 (0.2085) | 0.136 (0.1518) | 0.094 (0.1743) | 0.057 (0.0637)
  Eosinophils,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Eosinophils,Week 24,n=22,21,16,16,16 | 0.210 (0.4418) | 0.109 (0.1590) | 0.109 (0.1094) | 0.089 (0.2392) | 0.051 (0.0676)
  Eosinophils,Week 28,n=18,18,11,14,13: number analyzed (Participants) | 18 | 18 | 11 | 14 | 13
  Eosinophils,Week 28,n=18,18,11,14,13 | 0.163 (0.2562) | 0.068 (0.1340) | 0.120 (0.1340) | 0.046 (0.0714) | 0.051 (0.0538)
  Eosinophils,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Eosinophils,Week 32,n=19,15,10,12,13 | 0.244 (0.3707) | 0.069 (0.1580) | 0.092 (0.1253) | 0.038 (0.0597) | 0.056 (0.0733)
  Eosinophils,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Eosinophils,Week 36,n=15,12,10,12,12 | 0.282 (0.3117) | 0.076 (0.1753) | 0.153 (0.1166) | 0.049 (0.0720) | 0.059 (0.0585)
  Eosinophils,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Eosinophils,Week 40,n=14,11,8,10,10 | 0.191 (0.2175) | 0.075 (0.1924) | 0.104 (0.1161) | 0.065 (0.0737) | 0.071 (0.1140)
  Eosinophils,Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Eosinophils,Week 44,n=11,10,6,7,9 | 0.144 (0.1952) | 0.045 (0.1329) | 0.165 (0.1564) | 0.024 (0.0541) | 0.066 (0.0600)
  Eosinophils,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Eosinophils,Week 48,n=9,8,4,8,5 | 0.091 (0.0664) | 0.059 (0.1561) | 0.233 (0.2387) | 0.028 (0.0489) | 0.030 (0.0604)
  Eosinophils,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Eosinophils,Week 52,n=8,5,5,5,4 | 0.151 (0.1865) | 0.192 (0.1839) | 0.172 (0.1207) | 0.108 (0.1139) | 0.013 (0.0802)
  Leukocytes,Week 2,n=37,38,24,24,25: number analyzed (Participants) | 37 | 38 | 24 | 24 | 25
  Leukocytes,Week 2,n=37,38,24,24,25 | -3.12 (2.268) | -3.63 (1.971) | -3.32 (2.816) | -0.76 (2.145) | 0.34 (2.238)
  Leukocytes,Week 4,n=36,37,24,22,26: number analyzed (Participants) | 36 | 37 | 24 | 22 | 26
  Leukocytes,Week 4,n=36,37,24,22,26 | -3.66 (2.621) | -4.76 (2.411) | -4.07 (2.157) | -1.64 (2.247) | -0.16 (2.330)
  Leukocytes,Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Leukocytes,Week 8,n=34,29,23,22,21 | -4.04 (2.481) | -5.65 (3.672) | -4.42 (2.469) | -1.79 (2.682) | -0.26 (1.880)
  Leukocytes,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Leukocytes,Week 12,n=31,28,23,22,22 | -4.68 (2.666) | -5.67 (2.551) | -5.23 (2.581) | -2.66 (2.883) | -1.28 (1.810)
  Leukocytes,Week 16,n=27,26,20,19,19: number analyzed (Participants) | 27 | 26 | 20 | 19 | 19
  Leukocytes,Week 16,n=27,26,20,19,19 | -5.21 (2.244) | -5.61 (3.502) | -5.36 (2.309) | -2.98 (3.018) | -0.79 (3.018)
  Leukocytes,Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Leukocytes,Week 20,n=25,23,18,18,16 | -5.24 (1.950) | -5.20 (3.104) | -5.40 (2.414) | -3.24 (3.592) | -1.71 (2.840)
  Leukocytes,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Leukocytes,Week 24,n=22,21,16,16,16 | -5.14 (3.559) | -6.39 (2.952) | -5.01 (1.884) | -2.89 (3.892) | -1.52 (2.738)
  Leukocytes,Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Leukocytes,Week 28,n=18,18,12,14,13 | -5.46 (2.619) | -6.04 (3.274) | -4.58 (2.143) | -3.01 (3.368) | -1.97 (3.461)
  Leukocytes,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Leukocytes,Week 32,n=19,15,10,12,13 | -5.71 (2.419) | -5.61 (3.250) | -5.27 (1.696) | -3.43 (3.342) | -2.33 (3.011)
  Leukocytes,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Leukocytes,Week 36,n=15,12,10,12,12 | -5.76 (2.106) | -6.82 (2.814) | -5.58 (1.757) | -3.36 (3.612) | -2.95 (3.635)
  Leukocytes,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Leukocytes,Week 40,n=14,11,8,10,10 | -6.14 (1.987) | -7.10 (2.534) | -6.46 (2.130) | -3.18 (3.662) | -2.23 (3.142)
  Leukocytes,Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Leukocytes,Week 44,n=11,10,6,7,9 | -6.25 (2.300) | -6.95 (2.441) | -6.17 (1.726) | -2.83 (3.875) | -3.08 (3.056)
  Leukocytes,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Leukocytes,Week 48,n=9,8,4,8,5 | -6.88 (2.436) | -7.35 (2.853) | -6.48 (2.887) | -2.69 (2.979) | -3.00 (3.045)
  Leukocytes,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Leukocytes,Week 52,n=8,5,5,5,4 | -6.66 (2.654) | -7.36 (2.920) | -6.38 (2.262) | -3.84 (3.467) | -3.10 (4.090)
  Lymphocytes,Week 2,n=37,36,24,23,25: number analyzed (Participants) | 37 | 36 | 24 | 23 | 25
  Lymphocytes,Week 2,n=37,36,24,23,25 | 0.015 (1.1645) | 0.002 (1.2620) | -0.041 (1.3241) | -0.159 (0.9064) | -0.209 (0.9381)
  Lymphocytes,Week 4,n=36,37,24,22,26: number analyzed (Participants) | 36 | 37 | 24 | 22 | 26
  Lymphocytes,Week 4,n=36,37,24,22,26 | 0.027 (1.2460) | -0.255 (1.2225) | 0.057 (1.2338) | -0.002 (0.7340) | -0.382 (1.0808)
  Lymphocytes,Week 8,n=34,29,22,22,21: number analyzed (Participants) | 34 | 29 | 22 | 22 | 21
  Lymphocytes,Week 8,n=34,29,22,22,21 | -0.191 (1.3361) | -0.411 (1.2086) | -0.067 (1.2814) | -0.049 (1.0832) | -0.516 (0.8562)
  Lymphocytes,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Lymphocytes,Week 12,n=31,28,23,22,22 | -0.215 (1.3052) | -0.437 (1.2479) | -0.081 (1.2018) | -0.128 (1.0505) | -0.344 (0.7846)
  Lymphocytes,Week 16,n=27,26,20,19,19: number analyzed (Participants) | 27 | 26 | 20 | 19 | 19
  Lymphocytes,Week 16,n=27,26,20,19,19 | -0.450 (1.3450) | -0.704 (1.2994) | -0.153 (0.7804) | -0.327 (1.4269) | -0.635 (0.8037)
  Lymphocytes,Week 20,n=25,22,18,17,16: number analyzed (Participants) | 25 | 22 | 18 | 17 | 16
  Lymphocytes,Week 20,n=25,22,18,17,16 | -0.616 (1.2793) | -0.313 (1.3011) | -0.439 (1.4363) | -0.385 (0.8819) | -0.533 (0.7432)
  Lymphocytes,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Lymphocytes,Week 24,n=22,21,16,16,16 | -0.399 (1.4276) | -0.179 (1.8386) | -0.073 (0.7890) | -0.401 (1.2030) | -0.386 (0.7504)
  Lymphocytes,Week 28,n=18,18,11,14,13: number analyzed (Participants) | 18 | 18 | 11 | 14 | 13
  Lymphocytes,Week 28,n=18,18,11,14,13 | -0.614 (1.5450) | -0.273 (1.3296) | -0.192 (0.7271) | -0.258 (1.0211) | -0.565 (1.0397)
  Lymphocytes,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Lymphocytes,Week 32,n=19,15,10,12,13 | -0.602 (1.3438) | -0.407 (1.4002) | -0.476 (0.7997) | -0.402 (1.2625) | -0.492 (0.7877)
  Lymphocytes,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Lymphocytes,Week 36,n=15,12,10,12,12 | -0.625 (1.5738) | -0.672 (1.2263) | -0.430 (0.7690) | -0.417 (1.0538) | -0.078 (0.7182)
  Lymphocytes,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Lymphocytes,Week 40,n=14,11,8,10,10 | -0.929 (1.5351) | -0.845 (1.3603) | -0.570 (0.8261) | -0.519 (1.1491) | -0.681 (0.7363)
  Lymphocytes,Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Lymphocytes,Week 44,n=11,10,6,7,9 | -0.915 (1.2235) | -1.047 (1.3375) | -0.198 (0.9783) | -1.029 (1.0293) | -0.343 (0.8113)
  Lymphocytes,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Lymphocytes,Week 48,n=9,8,4,8,5 | -1.258 (1.2063) | -0.923 (1.4811) | 0.118 (1.0588) | -0.576 (1.1994) | -0.510 (1.1450)
  Lymphocytes,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Lymphocytes,Week 52,n=8,5,5,5,4 | -1.253 (1.2857) | -0.754 (1.0291) | -0.286 (1.0455) | 0.194 (0.8800) | -0.128 (1.2618)
  Neutrophils,Week 2,n=37,36,24,23,25: number analyzed (Participants) | 37 | 36 | 24 | 23 | 25
  Neutrophils,Week 2,n=37,36,24,23,25 | -3.208 (2.5761) | -3.454 (2.2265) | -3.367 (2.5781) | -0.748 (2.2688) | 0.387 (2.6156)
  Neutrophils,Week 4,n=36,37,24,22,26: number analyzed (Participants) | 36 | 37 | 24 | 22 | 26
  Neutrophils,Week 4,n=36,37,24,22,26 | -3.791 (2.5242) | -4.476 (2.3632) | -4.106 (2.4354) | -1.673 (1.9745) | 0.089 (3.1611)
  Neutrophils,Week 8,n=34,29,22,22,21: number analyzed (Participants) | 34 | 29 | 22 | 22 | 21
  Neutrophils,Week 8,n=34,29,22,22,21 | -3.949 (2.5477) | -5.271 (3.2214) | -4.354 (2.4128) | -1.869 (3.2525) | 0.192 (2.2180)
  Neutrophils,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Neutrophils,Week 12,n=31,28,23,22,22 | -4.590 (2.6603) | -5.340 (2.6437) | -5.250 (2.1872) | -2.678 (3.1106) | -1.019 (2.1306)
  Neutrophils,Week 16,n=27,26,20,19,19: number analyzed (Participants) | 27 | 26 | 20 | 19 | 19
  Neutrophils,Week 16,n=27,26,20,19,19 | -4.933 (2.4430) | -4.929 (3.7907) | -5.358 (2.2367) | -2.766 (3.3212) | -0.263 (3.3610)
  Neutrophils,Week 20,n=25,22,18,17,16: number analyzed (Participants) | 25 | 22 | 18 | 17 | 16
  Neutrophils,Week 20,n=25,22,18,17,16 | -4.867 (2.3110) | -4.997 (3.0763) | -5.168 (2.4898) | -2.856 (4.0311) | -1.355 (3.3883)
  Neutrophils,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Neutrophils,Week 24,n=22,21,16,16,16 | -4.985 (3.5051) | -6.257 (2.7551) | -5.030 (1.9579) | -2.570 (4.2089) | -1.342 (3.1038)
  Neutrophils,Week 28,n=18,18,11,14,13: number analyzed (Participants) | 18 | 18 | 11 | 14 | 13
  Neutrophils,Week 28,n=18,18,11,14,13 | -5.076 (2.3415) | -5.729 (3.1699) | -4.469 (2.1333) | -2.764 (3.5787) | -1.503 (4.3502)
  Neutrophils,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Neutrophils,Week 32,n=19,15,10,12,13 | -5.357 (2.5525) | -5.153 (3.1939) | -4.840 (1.9387) | -3.006 (3.7915) | -2.018 (3.5674)
  Neutrophils,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Neutrophils,Week 36,n=15,12,10,12,12 | -5.444 (2.1894) | -6.079 (3.0406) | -5.265 (1.8375) | -3.023 (3.9443) | -3.018 (4.1223)
  Neutrophils,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Neutrophils,Week 40,n=14,11,8,10,10 | -5.416 (2.4371) | -6.179 (2.8859) | -5.916 (1.7172) | -2.705 (3.4469) | -1.663 (3.4090)
  Neutrophils,Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Neutrophils,Week 44,n=11,10,6,7,9 | -5.432 (2.5555) | -5.799 (3.1785) | -6.185 (1.3944) | -1.807 (4.5472) | -2.883 (3.8690)
  Neutrophils,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Neutrophils,Week 48,n=9,8,4,8,5 | -5.628 (2.3471) | -6.396 (3.4832) | -6.790 (1.6060) | -2.160 (3.3843) | -2.650 (4.0017)
  Neutrophils,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Neutrophils,Week 52,n=8,5,5,5,4 | -5.520 (2.7316) | -6.774 (2.6817) | -6.256 (1.8929) | -4.214 (3.6948) | -2.990 (4.8629)
  Platelets,Week 2,n=37,38,24,23,25: number analyzed (Participants) | 37 | 38 | 24 | 23 | 25
  Platelets,Week 2,n=37,38,24,23,25 | -39.0 (39.46) | -49.2 (52.77) | -41.1 (40.29) | -1.9 (37.57) | -4.3 (49.32)
  Platelets,Week 4,n=36,37,24,22,26: number analyzed (Participants) | 36 | 37 | 24 | 22 | 26
  Platelets,Week 4,n=36,37,24,22,26 | -45.9 (41.70) | -64.3 (56.21) | -49.0 (35.74) | 2.1 (41.23) | -5.7 (43.51)
  Platelets,Week 8,n=34,29,22,22,21: number analyzed (Participants) | 34 | 29 | 22 | 22 | 21
  Platelets,Week 8,n=34,29,22,22,21 | -37.3 (31.22) | -72.2 (75.77) | -53.3 (37.10) | 14.2 (45.62) | 15.7 (57.21)
  Platelets,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Platelets,Week 12,n=31,28,23,22,22 | -51.2 (33.25) | -74.0 (52.17) | -55.4 (38.89) | 17.8 (50.58) | 4.3 (55.14)
  Platelets,Week 16,n=27,26,20,19,19: number analyzed (Participants) | 27 | 26 | 20 | 19 | 19
  Platelets,Week 16,n=27,26,20,19,19 | -53.8 (33.54) | -69.9 (53.79) | -54.8 (39.71) | 12.4 (52.98) | 13.8 (60.11)
  Platelets,Week 20,n=25,22,18,17,16: number analyzed (Participants) | 25 | 22 | 18 | 17 | 16
  Platelets,Week 20,n=25,22,18,17,16 | -52.2 (54.64) | -69.5 (58.27) | -53.5 (38.00) | 14.8 (44.55) | -0.1 (56.21)
  Platelets,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Platelets,Week 24,n=22,21,16,16,16 | -58.0 (39.58) | -72.4 (64.56) | -57.5 (44.46) | 6.3 (46.94) | 20.1 (45.30)
  Platelets,Week 28,n=18,18,11,14,13: number analyzed (Participants) | 18 | 18 | 11 | 14 | 13
  Platelets,Week 28,n=18,18,11,14,13 | -70.2 (45.09) | -61.3 (54.34) | -50.6 (27.71) | 15.4 (31.84) | 13.1 (47.56)
  Platelets,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Platelets,Week 32,n=19,15,10,12,13 | -57.6 (66.52) | -65.5 (51.20) | -50.8 (33.70) | -1.5 (45.26) | 10.7 (53.95)
  Platelets,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Platelets,Week 36,n=15,12,10,12,12 | -74.1 (32.84) | -70.6 (58.49) | -48.6 (23.64) | 13.4 (32.69) | 20.0 (85.28)
  Platelets,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Platelets,Week 40,n=14,11,8,10,10 | -77.4 (41.72) | -66.9 (62.21) | -42.0 (21.33) | 5.6 (45.38) | 5.3 (54.71)
  Platelets,Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Platelets,Week 44,n=11,10,6,7,9 | -69.5 (36.62) | -76.7 (64.91) | -58.2 (19.28) | 11.1 (48.18) | -3.3 (56.78)
  Platelets,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Platelets,Week 48,n=9,8,4,8,5 | -68.3 (41.94) | -71.4 (57.71) | -80.8 (22.98) | 14.4 (53.59) | 0.4 (61.59)
  Platelets,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Platelets,Week 52,n=8,5,5,5,4 | -81.9 (38.36) | -51.6 (43.90) | -58.6 (40.79) | -18.6 (55.44) | -17.5 (38.04)

26. Secondary Outcome: Part A: Change From Baseline in Hematology Parameters- Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin
Description: Blood samples were collected to analyze the hematology parameters including MCHC and Hemoglobin. Change from Baseline is presented for these parameters. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Grams per liter
  MCHC,Week 2,n=32,33,18,22,23: number analyzed (Participants) | 32 | 33 | 18 | 22 | 23
  MCHC,Week 2,n=32,33,18,22,23 | -0.5 (6.21) | 0.1 (9.47) | 1.9 (5.11) | -1.1 (6.56) | 1.2 (8.41)
  MCHC,Week 4,n=31,31,19,20,25: number analyzed (Participants) | 31 | 31 | 19 | 20 | 25
  MCHC,Week 4,n=31,31,19,20,25 | 1.6 (7.36) | 2.3 (11.94) | 2.6 (9.46) | 0.1 (5.17) | 2.4 (9.32)
  MCHC,Week 8,n=28,24,18,20,20: number analyzed (Participants) | 28 | 24 | 18 | 20 | 20
  MCHC,Week 8,n=28,24,18,20,20 | 6.1 (8.97) | 6.7 (10.98) | 6.4 (9.09) | 0.6 (9.53) | 6.7 (8.19)
  MCHC,Week 12,n=25,23,18,20,20: number analyzed (Participants) | 25 | 23 | 18 | 20 | 20
  MCHC,Week 12,n=25,23,18,20,20 | 6.5 (9.77) | 6.7 (9.03) | 5.9 (14.20) | 1.3 (9.55) | 4.9 (7.81)
  MCHC,Week 16,n=22,21,17,17,17: number analyzed (Participants) | 22 | 21 | 17 | 17 | 17
  MCHC,Week 16,n=22,21,17,17,17 | 8.3 (9.80) | 8.9 (12.41) | 10.2 (8.50) | 0.9 (11.52) | 4.5 (9.62)
  MCHC,Week 20,n=19,18,14,16,14: number analyzed (Participants) | 19 | 18 | 14 | 16 | 14
  MCHC,Week 20,n=19,18,14,16,14 | 7.7 (8.43) | 10.8 (9.53) | 9.0 (8.60) | 3.4 (10.38) | 4.6 (12.48)
  MCHC,Week 24,n=16,16,13,15,14: number analyzed (Participants) | 16 | 16 | 13 | 15 | 14
  MCHC,Week 24,n=16,16,13,15,14 | 4.7 (7.50) | 14.6 (11.04) | 4.9 (9.97) | 3.0 (7.46) | 4.9 (11.49)
  MCHC,Week 28,n=13,14,10,12,11: number analyzed (Participants) | 13 | 14 | 10 | 12 | 11
  MCHC,Week 28,n=13,14,10,12,11 | 4.5 (7.78) | 9.2 (11.52) | 8.9 (11.41) | 2.8 (13.57) | -0.4 (7.86)
  MCHC,Week 32,n=13,11,8,10,11: number analyzed (Participants) | 13 | 11 | 8 | 10 | 11
  MCHC,Week 32,n=13,11,8,10,11 | 6.9 (9.33) | 8.4 (10.45) | 8.8 (9.05) | 6.7 (8.88) | 1.4 (8.58)
  MCHC,Week 36,n=10,10,8,10,10: number analyzed (Participants) | 10 | 10 | 8 | 10 | 10
  MCHC,Week 36,n=10,10,8,10,10 | 6.9 (5.11) | 6.7 (9.72) | 13.5 (8.07) | 7.9 (11.44) | 4.2 (5.90)
  MCHC,Week 40,n=10,9,7,8,9: number analyzed (Participants) | 10 | 9 | 7 | 8 | 9
  MCHC,Week 40,n=10,9,7,8,9 | 11.5 (9.89) | 11.3 (7.75) | 14.4 (12.45) | 5.1 (15.30) | 13.9 (12.39)
  MCHC,Week 44,n=8,8,4,5,8: number analyzed (Participants) | 8 | 8 | 4 | 5 | 8
  MCHC,Week 44,n=8,8,4,5,8 | 12.5 (7.17) | 9.9 (9.86) | 13.5 (4.12) | 5.2 (4.60) | 12.1 (10.99)
  MCHC,Week 48,n=6,7,2,6,4: number analyzed (Participants) | 6 | 7 | 2 | 6 | 4
  MCHC,Week 48,n=6,7,2,6,4 | 13.3 (9.07) | 11.9 (9.84) | 10.5 (13.44) | 3.8 (11.48) | 9.3 (9.32)
  MCHC,Week 52,n=6,4,3,4,3: number analyzed (Participants) | 6 | 4 | 3 | 4 | 3
  MCHC,Week 52,n=6,4,3,4,3 | 16.5 (5.47) | 18.8 (5.68) | 24.0 (3.46) | 11.3 (5.06) | 5.0 (9.85)
  Hemoglobin,Week 2,n=38,39,24,24,25: number analyzed (Participants) | 38 | 39 | 24 | 24 | 25
  Hemoglobin,Week 2,n=38,39,24,24,25 | 1.2 (6.50) | 2.5 (6.85) | 1.3 (8.72) | -2.4 (7.08) | -0.9 (5.44)
  Hemoglobin,Week 4,n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Hemoglobin,Week 4,n=36,37,24,22,27 | 3.0 (6.37) | 2.8 (8.17) | 2.5 (6.55) | -1.0 (8.45) | -2.1 (6.86)
  Hemoglobin,Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Hemoglobin,Week 8,n=34,29,23,22,21 | 5.9 (9.57) | 4.7 (9.59) | 3.1 (7.00) | -1.4 (10.54) | -2.8 (7.41)
  Hemoglobin,Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Hemoglobin,Week 12,n=31,28,23,22,22 | 5.8 (7.85) | 8.4 (10.62) | 4.7 (6.24) | -3.2 (11.11) | -1.4 (7.10)
  Hemoglobin,Week 16,n=27,26,21,19,19: number analyzed (Participants) | 27 | 26 | 21 | 19 | 19
  Hemoglobin,Week 16,n=27,26,21,19,19 | 2.6 (6.00) | 5.8 (8.87) | 4.2 (7.03) | -3.8 (10.55) | -1.7 (7.47)
  Hemoglobin,Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Hemoglobin,Week 20,n=25,23,18,18,16 | 2.0 (7.89) | 7.4 (9.69) | 3.3 (5.58) | -4.6 (11.32) | -0.6 (6.22)
  Hemoglobin,Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Hemoglobin,Week 24,n=22,21,16,16,16 | 2.2 (8.67) | 7.0 (9.99) | 5.4 (6.38) | -3.1 (12.05) | -0.9 (6.43)
  Hemoglobin,Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Hemoglobin,Week 28,n=18,18,12,14,13 | 0.3 (9.68) | 5.8 (11.83) | 2.8 (6.92) | -4.4 (11.45) | -1.5 (8.88)
  Hemoglobin,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Hemoglobin,Week 32,n=19,15,10,12,13 | 0.9 (9.04) | 5.1 (10.88) | 2.0 (9.42) | -3.0 (10.05) | 0.8 (9.64)
  Hemoglobin,Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Hemoglobin,Week 36,n=15,12,10,12,12 | 4.4 (7.97) | 4.8 (11.91) | 4.0 (7.26) | -2.6 (10.93) | 1.3 (9.68)
  Hemoglobin,Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Hemoglobin,Week 40,n=14,11,8,10,10 | 1.3 (8.03) | 3.8 (12.40) | 6.3 (5.47) | -3.4 (11.24) | -0.4 (7.86)
  Hemoglobin,Week 44,n=11,10,6,8,9: number analyzed (Participants) | 11 | 10 | 6 | 8 | 9
  Hemoglobin,Week 44,n=11,10,6,8,9 | 0.0 (8.00) | 6.7 (14.60) | 2.3 (7.84) | -0.3 (11.70) | 2.8 (12.85)
  Hemoglobin,Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Hemoglobin,Week 48,n=9,8,4,8,5 | 2.4 (7.57) | 4.8 (12.62) | 2.8 (12.69) | -4.6 (14.66) | 7.6 (15.57)
  Hemoglobin,Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Hemoglobin,Week 52,n=8,5,5,5,4 | 2.9 (5.33) | 8.6 (12.84) | 10.4 (13.28) | 4.4 (6.47) | 2.8 (13.57)

27. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter-Hematocrit
Description: Blood samples were collected to analyze the hematology parameter Hematocrit. Change from Baseline is presented for this parameter. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Proportion of red blood cells in blood
  Week 2,n=38,39,24,24,25: number analyzed (Participants) | 38 | 39 | 24 | 24 | 25
  Week 2,n=38,39,24,24,25 | 0.0040 (0.01988) | 0.0060 (0.02186) | 0.0008 (0.02909) | -0.0063 (0.02491) | -0.0030 (0.01813)
  Week 4,n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4,n=36,37,24,22,27 | 0.0059 (0.01903) | 0.0048 (0.02635) | 0.0040 (0.01531) | -0.0035 (0.02676) | -0.0087 (0.02004)
  Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Week 8,n=34,29,23,22,21 | 0.0101 (0.02601) | 0.0054 (0.03213) | 0.0019 (0.02110) | -0.0054 (0.03286) | -0.0159 (0.01918)
  Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Week 12,n=31,28,23,22,22 | 0.0087 (0.02386) | 0.0148 (0.03272) | 0.0059 (0.01970) | -0.0118 (0.03281) | -0.0095 (0.02108)
  Week 16,n=27,26,21,19,19: number analyzed (Participants) | 27 | 26 | 21 | 19 | 19
  Week 16,n=27,26,21,19,19 | -0.0037 (0.02187) | 0.0049 (0.02833) | 0.0008 (0.01961) | -0.0135 (0.02976) | -0.0095 (0.02347)
  Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Week 20,n=25,23,18,18,16 | -0.0063 (0.02436) | 0.0066 (0.03019) | -0.0015 (0.01398) | -0.0184 (0.02972) | -0.0062 (0.02076)
  Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Week 24,n=22,21,16,16,16 | -0.0017 (0.02882) | 0.0010 (0.02839) | 0.0089 (0.01973) | -0.0133 (0.03478) | -0.0077 (0.01599)
  Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Week 28,n=18,18,12,14,13 | -0.0089 (0.02917) | 0.0039 (0.03455) | -0.0046 (0.01858) | -0.0186 (0.02814) | -0.0035 (0.02785)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -0.0076 (0.02782) | 0.0027 (0.02994) | -0.0060 (0.03161) | -0.0176 (0.02473) | 0.0025 (0.02741)
  Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Week 36,n=15,12,10,12,12 | 0.0012 (0.02603) | 0.0036 (0.03232) | -0.0054 (0.01811) | -0.0198 (0.02570) | 0.0018 (0.03090)
  Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Week 40,n=14,11,8,10,10 | -0.0115 (0.03075) | -0.0052 (0.03398) | -0.0009 (0.01086) | -0.0193 (0.02157) | -0.0160 (0.02099)
  Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Week 44,n=11,10,6,7,9 | -0.0185 (0.03039) | 0.0054 (0.03463) | -0.0097 (0.02548) | -0.0126 (0.03225) | -0.0037 (0.03048)
  Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Week 48,n=9,8,4,8,5 | -0.0136 (0.02709) | -0.0025 (0.03217) | -0.0053 (0.04366) | -0.0216 (0.03428) | 0.0144 (0.04123)
  Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Week 52,n=8,5,5,5,4 | -0.0135 (0.02112) | 0.0016 (0.04082) | 0.0058 (0.04370) | -0.0006 (0.01558) | 0.0025 (0.03288)

28. Secondary Outcome: Part A: Change From Baseline in Hematology Parameter -Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes Mean Corpuscular Volume. Change from Baseline is presented for this parameter. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Femtoliter
  Week 2,n=38,39,24,24,25: number analyzed (Participants) | 38 | 39 | 24 | 24 | 25
  Week 2,n=38,39,24,24,25 | 0.5 (1.35) | 0.5 (1.64) | 0.5 (1.38) | 0.6 (1.38) | 0.4 (1.44)
  Week 4,n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4,n=36,37,24,22,27 | 0.9 (1.95) | 1.1 (2.15) | 1.0 (1.69) | 0.6 (1.68) | 0.6 (2.28)
  Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Week 8,n=34,29,23,22,21 | 1.2 (2.54) | 1.8 (3.27) | 1.9 (2.72) | 1.7 (2.34) | -0.2 (2.91)
  Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Week 12,n=31,28,23,22,22 | 0.8 (3.41) | 2.0 (4.29) | 2.6 (3.14) | 0.9 (3.16) | 0.3 (4.07)
  Week 16,n=27,26,21,19,19: number analyzed (Participants) | 27 | 26 | 21 | 19 | 19
  Week 16,n=27,26,21,19,19 | 1.0 (4.14) | 2.2 (4.36) | 3.1 (3.37) | 0.4 (4.03) | -0.3 (4.98)
  Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Week 20,n=25,23,18,18,16 | 1.2 (4.42) | 1.8 (4.35) | 2.1 (3.12) | -0.5 (4.72) | 0.1 (3.54)
  Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Week 24,n=22,21,16,16,16 | 1.1 (4.20) | 1.1 (3.91) | 2.6 (3.36) | -1.0 (4.44) | -1.6 (4.84)
  Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Week 28,n=18,18,12,14,13 | 0.6 (4.02) | 1.4 (4.19) | 2.0 (2.26) | -0.4 (4.43) | -0.5 (3.95)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | 0.9 (4.42) | 2.0 (4.44) | 1.3 (3.13) | 0.3 (4.89) | -0.5 (3.64)
  Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Week 36,n=15,12,10,12,12 | 1.8 (3.49) | 1.6 (4.76) | 0.9 (2.47) | -0.5 (4.93) | -0.2 (2.55)
  Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Week 40,n=14,11,8,10,10 | 0.6 (3.73) | 1.8 (5.25) | 2.0 (2.83) | 0.4 (4.95) | -2.1 (3.00)
  Week 44,n=11,10,6,8,9: number analyzed (Participants) | 11 | 10 | 6 | 8 | 9
  Week 44,n=11,10,6,8,9 | -0.5 (3.50) | 2.5 (5.08) | 1.7 (3.50) | -0.7 (6.87) | -0.7 (2.83)
  Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Week 48,n=9,8,4,8,5 | -0.4 (3.50) | 3.3 (4.95) | 2.3 (4.50) | -1.1 (6.92) | 2.0 (2.12)
  Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Week 52,n=8,5,5,5,4 | -0.6 (3.02) | 3.2 (5.12) | 1.4 (4.16) | 3.2 (5.72) | 1.0 (2.58)

29. Secondary Outcome: Part A:Change From Baseline in Hematology Parameter-Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes Mean Corpuscular Hemoglobin. Change from Baseline is presented for this parameter. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Picograms
  Week 2,n=38,39,24,24,25: number analyzed (Participants) | 38 | 39 | 24 | 24 | 25
  Week 2,n=38,39,24,24,25 | 0.13 (0.571) | 0.29 (0.730) | 0.42 (0.512) | 0.12 (0.494) | 0.22 (0.678)
  Week 4,n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4,n=36,37,24,22,27 | 0.53 (0.786) | 0.58 (0.877) | 0.55 (0.672) | 0.25 (0.458) | 0.36 (0.892)
  Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Week 8,n=34,29,23,22,21 | 0.96 (1.041) | 1.20 (1.056) | 1.16 (1.178) | 0.60 (0.751) | 0.49 (1.022)
  Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Week 12,n=31,28,23,22,22 | 0.94 (1.341) | 1.43 (1.372) | 1.38 (1.630) | 0.44 (1.110) | 0.47 (1.480)
  Week 16,n=27,26,21,19,19: number analyzed (Participants) | 27 | 26 | 21 | 19 | 19
  Week 16,n=27,26,21,19,19 | 1.16 (1.345) | 1.59 (1.617) | 1.83 (1.424) | 0.24 (1.508) | 0.22 (1.927)
  Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Week 20,n=25,23,18,18,16 | 1.24 (1.529) | 1.69 (1.605) | 1.48 (1.256) | 0.14 (1.666) | 0.39 (1.696)
  Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Week 24,n=22,21,16,16,16 | 0.97 (1.491) | 1.80 (1.663) | 1.34 (1.230) | -0.04 (1.727) | -0.08 (2.041)
  Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Week 28,n=18,18,12,14,13 | 0.91 (1.659) | 1.48 (1.618) | 1.47 (1.409) | 0.21 (2.000) | -0.20 (1.493)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | 1.01 (1.498) | 1.57 (1.694) | 1.27 (1.111) | 0.68 (2.103) | -0.14 (1.413)
  Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Week 36,n=15,12,10,12,12 | 1.42 (0.944) | 1.29 (1.905) | 1.39 (1.005) | 0.68 (2.327) | 0.15 (0.971)
  Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Week 40,n=14,11,8,10,10 | 1.30 (0.818) | 1.75 (1.914) | 1.91 (1.373) | 0.71 (2.617) | 0.44 (1.492)
  Week 44,n=11,10,6,8,9: number analyzed (Participants) | 11 | 10 | 6 | 8 | 9
  Week 44,n=11,10,6,8,9 | 1.16 (0.727) | 1.83 (2.214) | 1.63 (1.178) | 0.30 (2.460) | 0.77 (1.261)
  Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Week 48,n=9,8,4,8,5 | 1.36 (0.633) | 2.25 (2.194) | 1.73 (1.389) | 0.14 (2.934) | 1.32 (1.119)
  Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Week 52,n=8,5,5,5,4 | 1.44 (0.950) | 2.70 (1.744) | 2.24 (1.484) | 1.84 (1.889) | 0.80 (1.068)

30. Secondary Outcome: Part A:Change From Baseline in Hematology Parameter- Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes. Change from Baseline is presented for this parameter. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: trillion cells per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
trillion cells per liter
  Week 2,n=38,39,24,24,25: number analyzed (Participants) | 38 | 39 | 24 | 24 | 25
  Week 2,n=38,39,24,24,25 | 0.01 (0.232) | 0.02 (0.265) | -0.01 (0.303) | -0.10 (0.254) | -0.07 (0.221)
  Week 4,n=36,37,24,22,27: number analyzed (Participants) | 36 | 37 | 24 | 22 | 27
  Week 4,n=36,37,24,22,27 | 0.01 (0.208) | -0.01 (0.311) | -0.01 (0.202) | -0.09 (0.268) | -0.14 (0.248)
  Week 8,n=34,29,23,22,21: number analyzed (Participants) | 34 | 29 | 23 | 22 | 21
  Week 8,n=34,29,23,22,21 | 0.04 (0.249) | -0.04 (0.406) | -0.08 (0.300) | -0.16 (0.372) | -0.17 (0.219)
  Week 12,n=31,28,23,22,22: number analyzed (Participants) | 31 | 28 | 23 | 22 | 22
  Week 12,n=31,28,23,22,22 | 0.03 (0.255) | 0.05 (0.417) | -0.07 (0.265) | -0.20 (0.379) | -0.11 (0.237)
  Week 16,n=27,26,21,19,19: number analyzed (Participants) | 27 | 26 | 21 | 19 | 19
  Week 16,n=27,26,21,19,19 | -0.09 (0.238) | -0.07 (0.312) | -0.14 (0.282) | -0.19 (0.399) | -0.11 (0.303)
  Week 20,n=25,23,18,18,16: number analyzed (Participants) | 25 | 23 | 18 | 18 | 16
  Week 20,n=25,23,18,18,16 | -0.13 (0.263) | -0.03 (0.305) | -0.12 (0.183) | -0.20 (0.461) | -0.08 (0.286)
  Week 24,n=22,21,16,16,16: number analyzed (Participants) | 22 | 21 | 16 | 16 | 16
  Week 24,n=22,21,16,16,16 | -0.09 (0.270) | -0.06 (0.282) | -0.04 (0.234) | -0.11 (0.464) | -0.01 (0.289)
  Week 28,n=18,18,12,14,13: number analyzed (Participants) | 18 | 18 | 12 | 14 | 13
  Week 28,n=18,18,12,14,13 | -0.14 (0.295) | -0.04 (0.327) | -0.16 (0.231) | -0.18 (0.377) | -0.02 (0.387)
  Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Week 32,n=19,15,10,12,13 | -0.13 (0.292) | -0.09 (0.259) | -0.13 (0.330) | -0.22 (0.321) | 0.04 (0.362)
  Week 36,n=15,12,10,12,12: number analyzed (Participants) | 15 | 12 | 10 | 12 | 12
  Week 36,n=15,12,10,12,12 | -0.08 (0.262) | -0.04 (0.378) | -0.10 (0.183) | -0.21 (0.358) | 0.03 (0.391)
  Week 40,n=14,11,8,10,10: number analyzed (Participants) | 14 | 11 | 8 | 10 | 10
  Week 40,n=14,11,8,10,10 | -0.16 (0.234) | -0.16 (0.380) | -0.09 (0.189) | -0.22 (0.301) | -0.10 (0.330)
  Week 44,n=11,10,6,7,9: number analyzed (Participants) | 11 | 10 | 6 | 7 | 9
  Week 44,n=11,10,6,7,9 | -0.18 (0.286) | -0.10 (0.333) | -0.17 (0.320) | -0.10 (0.216) | -0.03 (0.367)
  Week 48,n=9,8,4,8,5: number analyzed (Participants) | 9 | 8 | 4 | 8 | 5
  Week 48,n=9,8,4,8,5 | -0.14 (0.240) | -0.23 (0.266) | -0.18 (0.457) | -0.20 (0.251) | 0.04 (0.434)
  Week 52,n=8,5,5,5,4: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4
  Week 52,n=8,5,5,5,4 | -0.16 (0.283) | -0.18 (0.370) | -0.02 (0.531) | -0.18 (0.192) | -0.05 (0.332)

31. Secondary Outcome: Part A: Change From Baseline in Clinical Chemistry Parameters- Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea
Description: Blood samples were collected to analyze the chemistry parameters including Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea . Change from Baseline is presented for these parameters. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4 ,8,12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Millimoles per liter
  calcium,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  calcium,Week 2,n=38,39,26,24,26 | 0.002 (0.1056) | 0.006 (0.0853) | -0.008 (0.0817) | 0.008 (0.1050) | 0.013 (0.0812)
  calcium,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  calcium,Week 4,n=37,38,25,23,27 | 0.009 (0.0974) | 0.008 (0.0968) | 0.013 (0.0649) | -0.016 (0.0922) | -0.001 (0.0899)
  calcium,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  calcium,Week 8,n=34,31,24,22,23 | 0.032 (0.1114) | 0.049 (0.0879) | 0.005 (0.0764) | 0.020 (0.0918) | 0.013 (0.0615)
  calcium,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  calcium,Week 12,n=32,28,24,22,21 | 0.019 (0.1200) | 0.072 (0.0789) | -0.001 (0.0750) | 0.011 (0.0913) | 0.016 (0.0851)
  calcium,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  calcium,Week 16,n=28,26,22,19,18 | 0.009 (0.0974) | 0.050 (0.0808) | 0.018 (0.0954) | -0.008 (0.0707) | 0.044 (0.0768)
  calcium,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  calcium,Week 20,n=25,23,19,18,16 | 0.018 (0.1080) | 0.070 (0.0987) | 0.032 (0.0933) | 0.000 (0.0884) | 0.012 (0.0932)
  calcium,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  calcium,Week 24,n=22,21,16,17,16 | 0.008 (0.1029) | 0.064 (0.0927) | 0.032 (0.1077) | -0.002 (0.0748) | 0.009 (0.0702)
  calcium,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  calcium,Week 28,n=19,18,12,13,14 | 0.006 (0.1102) | 0.066 (0.1106) | 0.054 (0.1232) | 0.018 (0.0838) | 0.076 (0.1108)
  calcium,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  calcium,Week 32,n=19,15,10,12,13 | 0.029 (0.1119) | 0.044 (0.0923) | 0.059 (0.0737) | -0.008 (0.0978) | 0.075 (0.1271)
  calcium,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  calcium,Week 36,n=15,12,10,12,13 | 0.016 (0.0789) | 0.055 (0.0773) | 0.075 (0.0738) | -0.038 (0.1025) | 0.053 (0.0957)
  calcium,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  calcium,Week 40,n=15,11,9,10,10 | 0.077 (0.1012) | 0.016 (0.0662) | 0.008 (0.0930) | -0.042 (0.0561) | 0.037 (0.0589)
  calcium,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  calcium,Week 44,n=11,11,6,8,9 | 0.042 (0.1480) | 0.025 (0.0908) | -0.002 (0.0475) | -0.035 (0.1638) | 0.054 (0.1146)
  calcium,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  calcium,Week 48,n=9,8,5,8,5 | -0.007 (0.1126) | 0.028 (0.0956) | -0.018 (0.0769) | -0.035 (0.0769) | 0.142 (0.0782)
  calcium,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  calcium,Week 52,n=9,5,5,5,4 | 0.013 (0.0907) | 0.076 (0.1108) | 0.026 (0.0747) | -0.056 (0.1161) | 0.083 (0.0624)
  Carbon Dioxide,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Carbon Dioxide,Week 2,n=38,39,26,24,26 | 0.7 (2.42) | 0.6 (2.55) | 0.5 (2.53) | -0.3 (2.31) | 0.7 (2.24)
  Carbon Dioxide,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Carbon Dioxide,Week 4,n=37,38,25,23,27 | 0.1 (2.03) | 0.2 (2.68) | 0.4 (2.69) | 0.2 (1.75) | 0.1 (2.83)
  Carbon Dioxide,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Carbon Dioxide,Week 8,n=34,31,24,22,23 | 0.1 (3.39) | 0.3 (2.89) | 0.0 (2.69) | 0.0 (2.01) | 1.1 (2.24)
  Carbon Dioxide,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Carbon Dioxide,Week 12,n=32,28,24,22,21 | 0.1 (2.66) | 0.6 (2.53) | -0.4 (2.28) | 0.0 (1.94) | 1.2 (1.73)
  Carbon Dioxide,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Carbon Dioxide,Week 16,n=28,26,22,19,18 | 0.1 (2.97) | 0.5 (2.47) | 0.8 (2.94) | -0.1 (1.88) | 0.5 (2.55)
  Carbon Dioxide,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Carbon Dioxide,Week 20,n=25,23,19,18,16 | 0.1 (2.98) | -0.1 (3.17) | -0.1 (2.70) | -0.3 (2.83) | 0.5 (2.68)
  Carbon Dioxide,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Carbon Dioxide,Week 24,n=22,21,16,17,16 | 0.4 (3.10) | 0.4 (3.11) | -0.8 (2.65) | 0.5 (2.29) | -0.2 (2.61)
  Carbon Dioxide,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Carbon Dioxide,Week 28,n=19,18,12,13,14 | -1.6 (2.83) | 0.4 (3.63) | -1.0 (2.04) | -0.4 (2.36) | 0.4 (3.08)
  Carbon Dioxide,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Carbon Dioxide,Week 32,n=19,15,10,12,13 | -1.0 (3.65) | 0.8 (2.08) | -1.4 (2.17) | -0.6 (2.43) | 0.2 (2.24)
  Carbon Dioxide,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Carbon Dioxide,Week 36,n=15,12,10,12,13 | -1.1 (2.28) | 0.3 (3.72) | -0.9 (1.97) | -0.3 (3.63) | 1.0 (2.16)
  Carbon Dioxide,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Carbon Dioxide,Week 40,n=15,11,6,10,10 | -1.5 (3.16) | 0.9 (3.75) | -1.7 (2.35) | -0.8 (2.70) | 0.4 (1.43)
  Carbon Dioxide,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Carbon Dioxide,Week 44,n=11,11,6,8,9 | -1.7 (2.72) | 1.6 (3.50) | 0.0 (3.03) | -1.6 (1.60) | -0.1 (2.47)
  Carbon Dioxide,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Carbon Dioxide,Week 48,n=9,8,5,8,5 | -2.6 (2.70) | 0.5 (3.59) | -1.0 (2.65) | 0.0 (1.77) | -0.2 (2.17)
  Carbon Dioxide,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Carbon Dioxide,Week 52,n=9,5,5,5,4 | -1.1 (1.76) | 1.2 (2.68) | -1.2 (1.48) | -0.4 (1.34) | 1.8 (2.87)
  Chloride,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Chloride,Week 2,n=38,39,26,24,26 | 1.1 (2.36) | 0.6 (1.79) | 0.7 (1.76) | 1.0 (2.16) | 0.8 (2.77)
  Chloride,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Chloride,Week 4,n=37,38,25,23,27 | 1.8 (2.34) | 1.6 (2.10) | 1.4 (1.87) | 0.7 (2.14) | 1.4 (2.79)
  Chloride,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Chloride,Week 8,n=34,31,24,22,23 | 2.5 (2.12) | 2.4 (2.06) | 2.0 (2.65) | 1.0 (2.18) | 2.1 (3.24)
  Chloride,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Chloride,Week 12,n=32,28,24,22,21 | 2.9 (2.54) | 1.8 (3.03) | 2.4 (2.30) | 0.6 (2.06) | 2.0 (2.36)
  Chloride,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Chloride,Week 16,n=28,26,22,19,18 | 3.0 (2.27) | 2.3 (2.54) | 2.2 (2.46) | 1.1 (2.04) | 2.4 (3.40)
  Chloride,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Chloride,Week 20,n=25,23,19,18,16 | 3.3 (2.88) | 2.0 (2.11) | 2.1 (2.49) | 1.3 (2.22) | 2.5 (3.12)
  Chloride,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Chloride,Week 24,n=22,21,16,17,16 | 3.4 (3.42) | 2.7 (2.51) | 1.6 (3.16) | 1.0 (2.12) | 2.3 (3.55)
  Chloride,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Chloride,Week 28,n=19,18,12,13,14 | 3.9 (3.13) | 2.8 (2.80) | 2.8 (2.49) | 0.2 (3.49) | 2.9 (3.63)
  Chloride,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Chloride,Week 32,n=19,15,10,12,13 | 3.4 (2.73) | 1.9 (2.59) | 2.0 (2.26) | -0.1 (4.17) | 3.4 (3.43)
  Chloride,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Chloride,Week 36,n=15,12,10,12,13 | 3.8 (1.74) | 2.4 (2.78) | 1.9 (2.47) | 1.1 (1.88) | 2.8 (3.37)
  Chloride,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Chloride,Week 40,n=15,11,9,10,10 | 3.3 (2.49) | 3.6 (1.12) | 1.4 (1.94) | 1.9 (1.45) | 3.9 (3.03)
  Chloride,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Chloride,Week 44,n=11,11,6,8,9 | 3.8 (2.23) | 3.4 (1.91) | 0.2 (2.14) | 1.1 (2.03) | 2.2 (4.52)
  Chloride,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Chloride,Week 48,n=9,8,5,8,5 | 4.6 (1.88) | 2.1 (2.23) | 2.0 (1.58) | 1.8 (1.58) | 2.8 (3.11)
  Chloride,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Chloride,Week 52,n=9,5,5,5,4 | 4.8 (1.09) | 2.2 (1.64) | 0.2 (3.83) | 3.6 (1.95) | 3.8 (4.11)
  Glucose,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Glucose,Week 2,n=38,39,26,24,26 | -0.03 (2.568) | -0.46 (1.671) | 0.01 (1.237) | 0.29 (1.358) | -0.44 (3.578)
  Glucose,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Glucose,Week 4,n=37,38,25,23,27 | -0.10 (2.676) | -0.35 (1.929) | 0.38 (1.601) | 0.31 (1.466) | -0.03 (4.387)
  Glucose,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Glucose,Week 8,n=34,31,24,22,23 | -0.29 (2.507) | -0.58 (2.606) | -0.12 (1.265) | 0.10 (1.579) | -1.15 (5.685)
  Glucose,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Glucose,Week 12,n=32,28,24,22,21 | -0.64 (2.219) | -0.63 (2.134) | -0.33 (1.163) | -0.25 (1.164) | -1.76 (5.919)
  Glucose,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Glucose,Week 16,n=28,26,22,19,18 | -0.71 (2.485) | 0.33 (1.941) | -0.29 (1.113) | -0.12 (1.414) | -1.15 (6.411)
  Glucose,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Glucose,Week 20,n=25,23,19,18,16 | -0.66 (2.701) | -0.46 (1.550) | 0.46 (1.714) | -0.33 (1.435) | -1.96 (7.018)
  Glucose,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Glucose,Week 24,n=22,21,16,17,16 | -0.72 (2.701) | -0.44 (1.632) | -0.23 (1.217) | -0.38 (1.290) | -2.08 (6.953)
  Glucose,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Glucose,Week 28,n=19,18,12,13,14 | -0.91 (2.990) | -0.32 (1.510) | 0.58 (1.627) | -0.25 (1.278) | -2.05 (7.699)
  Glucose,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Glucose,Week 32,n=19,15,10,12,13 | -0.74 (3.492) | -0.48 (1.533) | 0.72 (1.795) | -0.05 (1.363) | -3.12 (7.818)
  Glucose,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Glucose,Week 36,n=15,12,10,12,13 | -1.14 (3.268) | -0.35 (1.861) | 0.05 (1.019) | -0.50 (1.261) | -2.98 (7.786)
  Glucose,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Glucose,Week 40,n=15,11,9,10,10 | -0.99 (3.465) | -0.33 (2.376) | 0.22 (1.203) | -0.22 (1.192) | -0.94 (3.589)
  Glucose,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Glucose,Week 44,n=11,11,6,8,9 | -1.39 (3.789) | -0.05 (1.954) | -0.27 (0.940) | 0.30 (0.739) | -0.23 (2.001)
  Glucose,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Glucose,Week 48,n=9,8,5,8,5 | -1.39 (4.249) | -0.93 (2.077) | -0.62 (1.441) | -0.88 (1.369) | -0.36 (2.196)
  Glucose,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Glucose,Week 52,n=9,5,5,5,4 | -1.51 (4.466) | -0.94 (2.707) | -0.26 (1.316) | -0.72 (1.308) | 0.45 (2.353)
  Phosphate,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Phosphate,Week 2,n=38,39,26,24,26 | 0.056 (0.2249) | -0.004 (0.1930) | 0.017 (0.1886) | -0.025 (0.1622) | 0.005 (0.1601)
  Phosphate,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Phosphate,Week 4,n=37,38,25,23,27 | 0.071 (0.1944) | -0.011 (0.2501) | 0.093 (0.1848) | 0.006 (0.1883) | 0.008 (0.2087)
  Phosphate,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Phosphate,Week 8,n=34,31,24,22,23 | 0.088 (0.1786) | 0.091 (0.2098) | 0.112 (0.1588) | 0.045 (0.1971) | 0.055 (0.1746)
  Phosphate,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Phosphate,Week 12,n=32,28,24,22,21 | 0.122 (0.2404) | 0.154 (0.2377) | 0.190 (0.1725) | 0.067 (0.1873) | 0.079 (0.1946)
  Phosphate,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Phosphate,Week 16,n=28,26,22,19,18 | 0.113 (0.1976) | 0.139 (0.2315) | 0.146 (0.1612) | 0.025 (0.1589) | 0.039 (0.2238)
  Phosphate,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Phosphate,Week 20,n=25,23,19,18,16 | 0.070 (0.1860) | 0.160 (0.2436) | 0.141 (0.2257) | 0.043 (0.1854) | 0.060 (0.2183)
  Phosphate,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Phosphate,Week 24,n=22,21,16,17,16 | 0.132 (0.2066) | 0.163 (0.2383) | 0.181 (0.1778) | 0.055 (0.1728) | 0.101 (0.1811)
  Phosphate,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Phosphate,Week 28,n=19,18,12,13,14 | 0.156 (0.1873) | 0.090 (0.2543) | 0.191 (0.1980) | 0.073 (0.2017) | 0.190 (0.3143)
  Phosphate,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Phosphate,Week 32,n=19,15,10,12,13 | 0.164 (0.1166) | 0.101 (0.2160) | 0.214 (0.2086) | 0.048 (0.1677) | 0.155 (0.2713)
  Phosphate,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Phosphate,Week 36,n=15,12,10,12,13 | 0.111 (0.1786) | 0.068 (0.2204) | 0.304 (0.2112) | 0.098 (0.1939) | 0.151 (0.2114)
  Phosphate,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Phosphate,Week 40,n=15,11,6,10,10 | 0.221 (0.1902) | -0.007 (0.2007) | 0.104 (0.1948) | 0.073 (0.1849) | 0.206 (0.2151)
  Phosphate,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Phosphate,Week 44,n=11,11,6,8,9 | 0.142 (0.2117) | 0.025 (0.1874) | 0.090 (0.2131) | -0.065 (0.2267) | 0.218 (0.2184)
  Phosphate,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Phosphate,Week 48,n=9,8,5,8,5 | 0.029 (0.2136) | -0.054 (0.2203) | 0.028 (0.2611) | -0.015 (0.1561) | 0.132 (0.1972)
  Phosphate,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Phosphate,Week 52,n=9,5,5,5,4 | 0.049 (0.2235) | -0.036 (0.2779) | 0.208 (0.1583) | 0.036 (0.0865) | 0.115 (0.1434)
  Potassium,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Potassium,Week 2,n=38,39,26,24,26 | 0.03 (0.372) | -0.03 (0.437) | -0.02 (0.401) | 0.18 (0.336) | 0.08 (0.375)
  Potassium,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Potassium,Week 4,n=37,38,25,23,27 | -0.13 (0.319) | -0.04 (0.412) | -0.10 (0.453) | 0.06 (0.329) | -0.03 (0.343)
  Potassium,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Potassium,Week 8,n=34,31,24,22,23 | 0.01 (0.364) | 0.05 (0.437) | -0.11 (0.422) | 0.10 (0.333) | 0.06 (0.399)
  Potassium,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Potassium,Week 12,n=32,28,24,22,21 | -0.12 (0.333) | 0.15 (0.810) | -0.10 (0.346) | 0.06 (0.336) | 0.04 (0.446)
  Potassium,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Potassium,Week 16,n=28,26,22,19,18 | 0.01 (0.376) | 0.03 (0.439) | -0.02 (0.358) | 0.15 (0.345) | 0.15 (0.279)
  Potassium,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Potassium,Week 20,n=25,23,19,18,16 | 0.04 (0.394) | 0.07 (0.556) | 0.02 (0.417) | 0.10 (0.287) | 0.16 (0.390)
  Potassium,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Potassium,Week 24,n=22,21,16,17,16 | 0.05 (0.447) | -0.01 (0.403) | -0.13 (0.368) | 0.15 (0.371) | 0.16 (0.411)
  Potassium,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Potassium,Week 28,n=19,18,12,13,14 | 0.12 (0.288) | 0.07 (0.470) | 0.17 (0.414) | 0.08 (0.297) | 0.23 (0.418)
  Potassium,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Potassium,Week 32,n=19,15,10,12,13 | 0.16 (0.437) | 0.01 (0.448) | 0.17 (0.333) | 0.19 (0.365) | 0.25 (0.443)
  Potassium,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Potassium,Week 36,n=15,12,10,12,13 | 0.16 (0.429) | -0.07 (0.475) | 0.18 (0.408) | 0.18 (0.341) | 0.21 (0.403)
  Potassium,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Potassium,Week 40,n=15,11,9,10,10 | 0.24 (0.534) | -0.03 (0.476) | 0.01 (0.276) | 0.03 (0.450) | 0.28 (0.355)
  Potassium,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Potassium,Week 44,n=11,11,6,8,9 | 0.16 (0.287) | -0.13 (0.478) | -0.13 (0.288) | 0.15 (0.385) | 0.16 (0.488)
  Potassium,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Potassium,Week 48,n=9,8,5,8,5 | 0.21 (0.352) | 0.06 (0.644) | -0.04 (0.182) | 0.16 (0.283) | 0.52 (0.432)
  Potassium,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Potassium,Week 52,n=9,5,5,5,4 | 0.22 (0.186) | -0.16 (0.434) | -0.10 (0.418) | 0.06 (0.445) | 0.20 (0.365)
  Sodium,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Sodium,Week 2,n=38,39,26,24,26 | 0.3 (2.11) | 0.0 (2.33) | -0.8 (2.37) | -0.2 (1.52) | 0.9 (2.92)
  Sodium,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Sodium,Week 4,n=37,38,25,23,27 | 0.7 (2.15) | 0.4 (2.11) | 0.2 (2.29) | 0.0 (1.43) | 0.6 (2.65)
  Sodium,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Sodium,Week 8,n=34,31,24,22,23 | 1.1 (2.10) | 0.9 (3.12) | 0.1 (2.32) | 0.5 (1.50) | 1.7 (2.91)
  Sodium,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Sodium,Week 12,n=32,28,24,22,21 | 1.8 (2.46) | 0.5 (3.90) | 0.6 (1.76) | 0.5 (1.79) | 2.1 (2.37)
  Sodium,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Sodium,Week 16,n=28,26,22,19,18 | 1.0 (2.28) | 0.6 (3.09) | -0.2 (2.25) | -0.3 (1.37) | 2.3 (3.59)
  Sodium,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Sodium,Week 20,n=25,23,19,18,16 | 1.0 (2.23) | 0.6 (2.79) | -0.3 (2.60) | -0.6 (0.92) | 2.3 (3.52)
  Sodium,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Sodium,Week 24,n=22,21,16,17,16 | 0.9 (2.31) | 1.0 (1.83) | -0.4 (2.00) | 0.4 (1.50) | 1.9 (2.96)
  Sodium,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Sodium,Week 28,n=19,18,12,13,14 | 0.9 (2.27) | 1.2 (2.75) | 0.5 (1.93) | -0.8 (3.22) | 2.4 (3.54)
  Sodium,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Sodium,Week 32,n=19,15,10,12,13 | 0.7 (2.31) | -0.3 (2.63) | -0.2 (2.04) | -0.8 (3.16) | 3.2 (4.13)
  Sodium,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Sodium,Week 36,n=15,12,10,12,13 | 0.5 (1.96) | 0.6 (2.43) | -0.4 (2.07) | -0.2 (1.85) | 2.8 (3.60)
  Sodium,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Sodium,Week 40,n=15,11,9,10,10 | 0.1 (2.17) | 1.2 (2.23) | -1.2 (2.49) | 0.5 (1.58) | 2.9 (3.07)
  Sodium,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Sodium,Week 44,n=11,11,6,8,9 | 0.5 (1.97) | 0.4 (2.58) | -2.0 (2.53) | -0.8 (1.28) | 1.8 (3.77)
  Sodium,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Sodium,Week 48,n=9,8,5,8,5 | -0.3 (1.87) | 0.8 (2.76) | -0.6 (2.07) | 0.3 (1.91) | 1.6 (2.70)
  Sodium,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Sodium,Week 52,n=9,5,5,5,4 | 0.7 (1.66) | 0.4 (2.51) | -0.8 (3.11) | 1.6 (1.14) | 3.5 (3.32)
  Urea,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Urea,Week 2,n=38,39,26,24,26 | 0.05 (1.210) | -0.16 (1.776) | 0.28 (1.439) | -0.31 (1.458) | -0.32 (1.240)
  Urea,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Urea,Week 4,n=37,38,25,23,27 | -0.09 (1.592) | -0.61 (1.514) | -0.06 (1.277) | -0.22 (1.022) | -0.27 (1.700)
  Urea,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Urea,Week 8,n=34,31,24,22,23 | -0.36 (1.938) | -0.99 (1.826) | -0.40 (1.574) | -0.91 (0.970) | -0.34 (0.965)
  Urea,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Urea,Week 12,n=32,28,24,22,21 | -0.65 (1.617) | -1.20 (1.778) | -0.62 (1.501) | -1.12 (1.457) | -0.35 (1.316)
  Urea,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Urea,Week 16,n=28,26,22,19,18 | -0.56 (2.009) | -0.52 (1.612) | -0.72 (1.232) | -0.40 (1.580) | -0.07 (1.701)
  Urea,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Urea,Week 20,n=25,23,19,18,16 | -0.30 (1.675) | -0.70 (1.379) | -0.70 (1.197) | -0.31 (1.470) | -0.77 (1.900)
  Urea,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Urea,Week 24,n=22,21,16,17,16 | -0.48 (1.901) | -0.22 (2.044) | -0.80 (1.717) | -0.65 (1.457) | -0.64 (2.019)
  Urea,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Urea,Week 28,n=19,18,12,13,14 | -0.45 (1.745) | -0.42 (1.510) | -0.73 (1.317) | 0.23 (1.111) | -0.31 (1.495)
  Urea,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Urea,Week 32,n=19,15,10,12,13 | -0.16 (2.086) | -0.64 (1.479) | -0.83 (1.382) | -0.76 (1.071) | 0.17 (2.609)
  Urea,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Urea,Week 36,n=15,12,10,12,13 | 0.06 (1.967) | -1.43 (1.828) | -0.93 (1.113) | -0.01 (0.973) | -0.22 (2.297)
  Urea,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Urea,Week 40,n=15,11,9,10,10 | -0.17 (1.775) | -0.78 (0.603) | -0.98 (1.237) | -0.76 (1.552) | 0.32 (1.886)
  Urea,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Urea,Week 44,n=11,11,6,8,9 | -0.46 (3.119) | -1.05 (1.234) | -0.63 (1.359) | -0.76 (1.274) | -1.09 (1.727)
  Urea,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Urea,Week 48,n=9,8,5,8,5 | -0.18 (3.535) | -1.58 (1.450) | -0.06 (1.311) | -0.51 (1.225) | 0.44 (1.282)
  Urea,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Urea,Week 52,n=9,5,5,5,4 | -0.26 (2.508) | -1.22 (1.671) | -0.76 (1.647) | -0.82 (0.782) | -0.45 (1.475)

32. Secondary Outcome: Part A: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected to analyze the chemistry parameters including Albumin and Protein. Change from Baseline is presented for these parameters. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Grams per liter
  Albumin,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Albumin,Week 2,n=38,39,26,24,26 | 0.3 (2.29) | 0.9 (1.79) | 0.8 (1.88) | -0.9 (2.64) | -0.7 (2.24)
  Albumin,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Albumin,Week 4,n=37,38,25,23,27 | 0.9 (2.41) | 2.0 (2.84) | 1.6 (1.50) | -1.4 (2.46) | -0.9 (2.46)
  Albumin,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Albumin,Week 8,n=34,31,24,22,23 | 1.9 (2.76) | 3.1 (2.35) | 2.1 (1.85) | -1.1 (2.35) | -0.6 (1.80)
  Albumin,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Albumin,Week 12,n=32,28,24,22,21 | 2.0 (2.26) | 3.4 (2.50) | 3.1 (1.54) | -0.5 (2.81) | 0.2 (1.87)
  Albumin,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Albumin,Week 16,n=28,26,22,19,18 | 1.7 (2.29) | 2.8 (2.52) | 2.8 (2.44) | -1.2 (2.41) | 0.6 (2.48)
  Albumin,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Albumin,Week 20,n=25,23,19,18,16 | 1.8 (2.46) | 3.9 (2.68) | 2.8 (2.15) | -0.9 (2.70) | 0.3 (2.11)
  Albumin,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Albumin,Week 24,n=22,21,16,17,16 | 1.6 (2.77) | 3.8 (2.36) | 3.7 (1.85) | 0.0 (2.83) | 0.3 (1.88)
  Albumin,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Albumin,Week 28,n=19,18,12,13,14 | 1.5 (1.61) | 3.5 (3.38) | 2.4 (2.78) | -0.5 (2.82) | 0.4 (2.98)
  Albumin,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Albumin,Week 32,n=19,15,10,12,13 | 2.2 (2.03) | 3.6 (3.68) | 2.2 (2.66) | -0.7 (3.20) | 1.1 (2.93)
  Albumin,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Albumin,Week 36,n=15,12,10,12,13 | 3.1 (2.61) | 4.3 (3.75) | 2.9 (2.08) | -1.3 (3.25) | 0.2 (3.02)
  Albumin,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Albumin,Week 40,n=15,11,9,10,10 | 3.2 (1.97) | 3.9 (3.78) | 2.4 (2.07) | -1.1 (2.96) | -0.5 (2.27)
  Albumin,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Albumin,Week 44,n=11,11,6,8,9 | 3.2 (2.36) | 4.1 (3.36) | 2.2 (2.23) | 0.4 (3.07) | 0.6 (2.19)
  Albumin,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Albumin,Week 48,n=9,8,5,8,5 | 3.4 (2.13) | 4.4 (3.20) | 1.6 (2.70) | -0.8 (3.28) | 2.0 (2.92)
  Albumin,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Albumin,Week 52,n=9,5,5,5,4 | 3.7 (2.45) | 5.2 (1.64) | 4.0 (2.55) | -1.2 (0.84) | 1.5 (4.12)
  Protein,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Protein,Week 2,n=38,39,26,24,26 | -2.6 (3.68) | -2.4 (3.13) | -1.9 (2.73) | -1.7 (3.31) | -1.7 (3.16)
  Protein,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Protein,Week 4,n=37,38,25,23,27 | -2.5 (3.49) | -2.4 (4.39) | -1.8 (2.81) | -2.0 (3.64) | -2.0 (4.05)
  Protein,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Protein,Week 8,n=34,31,24,22,23 | -1.9 (3.53) | -1.6 (4.16) | -2.2 (3.67) | -0.7 (3.10) | -0.7 (3.30)
  Protein,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Protein,Week 12,n=32,28,24,22,21 | -1.7 (3.19) | -1.3 (3.72) | -0.8 (3.06) | 1.0 (3.68) | 0.9 (3.67)
  Protein,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Protein,Week 16,n=28,26,22,19,18 | -2.3 (3.43) | -2.0 (3.67) | -1.9 (3.70) | 0.2 (3.20) | 1.0 (3.68)
  Protein,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Protein,Week 20,n=25,23,19,18,16 | -1.9 (3.44) | -0.4 (4.69) | -1.3 (2.84) | 0.6 (3.45) | 0.4 (2.63)
  Protein,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Protein,Week 24,n=22,21,16,17,16 | -1.1 (3.64) | -0.9 (4.39) | 0.0 (2.85) | 1.5 (4.86) | 0.8 (3.09)
  Protein,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Protein,Week 28,n=19,18,12,13,14 | -2.4 (3.30) | -0.8 (5.27) | -2.7 (2.67) | -0.2 (4.39) | 1.6 (4.20)
  Protein,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Protein,Week 32,n=19,15,10,12,13 | -1.4 (3.52) | -1.5 (4.67) | -2.1 (4.07) | -0.3 (4.45) | 2.6 (3.78)
  Protein,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Protein,Week 36,n=15,12,10,12,13 | -0.3 (3.48) | -0.8 (4.69) | -0.5 (2.51) | -0.3 (4.11) | 1.8 (3.51)
  Protein,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  Protein,Week 40,n=15,11,9,10,10 | -0.5 (3.38) | -1.5 (4.93) | -2.1 (1.76) | -0.4 (3.27) | 1.4 (3.03)
  Protein,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Protein,Week 44,n=11,11,6,8,9 | 0.3 (2.65) | -0.4 (4.06) | -2.0 (3.52) | 2.3 (5.50) | 1.7 (2.60)
  Protein,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Protein,Week 48,n=9,8,5,8,5 | 0.3 (4.69) | -0.1 (3.76) | -1.8 (4.49) | 1.4 (4.98) | 3.2 (2.28)
  Protein,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Protein,Week 52,n=9,5,5,5,4 | -0.4 (3.54) | 1.0 (4.69) | 0.6 (4.88) | -1.0 (3.54) | 1.8 (4.43)

33. Secondary Outcome: Part A: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the chemistry parameters including ALT,ALP and AST. Change from Baseline is presented for these parameters. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
International units per liter
  ALT,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  ALT,Week 2,n=38,39,26,24,26 | 8.2 (17.71) | 5.3 (14.63) | 10.1 (23.12) | -0.6 (3.27) | 1.8 (15.16)
  ALT,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  ALT,Week 4,n=37,38,25,23,27 | 6.6 (11.17) | 6.6 (16.09) | 5.2 (6.10) | -1.2 (4.20) | -3.1 (9.80)
  ALT,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  ALT,Week 8,n=34,31,24,22,23 | 6.0 (14.70) | 9.5 (12.71) | 4.7 (8.25) | -2.8 (4.19) | -6.8 (12.81)
  ALT,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  ALT,Week 12,n=32,28,24,22,21 | 4.7 (6.91) | 4.4 (10.82) | 4.0 (6.85) | -3.3 (5.39) | -7.0 (11.88)
  ALT,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  ALT,Week 16,n=28,26,22,19,18 | 4.1 (8.11) | 2.2 (9.86) | 5.2 (10.08) | -3.5 (5.23) | -6.6 (14.22)
  ALT,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  ALT,Week 20,n=25,23,19,18,16 | 16.1 (51.67) | 4.9 (15.83) | 8.6 (11.73) | 2.3 (22.33) | -8.1 (14.38)
  ALT,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  ALT,Week 24,n=22,21,16,17,16 | 8.3 (13.62) | 2.5 (14.71) | 16.4 (33.68) | -2.8 (6.58) | -9.4 (13.61)
  ALT,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  ALT,Week 28,n=19,18,12,13,14 | 6.7 (8.75) | 2.9 (14.59) | 12.1 (23.96) | -1.9 (3.95) | -8.9 (12.65)
  ALT,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  ALT,Week 32,n=19,15,10,12,13 | 6.6 (11.06) | 5.0 (14.05) | 5.1 (9.45) | -2.0 (4.45) | -10.0 (12.40)
  ALT,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  ALT,Week 36,n=15,12,10,12,13 | 8.7 (13.58) | 6.0 (15.22) | 4.5 (8.44) | -2.8 (2.77) | -10.0 (13.87)
  ALT,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  ALT,Week 40,n=15,11,9,10,10 | 5.3 (8.85) | 7.3 (19.52) | 5.4 (5.61) | 0.1 (11.82) | -2.1 (6.77)
  ALT,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  ALT,Week 44,n=11,11,6,8,9 | 1.8 (5.51) | 5.5 (15.53) | 2.7 (7.09) | -0.4 (7.15) | -7.0 (4.42)
  ALT,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  ALT,Week 48,n=9,8,5,8,5 | 2.3 (6.54) | 4.5 (16.52) | 3.6 (10.48) | -3.5 (3.12) | 0.2 (11.50)
  ALT,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  ALT,Week 52,n=9,5,5,5,4 | 1.3 (5.98) | 1.6 (19.63) | 8.8 (10.03) | -4.4 (1.52) | 5.3 (20.81)
  ALP,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  ALP,Week 2,n=38,39,26,24,26 | -9.3 (15.76) | -11.4 (7.46) | -11.4 (8.50) | -3.0 (5.88) | -2.6 (5.81)
  ALP,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  ALP,Week 4,n=37,38,25,23,27 | -15.5 (13.96) | -13.4 (12.75) | -14.2 (10.17) | -2.2 (8.83) | 5.3 (27.51)
  ALP,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  ALP,Week 8,n=34,31,24,22,23 | -16.8 (11.61) | -10.4 (13.73) | -15.3 (7.14) | 2.9 (9.95) | 1.6 (33.37)
  ALP,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  ALP,Week 12,n=32,28,24,22,21 | -19.2 (15.60) | -7.0 (10.15) | -15.0 (8.06) | 6.6 (13.21) | -5.3 (16.83)
  ALP,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  ALP,Week 16,n=28,26,22,19,18 | -18.2 (15.36) | -8.0 (12.61) | -14.6 (8.56) | 1.1 (12.90) | -0.3 (14.43)
  ALP,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  ALP,Week 20,n=25,23,19,18,16 | -14.4 (21.82) | -4.4 (12.89) | -13.3 (9.58) | 5.9 (19.44) | -1.0 (12.41)
  ALP,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  ALP,Week 24,n=22,21,16,17,16 | -16.3 (20.32) | -6.2 (13.76) | -12.5 (9.08) | 6.9 (16.34) | -1.8 (20.27)
  ALP,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  ALP,Week 28,n=19,18,12,13,14 | -17.6 (23.06) | -4.3 (14.99) | -17.5 (6.56) | 1.6 (13.28) | 2.9 (19.72)
  ALP,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  ALP,Week 32,n=19,15,10,12,13 | -15.9 (22.94) | -6.1 (11.89) | -12.6 (6.93) | -2.3 (17.00) | 5.2 (18.44)
  ALP,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  ALP,Week 36,n=15,12,10,12,13 | -20.3 (24.22) | -7.3 (11.18) | -9.6 (12.51) | -1.8 (15.49) | 7.3 (20.95)
  ALP,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  ALP,Week 40,n=15,11,9,10,10 | -14.5 (22.71) | -7.4 (10.16) | -9.9 (11.35) | -0.2 (15.17) | 12.3 (24.69)
  ALP,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  ALP,Week 44,n=11,11,6,8,9 | -19.4 (24.30) | -6.2 (13.48) | -4.0 (10.86) | 2.8 (19.93) | 11.9 (24.93)
  ALP,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  ALP,Week 48,n=9,8,5,8,5 | -24.4 (28.77) | -6.5 (8.45) | -4.4 (12.82) | 1.5 (18.31) | 7.2 (17.06)
  ALP,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  ALP,Week 52,n=9,5,5,5,4 | -26.0 (29.20) | -8.0 (9.14) | -3.6 (7.60) | 1.0 (19.34) | -1.5 (11.00)
  AST,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  AST,Week 2,n=38,39,26,24,26 | 6.1 (8.07) | 3.7 (4.81) | 4.5 (7.11) | -0.3 (2.66) | 0.4 (6.18)
  AST,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  AST,Week 4,n=37,38,25,23,27 | 5.4 (8.43) | 5.9 (6.74) | 5.0 (3.96) | -1.0 (2.75) | -0.7 (7.10)
  AST,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  AST,Week 8,n=34,31,24,22,23 | 6.4 (6.43) | 10.6 (8.90) | 6.7 (7.90) | 0.1 (2.74) | -1.6 (7.72)
  AST,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  AST,Week 12,n=32,28,24,22,21 | 7.6 (9.02) | 9.0 (5.64) | 6.5 (5.24) | 0.5 (3.62) | 0.1 (8.74)
  AST,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  AST,Week 16,n=28,26,22,19,18 | 8.5 (8.94) | 7.0 (5.79) | 8.0 (7.28) | 0.2 (4.45) | 1.0 (11.88)
  AST,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  AST,Week 20,n=25,23,19,18,16 | 14.6 (27.52) | 7.7 (7.24) | 9.0 (7.46) | 4.3 (20.22) | 1.4 (12.10)
  AST,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  AST,Week 24,n=22,21,16,17,16 | 9.8 (8.52) | 7.6 (6.75) | 10.5 (10.02) | 0.6 (4.40) | -1.3 (8.29)
  AST,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  AST,Week 28,n=19,18,12,13,14 | 9.0 (7.23) | 8.1 (7.30) | 9.4 (10.61) | 1.1 (3.88) | -0.1 (9.01)
  AST,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  AST,Week 32,n=19,15,10,12,13 | 8.8 (7.63) | 9.2 (7.72) | 8.0 (4.94) | 0.6 (3.65) | 1.2 (9.49)
  AST,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  AST,Week 36,n=15,12,10,12,13 | 10.6 (8.85) | 10.8 (8.09) | 7.6 (5.02) | 1.3 (2.56) | 0.2 (9.27)
  AST,Week 40,n=15,11,9,10,10: number analyzed (Participants) | 15 | 11 | 9 | 10 | 10
  AST,Week 40,n=15,11,9,10,10 | 8.9 (4.56) | 8.7 (10.82) | 9.1 (4.11) | 4.7 (13.17) | 6.7 (11.36)
  AST,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  AST,Week 44,n=11,11,6,8,9 | 8.1 (3.56) | 9.2 (8.91) | 8.3 (5.09) | 3.5 (4.81) | 2.3 (3.24)
  AST,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  AST,Week 48,n=9,8,5,8,5 | 8.1 (4.04) | 11.8 (12.63) | 9.8 (7.29) | 1.3 (4.68) | 6.4 (5.59)
  AST,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  AST,Week 52,n=9,5,5,5,4 | 7.1 (3.33) | 9.2 (4.97) | 11.6 (5.68) | -0.2 (3.63) | 4.3 (6.85)

34. Secondary Outcome: Part A: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin and Indirect Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters including bilirubin, creatinine, direct bilirubin and indirect bilirubin. Baseline was defined as the last non-missing value before first SC IP intake. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Groups:
- PartA:SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 42 | 39 | 26 | 27 | 27
Micromoles per liter
  Bilirubin,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Bilirubin,Week 2,n=38,39,26,24,26 | 1.8 (2.73) | 1.5 (3.12) | 1.9 (3.73) | -1.1 (1.94) | -1.0 (3.45)
  Bilirubin,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Bilirubin,Week 4,n=37,38,25,23,27 | 2.4 (5.05) | 1.9 (3.10) | 1.8 (2.76) | -1.8 (2.52) | -1.5 (5.22)
  Bilirubin,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Bilirubin,Week 8,n=34,31,24,22,23 | 3.0 (3.58) | 2.8 (4.81) | 0.9 (2.95) | -2.3 (2.50) | -3.2 (5.31)
  Bilirubin,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Bilirubin,Week 12,n=32,28,24,22,21 | 4.3 (8.49) | 2.8 (3.58) | 2.7 (3.44) | -1.0 (2.40) | -2.9 (4.52)
  Bilirubin,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Bilirubin,Week 16,n=28,26,22,19,18 | 2.7 (4.68) | 4.4 (4.53) | 3.9 (3.50) | -0.9 (1.85) | -3.3 (4.25)
  Bilirubin,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Bilirubin,Week 20,n=25,23,19,18,16 | 4.7 (9.09) | 4.3 (4.36) | 3.6 (3.58) | -1.4 (2.20) | -3.1 (4.67)
  Bilirubin,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Bilirubin,Week 24,n=22,21,16,17,16 | 4.9 (6.29) | 3.0 (4.41) | 4.8 (3.60) | -1.1 (1.80) | -1.7 (3.34)
  Bilirubin,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Bilirubin,Week 28,n=19,18,12,13,14 | 4.4 (5.86) | 3.7 (3.77) | 3.1 (3.18) | -0.8 (1.92) | -3.2 (3.72)
  Bilirubin,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Bilirubin,Week 32,n=19,15,10,12,13 | 4.2 (4.95) | 4.0 (4.54) | 2.7 (2.91) | -0.8 (2.53) | -3.0 (3.74)
  Bilirubin,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Bilirubin,Week 36,n=15,12,10,12,13 | 5.2 (4.66) | 5.3 (5.42) | 2.3 (2.91) | -0.9 (1.88) | -2.1 (4.91)
  Bilirubin,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Bilirubin,Week 40,n=15,11,6,10,10 | 5.1 (4.18) | 2.9 (4.13) | 2.6 (2.07) | -1.1 (2.02) | -1.9 (4.18)
  Bilirubin,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Bilirubin,Week 44,n=11,11,6,8,9 | 4.4 (6.14) | 1.8 (3.52) | 2.5 (2.17) | -0.1 (2.03) | -1.2 (3.23)
  Bilirubin,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Bilirubin,Week 48,n=9,8,5,8,5 | 6.7 (6.22) | 3.8 (3.62) | 2.2 (1.79) | -1.1 (1.96) | -1.8 (2.49)
  Bilirubin,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Bilirubin,Week 52,n=9,5,5,5,4 | 4.8 (5.09) | 1.6 (3.58) | 5.0 (4.36) | -1.0 (2.00) | 1.8 (6.85)
  Direct Bilirubin,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Direct Bilirubin,Week 2,n=38,39,26,24,26 | 0.1 (1.03) | -0.1 (0.92) | 0.1 (0.82) | 0.0 (0.59) | -0.3 (0.75)
  Direct Bilirubin,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Direct Bilirubin,Week 4,n=37,38,25,23,27 | 0.3 (0.97) | 0.1 (0.73) | 0.1 (0.76) | -0.2 (0.83) | -0.6 (1.31)
  Direct Bilirubin,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Direct Bilirubin,Week 8,n=34,31,24,22,23 | 0.2 (1.01) | 0.1 (0.72) | 0.0 (0.29) | -0.1 (0.75) | -0.8 (1.31)
  Direct Bilirubin,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Direct Bilirubin,Week 12,n=32,28,24,22,21 | 0.3 (1.12) | 0.1 (0.66) | 0.2 (0.96) | -0.1 (0.75) | -0.6 (1.29)
  Direct Bilirubin,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Direct Bilirubin,Week 16,n=28,26,22,19,18 | 0.3 (1.19) | 0.4 (0.98) | 0.3 (0.63) | -0.1 (0.46) | -0.8 (1.40)
  Direct Bilirubin,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Direct Bilirubin,Week 20,n=25,23,19,18,16 | 1.4 (3.29) | 0.1 (1.12) | 0.4 (0.77) | -0.2 (0.65) | -0.9 (1.45)
  Direct Bilirubin,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Direct Bilirubin,Week 24,n=22,21,16,17,16 | 1.0 (1.59) | 0.0 (0.89) | 0.4 (0.81) | -0.4 (0.79) | -0.8 (1.24)
  Direct Bilirubin,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Direct Bilirubin,Week 28,n=19,18,12,13,14 | 0.7 (1.34) | -0.1 (1.08) | 0.1 (0.90) | -0.5 (0.88) | -1.0 (1.52)
  Direct Bilirubin,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Direct Bilirubin,Week 32,n=19,15,10,12,13 | 0.5 (1.26) | 0.3 (1.03) | 0.1 (0.32) | -0.2 (0.58) | -1.2 (1.54)
  Direct Bilirubin,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Direct Bilirubin,Week 36,n=15,12,10,12,13 | 0.7 (1.22) | 0.3 (1.44) | -0.1 (0.74) | -0.2 (0.58) | -1.2 (1.54)
  Direct Bilirubin,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Direct Bilirubin,Week 40,n=15,11,6,10,10 | 0.6 (1.18) | -0.4 (0.81) | -0.3 (0.71) | 0.0 (0.00) | -1.4 (1.35)
  Direct Bilirubin,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Direct Bilirubin,Week 44,n=11,11,6,8,9 | 0.8 (0.98) | -0.4 (0.81) | 0.2 (0.41) | 0.0 (0.00) | -0.7 (1.00)
  Direct Bilirubin,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Direct Bilirubin,Week 48,n=9,8,5,8,5 | 1.2 (0.97) | -0.3 (0.71) | -0.6 (1.34) | 0.0 (0.00) | -1.2 (1.10)
  Direct Bilirubin,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Direct Bilirubin,Week 52,n=9,5,5,5,4 | 1.0 (1.00) | -0.8 (1.10) | -0.2 (1.10) | -0.4 (0.89) | -0.5 (1.00)
  Indirect Bilirubin,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Indirect Bilirubin,Week 2,n=38,39,26,24,26 | 1.7 (2.51) | 1.6 (2.84) | 1.8 (3.18) | -1.1 (1.75) | -0.7 (3.19)
  Indirect Bilirubin,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Indirect Bilirubin,Week 4,n=37,38,25,23,27 | 2.1 (4.93) | 1.9 (2.86) | 1.8 (2.31) | -1.6 (2.19) | -0.9 (4.27)
  Indirect Bilirubin,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Indirect Bilirubin,Week 8,n=34,31,24,22,23 | 2.8 (3.37) | 2.7 (4.37) | 0.9 (2.90) | -2.2 (2.47) | -2.4 (4.34)
  Indirect Bilirubin,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Indirect Bilirubin,Week 12,n=32,28,24,22,21 | 4.0 (7.94) | 2.7 (3.28) | 2.5 (2.87) | -1.0 (2.63) | -2.3 (3.79)
  Indirect Bilirubin,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Indirect Bilirubin,Week 16,n=28,26,22,19,18 | 2.4 (4.29) | 4.0 (3.88) | 3.6 (3.22) | -0.8 (1.84) | -2.5 (3.00)
  Indirect Bilirubin,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Indirect Bilirubin,Week 20,n=25,23,19,18,16 | 3.3 (6.22) | 4.2 (3.66) | 3.2 (3.21) | -1.2 (2.23) | -2.2 (3.47)
  Indirect Bilirubin,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Indirect Bilirubin,Week 24,n=22,21,16,17,16 | 4.0 (5.52) | 3.0 (3.88) | 4.4 (3.03) | -0.8 (1.64) | -0.9 (2.62)
  Indirect Bilirubin,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Indirect Bilirubin,Week 28,n=19,18,12,13,14 | 3.7 (5.05) | 3.8 (3.42) | 3.0 (3.02) | -0.3 (1.80) | -2.2 (2.55)
  Indirect Bilirubin,Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Indirect Bilirubin,Week 32,n=19,15,10,12,13 | 3.7 (4.24) | 3.7 (3.77) | 2.6 (2.99) | -0.6 (2.35) | -1.8 (2.52)
  Indirect Bilirubin,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Indirect Bilirubin,Week 36,n=15,12,10,12,13 | 4.5 (4.02) | 5.0 (4.47) | 2.4 (2.63) | -0.8 (1.66) | -0.8 (3.83)
  Indirect Bilirubin,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Indirect Bilirubin,Week 40,n=15,11,6,10,10 | 4.5 (3.94) | 3.3 (3.61) | 2.9 (2.03) | -1.1 (2.02) | -0.5 (2.95)
  Indirect Bilirubin,Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Indirect Bilirubin,Week 44,n=11,11,6,8,9 | 3.5 (5.43) | 2.2 (3.03) | 2.3 (2.34) | -0.1 (2.03) | -0.6 (2.88)
  Indirect Bilirubin,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Indirect Bilirubin,Week 48,n=9,8,5,8,5 | 5.4 (5.68) | 4.0 (3.21) | 2.8 (2.28) | -1.1 (1.96) | -0.6 (2.19)
  Indirect Bilirubin,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Indirect Bilirubin,Week 52,n=9,5,5,5,4 | 3.8 (4.52) | 2.4 (2.61) | 5.2 (5.02) | -0.6 (1.95) | 2.3 (6.13)
  Creatinine,Week 2,n=38,39,26,24,26: number analyzed (Participants) | 38 | 39 | 26 | 24 | 26
  Creatinine,Week 2,n=38,39,26,24,26 | 4.96 (9.319) | 4.10 (12.030) | 0.71 (5.170) | -1.65 (6.165) | 0.28 (7.485)
  Creatinine,,Week 4,n=37,38,25,23,27: number analyzed (Participants) | 37 | 38 | 25 | 23 | 27
  Creatinine,,Week 4,n=37,38,25,23,27 | 4.00 (11.061) | 3.03 (12.685) | 2.56 (6.760) | -0.64 (5.781) | 0.48 (7.222)
  Creatinine,Week 8,n=34,31,24,22,23: number analyzed (Participants) | 34 | 31 | 24 | 22 | 23
  Creatinine,Week 8,n=34,31,24,22,23 | 3.26 (10.522) | 1.48 (14.285) | 0.95 (6.027) | -2.93 (7.703) | 2.43 (8.688)
  Creatinine,,Week 12,n=32,28,24,22,21: number analyzed (Participants) | 32 | 28 | 24 | 22 | 21
  Creatinine,,Week 12,n=32,28,24,22,21 | 2.88 (11.590) | -0.84 (16.780) | 3.28 (6.334) | -3.09 (7.615) | 1.46 (6.093)
  Creatinine,,Week 16,n=28,26,22,19,18: number analyzed (Participants) | 28 | 26 | 22 | 19 | 18
  Creatinine,,Week 16,n=28,26,22,19,18 | 3.87 (9.387) | 1.16 (12.971) | 1.27 (6.604) | -0.14 (9.654) | 3.37 (15.068)
  Creatinine,,Week 20,n=25,23,19,18,16: number analyzed (Participants) | 25 | 23 | 19 | 18 | 16
  Creatinine,,Week 20,n=25,23,19,18,16 | -0.87 (8.652) | 0.33 (9.278) | -0.09 (5.721) | -0.18 (6.991) | 4.73 (12.179)
  Creatinine,Week 24,n=22,21,16,17,16: number analyzed (Participants) | 22 | 21 | 16 | 17 | 16
  Creatinine,Week 24,n=22,21,16,17,16 | 1.58 (9.671) | -0.45 (20.542) | 1.86 (9.364) | -1.14 (8.093) | 2.63 (7.834)
  Creatinine,,Week 28,n=19,18,12,13,14: number analyzed (Participants) | 19 | 18 | 12 | 13 | 14
  Creatinine,,Week 28,n=19,18,12,13,14 | 5.00 (12.803) | 0.46 (17.574) | -1.33 (5.372) | -0.28 (4.970) | 4.07 (7.431)
  Creatinine, Week 32,n=19,15,10,12,13: number analyzed (Participants) | 19 | 15 | 10 | 12 | 13
  Creatinine, Week 32,n=19,15,10,12,13 | 3.88 (11.182) | -2.52 (20.459) | -1.33 (7.598) | 0.59 (7.911) | 4.10 (7.264)
  Creatinine,,Week 36,n=15,12,10,12,13: number analyzed (Participants) | 15 | 12 | 10 | 12 | 13
  Creatinine,,Week 36,n=15,12,10,12,13 | 1.09 (11.330) | -3.82 (22.270) | 0.88 (7.151) | 4.56 (9.011) | 3.62 (11.433)
  Creatinine,,Week 40,n=15,11,6,10,10: number analyzed (Participants) | 15 | 11 | 6 | 10 | 10
  Creatinine,,Week 40,n=15,11,6,10,10 | 4.87 (11.617) | -1.45 (10.674) | -0.88 (9.831) | 1.67 (9.527) | 1.55 (10.630)
  Creatinine, Week 44,n=11,11,6,8,9: number analyzed (Participants) | 11 | 11 | 6 | 8 | 9
  Creatinine, Week 44,n=11,11,6,8,9 | 0.03 (14.182) | -7.06 (19.793) | -2.38 (7.847) | 0.23 (7.876) | 3.96 (14.656)
  Creatinine,,Week 48,n=9,8,5,8,5: number analyzed (Participants) | 9 | 8 | 5 | 8 | 5
  Creatinine,,Week 48,n=9,8,5,8,5 | 7.21 (14.144) | -7.15 (26.680) | 2.80 (8.917) | 1.43 (5.646) | 5.72 (18.804)
  Creatinine,,Week 52,n=9,5,5,5,4: number analyzed (Participants) | 9 | 5 | 5 | 5 | 4
  Creatinine,,Week 52,n=9,5,5,5,4 | 3.56 (6.903) | -5.10 (30.563) | 4.20 (9.195) | 1.78 (9.836) | 12.23 (16.814)

35. Secondary Outcome: Part A: Mean Serum Concentrations of Sirukumab
Description: Blood samples for Pharmacokinetic analysis of sirukumab serum concentrations were planned to be collected at specified time points.
Time Frame: Baseline (Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 44 and 52
Population: Safety Population. Data was not collected due to early termination of the study
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Part A: Mean Serum Anti-sirukumab Antibodies
Description: Blood samples for Pharmacokinetic analysis of Serum anti-sirukumab antibodies were planned to be collected at specified time points.
Time Frame: Baseline (Week 0) and up to 52 weeks
Population: Safety Population. Data was not collected due to early termination of the study
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Part A: Change From Baseline in Free and Total Interleukin-6 (IL-6) Over Time
Description: Blood samples for Pharmacodynamic analysis were planned but not collected due to early termination of study.
Time Frame: Baseline (Week 0) and up to 52 weeks
Population: Safety Population. Data was not collected due to early termination of the study
Arm/Group | PartA:SIR 100 mg SC q2w+6 Month Prednisone | PartA:SIR 100 mg SC q2w+3 Month Prednisone | PartA:SIR 50 mg SC q4w+6 Month Prednisone | PartA:Placebo SC q2w + 6 Month Prednisone | PartA:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Part B: Number of Participants With AEs, SAEs and Corticosteroid Related AEs Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinaemia were categorized as SAE. Number of participants with AEs, SAEs and corticosteroid related AEs for part B have been reported.
Time Frame: Up to 120 weeks
Population: Safety-Part B Population included all randomized participants who received at least 1 dose of SC IP in Part A and entered Part B
Measure: Count of Participants; unit: Participants
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Participants
  All AEs | 2 | 1 | 1 | 2 | 2
  All SAEs | 0 | 0 | 0 | 0 | 0
  Corticosteroid related AEs | 0 | 0 | 0 | 1 | 1

39. Secondary Outcome: Part B: Number of Participants With AEs, SAEs and Corticosteroid Related AEs Who Never Received 100mg OL Sirukumab in Part B
Description: as for outcome 38
Time Frame: Up to 120 weeks
Population: Safety-Part B Population
Measure: Count of Participants; unit: Participants
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Participants
  All AEs | 4 | 3 | 2 | 1 | 0
  All SAEs | 0 | 0 | 0 | 0 | 0
  Corticosteroid related AEs | 0 | 1 | 0 | 0 | 1

40. Secondary Outcome: Part B: Change From Baseline in SBP and DBP for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participant. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2,4,8,12,14,16,24,36,38,40 and follow up (Week 120)
Population: Safety-Part B Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Millimeters of mercury
  SBP,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  SBP,Week 2,n=1,1,0,1,2 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.5 (19.09)
  SBP,Week 4,n=2,1,1,2,2 | 5.0 (21.21) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.5 (3.54) | 1.5 (0.71)
  SBP,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  SBP,Week 8,n=2,1,1,2,1 | 14.0 (8.49) | 18.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -12.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -11.5 (10.61) | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  SBP,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  SBP,Week 12,n=2,1,1,1,0 | 7.0 (1.41) | 14.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  SBP,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  SBP,Week 14,n=0,0,0,1,0 |  |  |  | 9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  SBP,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  SBP,Week 16,n=2,0,0,1,0 | 0.0 (0.00) |  |  | 11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  SBP,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  SBP,Week 24,n=2,0,0,0,0 | 8.0 (0.00) |  |  |  |
  SBP,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  SBP,Week 36,n=2,0,0,0,0 | 11.0 (9.90) |  |  |  |
  SBP,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  SBP,Week 38,n=1,0,0,0,0 | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  SBP,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  SBP,Week 40,n=1,0,0,0,0 | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  SBP,Week follow up,n=2,1,0,1,1: number analyzed (Participants) | 2 | 1 | 0 | 1 | 1
  SBP,Week follow up,n=2,1,0,1,1 | 3.0 (18.38) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 22.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 12.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  DBP,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  DBP,Week 2,n=1,1,0,1,2 | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 7.0 (9.90)
  DBP,Week 4,n=2,1,1,2,2 | -3.0 (12.73) | -15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (5.66) | 4.5 (3.54)
  DBP,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  DBP,Week 8,n=2,1,1,2,1 | 3.0 (4.24) | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (2.83) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  DBP,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  DBP,Week 12,n=2,1,1,1,0 | -5.0 (7.07) | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  DBP,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  DBP,Week 14,n=0,0,0,1,0 |  |  |  | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  DBP,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  DBP,Week 16,n=2,0,0,1,0 | -5.0 (7.07) |  |  | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  DBP,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  DBP,Week 24,n=2,0,0,0,0 | 1.0 (1.41) |  |  |  |
  DBP,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  DBP,Week 36,n=2,0,0,0,0 | -2.0 (2.83) |  |  |  |
  DBP,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  DBP,Week 38,n=1,0,0,0,0 | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  DBP,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  DBP,Week 40,n=1,0,0,0,0 | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  DBP,Week follow up,n=2,1,0,1,1: number analyzed (Participants) | 2 | 1 | 0 | 1 | 1
  DBP,Week follow up,n=2,1,0,1,1 | -2.0 (5.66) | -7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 21.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis

41. Secondary Outcome: Part B: Change From Baseline in SBP and DBP for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participant. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24,36 and follow up (Week 120)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Millimeters of mercury
  SBP,Week 4,n=3,3,3,1,2: number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  SBP,Week 4,n=3,3,3,1,2 | -23.7 (4.73) | -6.3 (5.51) | 7.0 (25.36) | 10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (8.49)
  SBP,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  SBP,Week 8,n=2,1,2,0,2 | -32.5 (14.85) | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -7.5 (17.68) |  | -1.5 (0.71)
  SBP,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  SBP,Week 12,n=1,1,1,1,1 | -59.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 13.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  SBP,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  SBP,Week 16,n=0,1,1,1,0 |  | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 25.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  SBP,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SBP,Week 24,n=0,1,0,0,0 |  | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  SBP,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  SBP,Week 36,n=0,1,0,0,0 |  | -26.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  SBP,Week follow up,n=5,4,2,3,2: number analyzed (Participants) | 5 | 4 | 2 | 3 | 2
  SBP,Week follow up,n=5,4,2,3,2 | -7.4 (19.62) | -3.3 (8.54) | -17.5 (31.82) | 10.7 (10.07) | 5.0 (1.41)
  DBP,Week 4,n=3,3,3,1,2: number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  DBP,Week 4,n=3,3,3,1,2 | -8.3 (14.29) | 0.3 (4.51) | 7.7 (8.74) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | -11.0 (11.31)
  DBP,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  DBP,Week 8,n=2,1,2,0,2 | -9.0 (2.83) | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | 16.5 (2.12) |  | -6.0 (8.49)
  DBP,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  DBP,Week 12,n=1,1,1,1,1 | -22.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis.
  DBP,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  DBP,Week 16,n=0,1,1,1,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | -17.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |
  DBP,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  DBP,Week 24,n=0,1,0,0,0 |  | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |  |  |
  DBP,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  DBP,Week 36,n=0,1,0,0,0 |  | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |  |  |
  DBP,Week follow up,n=5,4,2,3,2: number analyzed (Participants) | 5 | 4 | 2 | 3 | 2
  DBP,Week follow up,n=5,4,2,3,2 | 3.4 (12.34) | -2.8 (4.57) | 12.5 (10.61) | 6.0 (4.36) | -2.0 (4.24)

42. Secondary Outcome: Part B: Change From Baseline in Pulse Rate for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Pulse rate was measured in semi-supine position after 5 minutes rest. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2,4,8,12,14,16,24,36,38,40 and follow up (Week 120)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
beats per minute
  Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2,n=1,1,0,1,2 | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (8.49)
  Week 4,n=2,1,1,2,2 | -2.0 (8.49) | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -17.0 (2.83) | -5.5 (9.19)
  Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Week 8,n=2,1,1,2,1 | 0.0 (5.66) | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -12.5 (9.19) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12,n=2,1,1,1,0 | -2.0 (2.83) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. | -12.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | -24.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |
  Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16,n=2,0,0,1,0 | 2.0 (2.83) |  |  | -14.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |
  Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24,n=2,0,0,0,0 | 5.0 (1.41) |  |  |  |
  Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36,n=2,0,0,0,0 | -2.0 (8.49) |  |  |  |
  Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis. |  |  |  |
  Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week follow up,n=2,1,0,1,1: number analyzed (Participants) | 2 | 1 | 0 | 1 | 1
  Week follow up,n=2,1,0,1,1 | 5.0 (12.73) | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -22.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis

43. Secondary Outcome: Part B: Change From Baseline in Pulse Rate for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Pulse rate was measured in semi-supine position after 5 minutes rest. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24,36 and follow up (Week 120)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
beats per minute
  Week 4,n=3,3,3,1,2: number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  Week 4,n=3,3,3,1,2 | 3.7 (1.53) | 0.3 (3.51) | -14.7 (2.31) | -29.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.5 (6.36)
  Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8,n=2,1,2,0,2 | 8.0 (4.24) | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.5 (2.12) |  | -0.5 (0.71)
  Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12,n=1,1,1,1,1 | 11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16,n=0,1,1,1,0 |  | -4.0 | -4.0 | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week follow up,n=5,4,2,3,2: number analyzed (Participants) | 5 | 4 | 2 | 3 | 2
  Week follow up,n=5,4,2,3,2 | 1.4 (10.11) | 4.0 (6.53) | -1.5 (2.12) | -7.7 (17.62) | 7.5 (4.95)

44. Secondary Outcome: Part B: Change From Baseline in Temperature for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Temperature was measured in semi-supine position after 5 minutes rest.. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2,4,8,12,14,16,24,36,38,40 and follow up (Week 120)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Celsius
  Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2,n=1,1,0,1,2 | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.65 (0.071)
  Week 4,n=2,1,1,2,2 | 0.15 (0.071) | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (0.141) | 0.30 (1.414)
  Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Week 8,n=2,1,1,2,1 | -0.15 (0.212) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (0.000) | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12,n=2,1,1,1,0 | -0.25 (0.071) | 0.90 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16,n=2,0,0,1,0 | -0.05 (0.071) |  |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24,n=2,0,0,0,0 | -0.42 (0.163) |  |  |  |
  Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36,n=2,0,0,0,0 | -0.25 (0.071) |  |  |  |
  Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38,n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40,n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week follow up,n=2,1,0,1,1: number analyzed (Participants) | 2 | 1 | 0 | 1 | 1
  Week follow up,n=2,1,0,1,1 | 0.15 (0.071) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis

45. Secondary Outcome: Part B: Change From Baseline in Temperature for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Temperature was measured in semi-supine position after 5 minutes rest.. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24,36 and follow up (Week 120)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Celsius
  Week 4,n=3,3,3,1,2: number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  Week 4,n=3,3,3,1,2 | 0.10 (0.458) | 0.07 (0.115) | 0.00 (0.300) | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (0.283)
  Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8,n=2,1,2,0,2 | -0.10 (0.566) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (0.283) |  | 0.05 (0.354)
  Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12,n=1,1,1,1,1 | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16,n=0,1,1,1,0 |  | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24,n=0,1,0,0,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36,n=0,1,0,0,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week follow up,n=5,4,2,3,2: number analyzed (Participants) | 5 | 4 | 2 | 3 | 2
  Week follow up,n=5,4,2,3,2 | 0.06 (0.305) | 0.15 (0.265) | 0.00 (0.283) | -0.13 (0.252) | 0.20 (0.283)

46. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters- Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameters including Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets. Change from Baseline is presented for these parameters.Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Giga cells per liter
  Eosinophils,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Eosinophils,Week 2,n=1,1,0,1,2 | -0.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.110 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.010 (0.0141)
  Eosinophils,Week 4,n=2,1,1,2,2 | -0.015 (0.0212) | -0.210 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.030 (0.0283) | 0.035 (0.0495)
  Eosinophils,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Eosinophils,Week 8,n=2,1,1,2,1 | -0.010 (0.0424) | -0.180 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.120 (0.1838) | 0.045 (0.0636)
  Eosinophils,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Eosinophils,Week 12,n=2,0,1,1,0 | -0.030 (0.0000) |  | 0.030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.160 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Eosinophils,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Eosinophils,Week 14,n=0,0,0,1,0 |  |  |  | -0.290 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Eosinophils,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Eosinophils,Week 16,n=2,0,0,1,0 | 0.030 (0.0141) |  |  | -0.270 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Eosinophils,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Eosinophils,Week 24,n=2,0,0,0,0 | -0.015 (0.0212) |  |  |  |
  Eosinophils,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Eosinophils,Week 36,n=2,0,0,0,0 | -0.010 (0.0566) |  |  |  |
  Eosinophils,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Eosinophils,Week 38,n=1,0,0,0,0 | 0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Eosinophils,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Eosinophils,Week 40,n=1,0,0,0,0 | -0.030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Leukocytes,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Leukocytes,Week 2,n=1,1,0,1,2 | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 2.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.30 (0.424)
  Leukocytes,Week 4,n=2,1,1,2,2 | 0.25 (0.778) | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.60 (1.697) | -1.45 (0.071)
  Leukocytes,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Leukocytes,Week 8,n=2,1,1,2,1 | -0.25 (1.061) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (0.000) | -0.95 (2.333)
  Leukocytes,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Leukocytes,Week 12,n=2,0,1,1,0 | -0.10 (0.990) |  | 0.90 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Leukocytes,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Leukocytes,Week 14,n=0,0,0,1,0 |  |  |  | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Leukocytes,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Leukocytes,Week 16,n=2,0,0,1,0 | -0.45 (0.778) |  |  | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Leukocytes,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Leukocytes,Week 24,n=2,0,0,0,0 | -0.20 (0.424) |  |  |  |
  Leukocytes,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Leukocytes,Week 36,n=2,0,0,0,0 | 0.65 (0.354) |  |  |  |
  Leukocytes,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Leukocytes,Week 38,n=1,0,0,0,0 | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Leukocytes,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Leukocytes,Week 40,n=1,0,0,0,0 | -1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Lymphocytes,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Lymphocytes,Week 2,n=1,1,0,1,2 | -0.170 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -0.400 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.160 (0.0990)
  Lymphocytes,Week 4,n=2,1,1,2,2 | 0.110 (0.0566) | -0.340 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.035 (0.2051) | -0.115 (0.5162)
  Lymphocytes,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Lymphocytes,Week 8,n=2,1,1,2,1 | -0.120 (0.0283) | 0.160 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.185 (0.3323) | -0.275 (0.4172)
  Lymphocytes,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Lymphocytes,Week 12,n=2,0,1,1,0 | -0.030 (0.0283) |  | 0.300 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.190 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Lymphocytes,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Lymphocytes,Week 14,n=0,0,0,1,0 |  |  |  | 0.490 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Lymphocytes,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Lymphocytes,Week 16,n=2,0,0,1,0 | -0.230 (0.2828) |  |  | 0.540 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Lymphocytes,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Lymphocytes,Week 24,n=2,0,0,0,0 | -0.320 (0.1697) |  |  |  |
  Lymphocytes,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Lymphocytes,Week 36,n=2,0,0,0,0 | 0.195 (0.1768) |  |  |  |
  LymphocytesWeek 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  LymphocytesWeek 38,n=1,0,0,0,0 | 0.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Lymphocytes,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Lymphocytes,Week 40,n=1,0,0,0,0 | -0.160 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Neutrophils ,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Neutrophils ,Week 2,n=1,1,0,1,2 | -0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.510 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 3.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.210 (0.5233)
  Neutrophils ,Week 4,n=2,1,1,2,2 | 0.205 (0.5728) | 0.400 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.230 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.740 (1.8950) | -1.420 (0.4950)
  Neutrophils ,Week 8,n=2,1,1,2,2 | -0.265 (0.6435) | 0.060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.620 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.485 (0.1909) | -0.790 (1.8385)
  Neutrophils ,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Neutrophils ,Week 12,n=2,0,1,1,0 | 0.020 (0.8061) |  | 0.630 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.320 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Neutrophils ,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Neutrophils ,Week 14,n=0,0,0,1,0 |  |  |  | 0.590 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Neutrophils ,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Neutrophils ,Week 16,n=2,0,0,1,0 | -0.235 (0.4879) |  |  | -0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Neutrophils ,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Neutrophils ,Week 24,n=2,0,0,0,0 | 0.085 (0.6859) |  |  |  |
  Neutrophils ,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Neutrophils ,Week 36,n=2,0,0,0,0 | 0.540 (0.6788) |  |  |  |
  Neutrophils ,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Neutrophils ,Week 38,n=1,0,0,0,0 | -0.460 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Neutrophils,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Neutrophils,Week 40,n=1,0,0,0,0 | -0.770 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Platelets ,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Platelets ,Week 2,n=1,1,0,1,2 | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -27.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -20.5 (57.28)
  Platelets,Week 4,n=2,1,1,2,2 | -1.0 (4.24) | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -33.5 (30.41) | -42.0 (11.31)
  Platelets,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Platelets,Week 8,n=2,1,1,2,1 | 7.0 (11.31) | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -20.5 (28.99) | -40.0 (0.00)
  Platelets,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Platelets,Week 12,n=2,0,1,1,0 | 7.0 (7.07) |  | 52.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 12.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Platelets,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Platelets,Week 14,n=0,0,0,1,0 |  |  |  | -31.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Platelets,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Platelets,Week 16,n=2,0,0,1,0 | 2.0 (1.41) |  |  | -97.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Platelets,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Platelets,Week 24,n=2,0,0,0,0 | -18.5 (9.19) |  |  |  |
  Platelets,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Platelets,Week 36,n=2,0,0,0,0 | 10.0 (21.21) |  |  |  |
  Platelets,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Platelets,Week 38,n=1,0,0,0,0 | -15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Platelets,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Platelets,Week 40,n=1,0,0,0,0 | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

47. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters- Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameters including Eosinophils, Leukocytes, Lymphocytes, Neutrophils and Platelets. Change from Baseline is presented for these parameters.Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Giga cells per liter
  Eosinophils,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Eosinophils,Week 4,n=3,3,2,1,2 | -0.110 (0.1735) | -0.013 (0.0551) | -0.050 (0.0849) | -0.030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.415 (0.5869)
  Eosinophils,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Eosinophils,Week 8,n=2,1,2,0,2 | -0.070 (0.0707) | 0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.020 (0.2546) |  | 0.330 (0.4101)
  Eosinophils,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Eosinophils,Week 12,n=1,1,1,1,1 | -0.120 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.120 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.190 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.070 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Eosinophils,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Eosinophils,Week 16,n=0,1,1,1,0 |  | -0.200 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.180 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Eosinophils,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Eosinophils,Week 24,n=0,1,0,0,0 |  | -0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Eosinophils,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Eosinophils,Week 36,n=0,1,0,0,0 |  | -0.240 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Leukocytes,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Leukocytes,Week 4,n=3,3,2,1,2 | 0.40 (0.500) | 0.30 (1.229) | 0.50 (0.000) | -0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.30 (0.990)
  Leukocytes,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Leukocytes,Week 8,n=2,1,2,0,2 | 0.25 (0.071) | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.90 (0.424) |  | 0.65 (0.071)
  Leukocytes,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Leukocytes,Week 12,n=1,1,1,1,1 | -1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Leukocytes,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Leukocytes,Week 16,n=0,1,1,1,0 |  | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Leukocytes,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Leukocytes,Week 24,n=0,1,0,0,0 |  | -0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Leukocytes,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Leukocytes,Week 36,n=0,1,0,0,0 |  | -1.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Lymphocytes,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Lymphocytes,Week 4,n=3,3,2,1,2 | 0.293 (0.2136) | 0.077 (0.2442) | 0.370 (0.0990) | -0.960 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.015 (0.2475)
  Lymphocytes,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Lymphocytes,Week 8,n=2,1,2,0,2 | 0.470 (0.0707) | 0.090 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.205 (0.0495) |  | -0.180 (0.4243)
  Lymphocytes,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Lymphocytes,Week 12,n=1,1,1,1,1 | -0.210 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.140 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.190 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.380 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.610 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Lymphocytes,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Lymphocytes,Week 16,n=0,1,1,1,0 |  | -0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.340 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.520 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Lymphocytes,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Lymphocytes,Week 24,n=0,1,0,0,0 |  | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Lymphocytes,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Lymphocytes,Week 36,n=0,1,0,0,0 |  | -0.240 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Neutrophils ,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Neutrophils ,Week 4,n=3,3,2,1,2 | 0.183 (0.4196) | 0.333 (1.0108) | 0.180 (0.1414) | 0.390 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.815 (0.0212)
  Neutrophils ,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Neutrophils ,Week 8,n=2,1,2,0,2 | -0.205 (0.1909) | 0.010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.600 (0.0283) |  | 0.500 (0.8627)
  Neutrophils ,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Neutrophils ,Week 12,n=1,1,1,1,1 | -0.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.440 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.820 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.770 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.140 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Neutrophils ,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Neutrophils ,Week 16,n=0,1,1,1,0 |  | -0.220 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.230 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.210 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Neutrophils ,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Neutrophils ,Week 24,n=0,1,0,0,0 |  | -0.350 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Neutrophils ,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Neutrophils ,Week 36,n=0,1,0,0,0 |  | -0.420 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Platelets,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Platelets,Week 4,n=3,3,2,1,2 | 15.0 (31.43) | -6.0 (9.64) | 10.5 (3.54) | 26.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -14.0 (4.24)
  Platelets,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Platelets,Week 8,n=2,1,2,0,2 | 17.5 (23.33) | -25.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 10.0 (22.63) |  | 31.5 (4.95)
  Platelets,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Platelets,Week 12,n=1,1,1,1,1 | 27.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -20.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 14.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 14.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Platelets,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Platelets,Week 16,n=0,1,1,1,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -19.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Platelets,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Platelets,Week 24,n=0,1,0,0,0 |  | -20.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Platelets,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Platelets,Week 36,n=0,1,0,0,0 |  | -16.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

48. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters- MCHC and Hemoglobin for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameters including MCHC and Hemoglobin. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Grams per liter
  MCHC,Week 2,n=1,1,0,1,1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  MCHC,Week 2,n=1,1,0,1,1 | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 20.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  MCHC,Week 4,n=2,1,0,2,1: number analyzed (Participants) | 2 | 1 | 0 | 2 | 1
  MCHC,Week 4,n=2,1,0,2,1 | -1.5 (3.54) | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 3.5 (2.12) | 23.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  MCHC,Week 8,n=2,1,0,2,1: number analyzed (Participants) | 2 | 1 | 0 | 2 | 1
  MCHC,Week 8,n=2,1,0,2,1 | 0.0 (12.73) | 16.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 3.5 (14.85) | 9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  MCHC,Week 12,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  MCHC,Week 12,n=2,0,0,1,0 | -5.5 (0.71) |  |  | 19.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  MCHC,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  MCHC,Week 14,n=0,0,0,1,0 |  |  |  | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  MCHC,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  MCHC,Week 16,n=2,0,0,1,0 | 0.0 (1.41) |  |  | 11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  MCHC,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  MCHC,Week 24,n=2,0,0,0,0 | -3.0 (2.83) |  |  |  |
  MCHC,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  MCHC,Week 36,n=2,0,0,0,0 | -4.0 (4.24) |  |  |  |
  MCHC,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  MCHC,Week 38,n=1,0,0,0,0 | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  MCHC,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  MCHC,Week 40,n=1,0,0,0,0 | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Hemoglobin,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Hemoglobin,Week 2,n=1,1,0,1,2 | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 10.0 (4.24)
  Hemoglobin,Week 4,n=2,1,1,2,2 | 0.5 (0.71) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (10.61) | 8.0 (8.49)
  Hemoglobin,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Hemoglobin,Week 8,n=2,1,1,2,1 | 4.0 (1.41) | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (10.61) | 9.0 (4.24)
  Hemoglobin,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Hemoglobin,Week 12,n=2,0,1,1,0 | 1.5 (3.54) |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hemoglobin,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Hemoglobin,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hemoglobin,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Hemoglobin,Week 16,n=2,0,0,1,0 | 0.0 (0.00) |  |  | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hemoglobin,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Hemoglobin,Week 24,n=2,0,0,0,0 | -0.5 (7.78) |  |  |  |
  Hemoglobin,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Hemoglobin,Week 36,n=2,0,0,0,0 | -1.5 (3.54) |  |  |  |
  Hemoglobin,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Hemoglobin,Week 38,n=1,0,0,0,0 | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Hemoglobin,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Hemoglobin,Week 40,n=1,0,0,0,0 | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

49. Secondary Outcome: Part B: Change From Baseline in Hematology Parameters- MCHC and Hemoglobin for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameters including MCHC and Hemoglobin. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Grams per liter
Groups:
- PartB:Placebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimenin Part A
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Grams per liter
  MCHC,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  MCHC,Week 4,n=3,3,2,1,2 | -18.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -14.0 (4.24) | -3.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -7.0 (11.31)
  MCHC,Week 8,n=0,1,2,0,2: number analyzed (Participants) | 0 | 1 | 2 | 0 | 2
  MCHC,Week 8,n=0,1,2,0,2 |  | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (16.26) |  | 8.0 (19.80)
  MCHC,Week 12,n=0,1,1,1,1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1
  MCHC,Week 12,n=0,1,1,1,1 |  | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 21.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  MCHC,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  MCHC,Week 16,n=0,1,1,1,0 |  | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  MCHC,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  MCHC,Week 24,n=0,1,0,0,0 |  | -17.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  MCHC,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  MCHC,Week 36,n=0,1,0,0,0 |  | -15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Hemoglobin,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Hemoglobin,Week 4,n=3,3,2,1,2 | -4.0 (5.29) | -6.3 (3.51) | 2.0 (9.90) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.5 (3.54)
  Hemoglobin,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Hemoglobin,Week 8,n=2,1,2,0,2 | -6.0 (14.14) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (12.73) |  | -1.5 (10.61)
  Hemoglobin,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Hemoglobin,Week 12,n=1,1,1,1,1 | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 20.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Hemoglobin,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Hemoglobin,Week 16,n=0,1,1,1,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 19.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hemoglobin,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Hemoglobin,Week 24,n=0,1,0,0,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Hemoglobin,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Hemoglobin,Week 36,n=0,1,0,0,0 |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

50. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter-Hematocrit for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Hematocrit. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Proportion of red blood cells in blood
  Hematocrit,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Hematocrit,Week 2,n=1,1,0,1,2 | -0.0080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0235 (0.01202)
  Hematocrit,Week 4,n=2,1,1,2,2 | 0.0030 (0.00141) | -0.0080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0060 (0.03111) | 0.0105 (0.00354)
  Hematocrit,Week 8,n=2,1,1,2,2 | 0.0115 (0.01909) | -0.0110 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0040 (0.01414) | 0.0260 (0.02546)
  Hematocrit,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Hematocrit,Week 12,n=2,0,1,1,0 | 0.0125 (0.01202) |  | -0.0060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0420 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hematocrit,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Hematocrit,Week 14,n=0,0,0,1,0 |  |  |  | -0.0080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hematocrit,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Hematocrit,Week 16,n=2,0,0,1,0 | 0.0000 (0.00141) |  |  | 0.0080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hematocrit,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Hematocrit,Week 24,n=2,0,0,0,0 | 0.0040 (0.02687) |  |  |  |
  Hematocrit,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Hematocrit,Week 36,n=2,0,0,0,0 | 0.0005 (0.01626) |  |  |  |
  Hematocrit,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Hematocrit,Week 38,n=1,0,0,0,0 | -0.0050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Hematocrit,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Hematocrit,Week 40,n=1,0,0,0,0 | -0.0140 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

51. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter-Hematocrit for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Hematocrit. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Proportion of red blood cells in blood
  Hematocrit,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Hematocrit,Week 4,n=3,3,2,1,2 | -0.0047 (0.02570) | -0.0057 (0.01834) | 0.0115 (0.02616) | -0.0040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0070 (0.00849)
  Hematocrit,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Hematocrit,Week 8,n=2,1,2,0,2 | -0.0185 (0.04879) | 0.0000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0135 (0.01768) |  | -0.0120 (0.00424)
  Hematocrit,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Hematocrit,Week 12,n=1,1,1,1,1 | -0.0120 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0470 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0010 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Hematocrit,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Hematocrit,Week 16,n=0,1,1,1,0 |  | 0.0060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0610 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.0030 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Hematocrit,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Hematocrit,Week 24,n=0,1,0,0,0 |  | 0.0100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Hematocrit,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Hematocrit,Week 36,n=0,1,0,0,0 |  | 0.0280 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

52. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter -Erythrocytes Mean Corpuscular Volume for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes Mean Corpuscular Volume. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Femtoliter
  Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2,n=1,1,0,1,2 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.5 (3.54)
  Week 4,n=2,1,1,2,2 | 1.5 (0.71) | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.5 (0.71) | 0.5 (2.12)
  Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Week 8,n=2,1,1,2,1 | 1.5 (2.12) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.5 (0.71) | 2.0 (2.83)
  Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Week 12,n=2,0,1,1,0 | 2.5 (0.71) |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16,n=2,0,0,1,0 | 0.5 (0.71) |  |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24,n=2,0,0,0,0 | 1.5 (0.71) |  |  |  |
  Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36,n=2,0,0,0,0 | 2.5 (2.12) |  |  |  |
  Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40,n=1,0,0,0,0 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

53. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter -Erythrocytes Mean Corpuscular Volume for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: as for outcome 51
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Femtoliter
  Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Week 4,n=3,3,2,1,2 | 0.7 (1.15) | 1.3 (1.53) | 0.0 (0.00) | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (1.41)
  Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8,n=2,1,2,0,2 | -0.5 (0.71) | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (1.41) |  | 1.5 (0.71)
  Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12,n=1,1,1,1,1 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16,n=0,1,1,1,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24,n=0,1,0,0,0 |  | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36,n=0,1,0,0,0 |  | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

54. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter-Erythrocytes Mean Corpuscular Hemoglobin for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes Mean Corpuscular Hemoglobin. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL Sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Picograms
  Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2,n=1,1,0,1,2 | -1.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.60 (0.990)
  Week 4,n=2,1,1,2,2 | 0.30 (0.000) | 0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.05 (0.354) | 1.00 (1.273)
  Week 8,n=2,1,1,2,2 | 0.30 (0.424) | 1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.45 (0.919) | 0.70 (0.141)
  Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12,n=2,1,1,1,0 | 0.25 (0.212) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | -0.90 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16,n=2,0,0,1,0 | 0.00 (0.00) |  |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24,n=2,0,0,0,0 | 0.10 (0.141) |  |  |  |
  Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36,n=2,0,0,0,0 | 0.25 (0.354) |  |  |  |
  Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38,n=1,0,0,0,0 | -0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40,n=1,0,0,0,0 | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

55. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter-Erythrocytes Mean Corpuscular Hemoglobin for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes Mean Corpuscular Hemoglobin. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Picograms
  Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Week 4,n=3,3,2,1,2 | -0.33 (0.757) | -0.47 (0.451) | -0.25 (0.354) | -1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (0.849)
  Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8,n=2,1,2,0,2 | -0.15 (0.354) | -0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (1.273) |  | 1.10 (2.121)
  Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12,n=1,1,1,1,1 | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16,n=0,1,1,1,0 |  | -0.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24,n=0,1,0,0,0 |  | -0.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36,n=0,1,0,0,0 |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

56. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter- Erythrocytes for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL Sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Trillion cells per liter
  Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2,n=1,1,0,1,2 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.25 (0.071)
  Week 4,n=2,1,1,2,2 | 0.00 (0.000) | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (0.283) | 0.10 (0.141)
  Week 8,n=2,1,1,2,2 | 0.10 (0.141) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.05 (0.212) | 0.15 (0.071)
  Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12,n=2,1,1,1,0 | 0.10 (0.141) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16,n=2,0,0,1,0 | 0.00 (0.00) |  |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24,n=2,0,0,0,0 | 0.00 (0.283) |  |  |  |
  Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36,n=2,0,0,0,0 | -0.05 (0.071) |  |  |  |
  Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38,n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40,n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

57. Secondary Outcome: Part B: Change From Baseline in Hematology Parameter- Erythrocytes for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the hematology parameter Erythrocytes. Change from Baseline is presented for this parameter. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Trillion cells per liter
  Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Week 4,n=3,3,2,1,2 | -0.03 (0.252) | -0.10 (0.173) | 0.10 (0.283) | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (0.000)
  Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8,n=2,1,2,0,2 | -0.15 (0.495) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (0.283) |  | -0.20 (0.000)
  Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12,n=1,1,1,1,1 | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16,n=0,1,1,1,0 |  | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24,n=0,1,0,0,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36,n=0,1,0,0,0 |  | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

58. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters- Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL Sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Millimoles per liter
  Calcium,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Calcium,Week 2,n=1,1,0,1,2 | 0.060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.040 (0.0000)
  Calcium,Week 4,n=2,1,1,2,2 | 0.070 (0.0707) | -0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.080 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.050 (0.1273) | 0.000 (0.0566)
  Calcium,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Calcium,Week 8,n=2,1,1,2,1 | 0.120 (0.0283) | -0.140 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.020 (0.0849) | 0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Calcium,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Calcium,Week 12,n=2,1,1,1,0 | 0.110 (0.0990) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Calcium,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Calcium,Week 14,n=0,0,0,1,0 |  |  |  | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Calcium,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Calcium,Week 16,n=2,0,0,1,0 | 0.000 (0.1131) |  |  | 0.140 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Calcium,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Calcium,Week 24,n=2,0,0,0,0 | 0.040 (0.0566) |  |  |  |
  Calcium,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Calcium,Week 36,n=2,0,0,0,0 | -0.050 (0.0707) |  |  |  |
  Calcium,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Calcium,Week 38,n=1,0,0,0,0 | -0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Calcium,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Calcium,Week 40,n=1,0,0,0,0 | -0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Carbon Dioxide,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Carbon Dioxide,Week 2,n=1,1,0,1,2 | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (0.00)
  Carbon Dioxide,Week 4,n=2,1,1,2,2 | 3.5 (3.54) | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.5 (2.12) | -3.5 (2.12)
  Carbon Dioxide,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Carbon Dioxide,Week 8,n=2,1,1,2,1 | 2.5 (2.12) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (0.00) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Carbon Dioxide,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Carbon Dioxide,Week 12,n=2,1,1,1,0 | 3.5 (2.12) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Carbon Dioxide,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Carbon Dioxide,Week 14,n=0,0,0,1,0 |  |  |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Carbon Dioxide,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Carbon Dioxide,Week 16,n=2,0,0,1,0 | 0.5 (0.71) |  |  | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Carbon Dioxide,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Carbon Dioxide,Week 24,n=2,0,0,0,0 | 3.0 (0.00) |  |  |  |
  Carbon Dioxide,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Carbon Dioxide,Week 36,n=2,0,0,0,0 | 1.5 (4.95) |  |  |  |
  Carbon Dioxide,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Carbon Dioxide,Week 38,n=1,0,0,0,0 | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Carbon Dioxide,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Carbon Dioxide,Week 40,n=1,0,0,0,0 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Chloride,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Chloride,Week 2,n=1,1,0,1,2 | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (1.41)
  Chloride,Week 4,n=2,1,1,2,2 | -2.5 (0.71) | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.5 (2.12) | 1.5 (0.71)
  Chloride,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Chloride,Week 8,n=2,1,1,2,1 | -3.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (1.41) | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Chloride,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Chloride,Week 12,n=2,1,1,1,0 | -2.5 (0.71) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Chloride,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Chloride,Week 14,n=0,0,0,1,0 |  |  |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Chloride,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Chloride,Week 16,n=2,0,0,1,0 | -1.0 (0.00) |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Chloride,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Chloride,Week 24,n=2,0,0,0,0 | -2.0 (1.41) |  |  |  |
  Chloride,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Chloride,Week 36,n=2,0,0,0,0 | 0.5 (0.71) |  |  |  |
  Chloride,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Chloride,Week 38,n=1,0,0,0,0 | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Chloride,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Chloride,Week 40,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Glucose,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Glucose,Week 2,n=1,1,0,1,2 | 0.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 1.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.25 (1.202)
  Glucose,Week 4,n=2,1,1,2,2 | 0.95 (1.202) | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.05 (2.192) | -0.05 (0.212)
  Glucose,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Glucose,Week 8,n=2,1,1,2,1 | 0.70 (0.424) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (1.414) | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Glucose,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Glucose,Week 12,n=2,1,1,1,0 | 0.60 (0.566) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Glucose,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Glucose,Week 14,n=0,0,0,1,0 |  |  |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Glucose,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Glucose,Week 16,n=2,0,0,1,0 | 0.55 (0.071) |  |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Glucose,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Glucose,Week 24,n=2,0,0,0,0 | 0.65 (0.354) |  |  |  |
  Glucose,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Glucose,Week 36,n=2,0,0,0,0 | 0.35 (0.071) |  |  |  |
  Glucose,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Glucose,Week 38,n=1,0,0,0,0 | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Glucose,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Glucose,Week 40,n=1,0,0,0,0 | 3.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Phosphate,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Phosphate,Week 2,n=1,1,0,1,2 | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -0.300 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (0.0707)
  Phosphate,Week 4,n=2,1,1,2,2 | -0.125 (0.1768) | -0.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.050 (0.2828) | -0.050 (0.1414)
  Phosphate,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Phosphate,Week 8,n=2,1,1,2,1 | 0.025 (0.1061) | -0.200 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.150 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.075 (0.3182) | -0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Phosphate,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Phosphate,Week 12,n=2,1,1,1,0 | -0.025 (0.1768) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.200 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Phosphate,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Phosphate,Week 14,n=0,0,0,1,0 |  |  |  | 0.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Phosphate,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Phosphate,Week 16,n=2,0,0,1,0 | -0.050 (0.0707) |  |  | 0.300 |
  Phosphate,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Phosphate,Week 24,n=2,0,0,0,0 | 0.050 (0.0000) |  |  |  |
  Phosphate,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Phosphate,Week 36,n=2,0,0,0,0 | -0.025 (0.0354) |  |  |  |
  Phosphate,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Phosphate,Week 38,n=1,0,0,0,0 | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Phosphate,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Phosphate,Week 40,n=1,0,0,0,0 | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Potassium,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Potassium,Week 2,n=1,1,0,1,2 | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (0.283)
  Potassium,Week 4,n=2,1,1,2,2 | 0.20 (0.283) | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.30 (0.141) | 0.00 (0.141)
  Potassium,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Potassium,Week 8,n=2,1,1,2,1 | 0.10 (0.424) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.30 (0.424) | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Potassium,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Potassium,Week 12,n=2,1,1,1,0 | 0.25 (0.636) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Potassium,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Potassium,Week 14,n=0,0,0,1,0 |  |  |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Potassium,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Potassium,Week 16,n=2,0,0,1,0 | 0.00 (0.141) |  |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Potassium,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Potassium,Week 24,n=2,0,0,0,0 | 0.40 (0.283) |  |  |  |
  Potassium,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Potassium,Week 36,n=2,0,0,0,0 | 0.20 (0.424) |  |  |  |
  Potassium,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Potassium,Week 38,n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Potassium,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Potassium,Week 40,n=1,0,0,0,0 | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Sodium,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Sodium,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (0.00)
  Sodium,Week 4,n=2,1,1,2,2 | -0.5 (0.71) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.5 (4.95) | 0.5 (0.71)
  Sodium,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Sodium,Week 8,n=2,1,1,2,1 | -2.0 (1.41) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (3.54) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Sodium,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Sodium,Week 12,n=2,1,1,1,0 | -1.0 (1.41) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Sodium,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Sodium,Week 14,n=0,0,0,1,0 |  |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Sodium,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Sodium,Week 16,n=2,0,0,1,0 | -1.5 (0.71) |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Sodium,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Sodium,Week 24,n=2,0,0,0,0 | -0.5 (0.71) |  |  |  |
  Sodium,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Sodium,Week 36,n=2,0,0,0,0 | 2.0 (0.00) |  |  |  |
  Sodium,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Sodium,Week 38,n=1,0,0,0,0 | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Sodium,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Sodium,Week 40,n=1,0,0,0,0 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Urea,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Urea,Week 2,n=1,1,0,1,2 | -1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.75 (0.354)
  Urea,Week 4,n=2,1,1,2,2 | 1.25 (0.354) | -1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.50 (0.707) | 0.25 (0.354)
  Urea,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Urea,Week 8,n=2,1,1,2,1 | 2.00 (2.121) | -2.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.25 (0.354) | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Urea,Week 12,n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Urea,Week 12,n=2,1,1,1,0 | -0.50 (2.121) | NA (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Urea,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Urea,Week 14,n=0,0,0,1,0 |  |  |  | 1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Urea,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Urea,Week 16,n=2,0,0,1,0 | 1.25 (1.768) |  |  | 1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Urea,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Urea,Week 24,n=2,0,0,0,0 | 0.00 (0.000) |  |  |  |
  Urea,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Urea,Week 36,n=2,0,0,0,0 | 0.00 (0.707) |  |  |  |
  Urea,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Urea,Week 38,n=1,0,0,0,0 | 1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Urea,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Urea,Week 40,n=1,0,0,0,0 | 1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

59. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters- Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including Calcium, Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Millimoles per liter
  Calcium,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Calcium,Week 4,n=3,3,2,1,2 | 0.067 (0.0643) | -0.093 (0.0462) | 0.060 (0.1414) | 0.120 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.040 (0.0566)
  Calcium,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Calcium,Week 8,n=2,1,2,0,2 | 0.010 (0.0707) | -0.060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.050 (0.0707) |  | 0.020 (0.0000)
  Calcium,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Calcium,Week 12,n=1,1,1,1,1 | 0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.160 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Calcium,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Calcium,Week 16,n=0,1,1,1,0 |  | 0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.180 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.060 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Calcium,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Calcium,Week 24,n=0,1,0,0,0 |  | -0.040 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Calcium,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Calcium,Week 36,n=0,1,0,0,0 |  | -0.020 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Carbon Dioxide,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Carbon Dioxide,Week 4,n=3,3,2,1,2 | 0.0 (2.00) | -2.7 (1.15) | 0.0 (2.83) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (0.00)
  Carbon Dioxide,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Carbon Dioxide,Week 8,n=2,1,2,0,2 | -0.5 (0.71) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.5 (3.54) |  | -1.5 (0.71)
  Carbon Dioxide,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Carbon Dioxide,Week 12,n=1,1,1,1,1 | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Carbon Dioxide,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Carbon Dioxide,Week 16,n=0,1,1,1,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Carbon Dioxide,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Carbon Dioxide,Week 24,n=0,1,0,0,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Carbon Dioxide,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Carbon Dioxide,Week 36,n=0,1,0,0,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Chloride,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Chloride,Week 4,n=3,3,2,1,2 | 0.7 (1.15) | 0.3 (3.06) | -2.5 (4.95) | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.5 (0.71)
  Chloride,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Chloride,Week 8,n=2,1,2,0,2 | -2.0 (0.00) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.5 (2.12) |  | 0.5 (2.12)
  Chloride,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Chloride,Week 12,n=1,1,1,1,1 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Chloride,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Chloride,Week 16,n=0,1,1,1,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Chloride,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Chloride,Week 24,n=0,1,0,0,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Chloride,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Chloride,Week 36,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Glucose,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Glucose,Week 4,n=3,3,2,1,2 | -0.10 (0.608) | 0.33 (1.115) | -0.80 (0.849) | 0.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.40 (0.707)
  Glucose,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Glucose,Week 8,n=2,1,2,0,2 | 0.15 (1.061) | 0.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.85 (0.071) |  | 0.55 (0.354)
  Glucose,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Glucose,Week 12,n=1,1,1,1,1 | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Glucose,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Glucose,Week 16,n=0,1,1,1,0 |  | 1.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Glucose,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Glucose,Week 24,n=0,1,0,0,0 |  | 1.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Glucose,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Glucose,Week 36,n=0,1,0,0,0 |  | 2.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Phosphate,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Phosphate,Week 4,n=3,3,2,1,2 | 0.050 (0.2646) | -0.033 (0.1155) | -0.125 (0.1768) | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.025 (0.1061)
  Phosphate,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Phosphate,Week 8,n=2,1,2,0,2 | 0.150 (0.1414) | -0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.250 (0.2121) |  | -0.075 (0.0354)
  Phosphate,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Phosphate,Week 12,n=1,1,1,1,1 | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Phosphate,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Phosphate,Week 16,n=0,1,1,1,0 |  | 0.100 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Phosphate,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Phosphate,Week 24,n=0,1,0,0,0 |  | 0.050 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Phosphate,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Phosphate,Week 36,n=0,1,0,0,0 |  | -0.150 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Potassium,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Potassium,Week 4,n=3,3,2,1,2 | -0.27 (0.289) | 0.03 (0.321) | 0.10 (0.141) | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (0.141)
  Potassium,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Potassium,Week 8,n=2,1,2,0,2 | -0.25 (0.212) | -0.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (0.424) |  | -0.10 (0.283)
  Potassium,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Potassium,Week 12,n=1,1,1,1,1 | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Potassium,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Potassium,Week 16,n=0,1,1,1,0 |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Potassium,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Potassium,Week 24,n=0,1,0,0,0 |  | -0.10 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Potassium,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Potassium,Week 36,n=0,1,0,0,0 |  | -0.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Sodium,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Sodium,Week 4,n=3,3,2,1,2 | 0.3 (1.53) | -1.0 (2.65) | -3.0 (2.83) | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (1.41)
  Sodium,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Sodium,Week 8,n=2,1,2,0,2 | -2.5 (0.71) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.5 (3.54) |  | -1.0 (1.41)
  Sodium,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Sodium,Week 12,n=1,1,1,1,1 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Sodium,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Sodium,Week 16,n=0,1,1,1,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Sodium,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Sodium,Week 24,n=0,1,0,0,0 |  | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Sodium,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Sodium,Week 36,n=0,1,0,0,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Urea,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Urea,Week 4,n=3,3,2,1,2 | -0.83 (0.577) | -0.50 (1.323) | -0.50 (0.707) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.25 (1.061)
  Urea,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Urea,Week 8,n=2,1,2,0,2 | -0.50 (0.707) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.75 (0.354) |  | 0.50 (0.707)
  Urea,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Urea,Week 12,n=1,1,1,1,1 | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Urea,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Urea,Week 16,n=0,1,1,1,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Urea,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Urea,Week 24,n=0,1,0,0,0 |  | -0.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Urea,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Urea,Week 36,n=0,1,0,0,0 |  | -1.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

60. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including Albumin and Protein. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Grams per liter
  Albumin,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Albumin,Week 2,n=1,1,0,1,2 | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.5 (0.71)
  Albumin,Week 4,n=2,1,1,2,2 | 0.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (2.83) | 3.0 (1.41)
  Albumin,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Albumin,Week 8,n=2,1,1,2,1 | 1.0 (2.83) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (2.83) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Albumin,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Albumin,Week 12,n=2,0,1,1,0 | 1.0 (0.00) |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Albumin,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Albumin,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Albumin,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Albumin,Week 16,n=2,0,0,1,0 | -0.5 (2.12) |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Albumin,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Albumin,Week 24,n=2,0,0,0,0 | -0.5 (3.54) |  |  |  |
  Albumin,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Albumin,Week 36,n=2,0,0,0,0 | -1.0 (2.83) |  |  |  |
  Albumin,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Albumin,Week 38,n=1,0,0,0,0 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Albumin,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Albumin,Week 40,n=1,0,0,0,0 | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Protein,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Protein,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.5 (2.12)
  Protein,Week 4,n=2,1,1,2,2 | 1.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (4.95) | -0.5 (2.12)
  Protein,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Protein,Week 8,n=2,1,1,2,1 | 3.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.5 (4.95) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Protein,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Protein,Week 12,n=2,0,1,1,0 | 2.5 (2.12) |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Protein,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Protein,Week 14,n=0,0,0,1,0 |  |  |  | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Protein,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Protein,Week 16,n=2,0,0,1,0 | 1.0 (1.41) |  |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Protein,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Protein,Week 24,n=2,0,0,0,0 | 0.5 (3.54) |  |  |  |
  Protein,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Protein,Week 36,n=2,0,0,0,0 | 1.5 (0.71) |  |  |  |
  Protein,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Protein,Week 38,n=1,0,0,0,0 | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Protein,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Protein,Week 40,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

61. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including Albumin and Protein. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Grams per liter
  Albumin,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Albumin,Week 4,n=3,3,2,1,2 | -0.3 (1.53) | -1.3 (0.58) | 1.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.5 (0.71)
  Albumin,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Albumin,Week 8,n=2,1,2,0,2 | 1.5 (2.12) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (2.83) |  | -1.5 (0.71)
  Albumin,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Albumin,Week 12,n=1,1,1,1,1 | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Albumin,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Albumin,Week 16,n=0,1,1,1,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Albumin,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Albumin,Week 24,n=0,1,0,0,0 |  | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Albumin,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Albumin,Week 36,n=0,1,0,0,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Protein,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Protein,Week 4,n=3,3,2,1,2 | -0.3 (3.21) | -2.7 (1.53) | 1.0 (5.66) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.0 (2.83)
  Protein,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Protein,Week 8,n=2,1,2,0,2 | 1.5 (3.54) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.5 (4.95) |  | -1.5 (3.54)
  Protein,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Protein,Week 12,n=1,1,1,1,1 | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Protein,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Protein,Week 16,n=0,1,1,1,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 12.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Protein,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Protein,Week 24,n=0,1,0,0,0 |  | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Protein,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Protein,Week 36,n=0,1,0,0,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

62. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP and AST for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including ALT,ALP and AST. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who received at least one dose of 100 mg OL sirukumab is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
International units per liter
  ALT,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  ALT,Week 2,n=1,1,0,1,2 | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 72.5 (101.12)
  ALT,Week 4,n=2,1,1,2,2 | -1.5 (3.54) | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (9.90) | 51.5 (64.35)
  ALT,Week 8,n=2,1,1,2,2 | 2.5 (4.95) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.5 (7.78) | 31.5 (24.75)
  ALT,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  ALT,Week 12,n=2,0,1,1,0 | -3.0 (7.07) |  | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALT,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  ALT,Week 14,n=0,0,0,1,0 |  |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALT,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  ALT,Week 16,n=2,0,0,1,0 | -1.0 (2.83) |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALT,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  ALT,Week 24,n=2,0,0,0,0 | -2.5 (6.36) |  |  |  |
  ALT,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  ALT,Week 36,n=2,0,0,0,0 | -4.5 (9.19) |  |  |  |
  ALT,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  ALT,Week 38,n=1,0,0,0,0 | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  ALT,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  ALT,Week 40,n=1,0,0,0,0 | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  ALP,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  ALP,Week 2,n=1,1,0,1,2 | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | -17.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.0 (5.66)
  ALP,Week 4,n=2,1,1,2,2 | 5.5 (0.71) | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -9.0 (14.14) | -7.0 (5.66)
  ALP,Week 8,n=2,1,1,2,2 | 7.0 (1.41) | -16.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.5 (26.16) | -12.0 (5.66)
  ALP,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  ALP,Week 12,n=2,0,1,1,0 | 5.0 (1.41) |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALP,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  ALP,Week 14,n=0,0,0,1,0 |  |  |  | -15.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALP,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  ALP,Week 16,n=2,0,0,1,0 | -0.5 (0.71) |  |  | -9.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALP,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  ALP,Week 24,n=2,0,0,0,0 | 2.5 (2.12) |  |  |  |
  ALP,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  ALP,Week 36,n=2,0,0,0,0 | 2.0 (5.66) |  |  |  |
  ALP,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  ALP,Week 38,n=1,0,0,0,0 | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  ALP,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  ALP,Week 40,n=1,0,0,0,0 | 18.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  AST,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  AST,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 44.5 (57.28)
  AST,Week 4,n=2,1,1,2,2 | -4.5 (0.71) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.5 (3.54) | 23.0 (25.46)
  AST,Week 8,n=2,1,1,2,2 | 1.5 (0.71) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (4.24) | 14.0 (5.66)
  AST,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  AST,Week 12,n=2,0,1,1,0 | -4.0 (1.41) |  | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  AST,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  AST,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  AST,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  AST,Week 16,n=2,0,0,1,0 | -3.0 (2.83) |  |  | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  AST,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  AST,Week 24,n=2,0,0,0,0 | -3.5 (2.12) |  |  |  |
  AST,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  AST,Week 36,n=2,0,0,0,0 | -4.5 (4.95) |  |  |  |
  AST,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  AST,Week 38,n=1,0,0,0,0 | -7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  AST,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  AST,Week 40,n=1,0,0,0,0 | -7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

63. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP and AST for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Blood samples were collected to analyze the chemistry parameters including ALT,ALP and AST. Change from Baseline is presented for these parameters. Baseline was defined as the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Data for participants who never received 100 mg open label Sirukumab has been presented
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
International units per liter
  ALT,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  ALT,Week 4,n=3,3,2,1,2 | 2.3 (1.15) | 2.7 (7.23) | -8.0 (4.24) | 103.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (0.00)
  ALT,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  ALT,Week 8,n=2,1,2,0,2 | 9.0 (7.07) | 13.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -9.5 (9.19) |  | -1.5 (3.54)
  ALT,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  ALT,Week 12,n=1,1,1,1,1 | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  ALT,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  ALT,Week 16,n=0,1,1,1,0 |  | -5.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALT,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ALT,Week 24,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  ALT,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ALT,Week 36,n=0,1,0,0,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  ALP,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  ALP,Week 4,n=3,3,2,1,2 | -0.7 (3.79) | 0.0 (4.36) | 0.5 (3.54) | 81.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (14.14)
  ALP,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  ALP,Week 8,n=2,1,2,0,2 | 1.5 (2.12) | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (4.24) |  | -3.0 (0.00)
  ALP,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  ALP,Week 12,n=1,1,1,1,1 | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 17.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -11.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  ALP,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  ALP,Week 16,n=0,1,1,1,0 |  | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -10.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  ALP,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ALP,Week 24,n=0,1,0,0,0 |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  ALP,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ALP,Week 36,n=0,1,0,0,0 |  | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  AST,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  AST,Week 4,n=3,3,2,1,2 | 0.7 (1.53) | 2.0 (3.00) | -5.0 (1.41) | 24.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.5 (3.54)
  AST,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  AST,Week 8,n=2,1,2,0,2 | 10.5 (9.19) | 7.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (2.83) |  | 0.0 (5.66)
  AST,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  AST,Week 12,n=1,1,1,1,1 | 1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  AST,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  AST,Week 16,n=0,1,1,1,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  AST,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  AST,Week 24,n=0,1,0,0,0 |  | -1.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  AST,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  AST,Week 36,n=0,1,0,0,0 |  | -3.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

64. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin and Indirect Bilirubin for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: as for outcome 60
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Micromoles per liter
  Bilirubin,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Bilirubin,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (1.41)
  Bilirubin,Week 4,n=2,1,1,2,2 | 5.0 (1.41) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (1.41) | 1.0 (1.41)
  Bilirubin,Week 8,n=2,1,1,2,2 | -1.0 (4.24) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (4.24) | 2.0 (0.00)
  Bilirubin,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Bilirubin,Week 12,n=2,0,1,1,0 | 0.0 (8.49) |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Bilirubin,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Bilirubin,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Bilirubin,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Bilirubin,Week 16,n=2,0,0,1,0 | 5.0 (4.24) |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Bilirubin,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Bilirubin,Week 24,n=2,0,0,0,0 | -2.0 (5.66) |  |  |  |
  Bilirubin,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Bilirubin,Week 36,n=2,0,0,0,0 | 1.0 (7.07) |  |  |  |
  Bilirubin,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Bilirubin,Week 38,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Bilirubin,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Bilirubin,Week 40,n=1,0,0,0,0 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Direct Bilirubin,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Direct Bilirubin,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (0.00)
  Direct Bilirubin,Week 4,n=2,1,1,2,2 | 1.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (1.41) | 0.0 (0.00)
  Direct Bilirubin,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Direct Bilirubin,Week 8,n=2,1,1,2,1 | 0.0 (2.83) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 1.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Direct Bilirubin,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Direct Bilirubin,Week 12,n=2,0,1,1,0 | 0.0 (2.83) |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Direct Bilirubin,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Direct Bilirubin,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Direct Bilirubin,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Direct Bilirubin,Week 16,n=2,0,0,1,0 | 1.0 (1.41) |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Direct Bilirubin,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Direct Bilirubin,Week 24,n=2,0,0,0,0 | 0.0 (0.00) |  |  |  |
  Direct Bilirubin,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Direct Bilirubin,Week 36,n=2,0,0,0,0 | -1.0 (1.41) |  |  |  |
  Direct Bilirubin,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin,Week 38,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Direct Bilirubin,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin,Week 40,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Indirect Bilirubin,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Indirect Bilirubin,Week 2,n=1,1,0,1,2 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.0 (1.41)
  Indirect Bilirubin,Week 4,n=2,1,1,2,2 | 4.0 (0.00) | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (0.00) | 1.0 (1.41)
  Indirect Bilirubin,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Indirect Bilirubin,Week 8,n=2,1,1,2,1 | -1.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (2.83) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Indirect Bilirubin,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Indirect Bilirubin,Week 12,n=2,0,1,1,0 | 0.0 (5.66) |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Indirect Bilirubin,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Indirect Bilirubin,Week 14,n=0,0,0,1,0 |  |  |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Indirect Bilirubin,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Indirect Bilirubin,Week 16,n=2,0,0,1,0 | 4.0 (5.66) |  |  | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Indirect Bilirubin,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Indirect Bilirubin,Week 24,n=2,0,0,0,0 | -2.0 (5.66) |  |  |  |
  Indirect Bilirubin,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Indirect Bilirubin,Week 36,n=2,0,0,0,0 | 2.0 (8.49) |  |  |  |
  Indirect Bilirubin,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Indirect Bilirubin,Week 38,n=1,0,0,0,0 | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Indirect Bilirubin,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Indirect Bilirubin,Week 40,n=1,0,0,0,0 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Creatinine,Week 2,n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Creatinine,Week 2,n=1,1,0,1,2 | -3.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  | 1.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.10 (1.838)
  Creatinine,Week 4,n=2,1,1,2,2 | -11.05 (9.405) | -12.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -1.30 (0.566) | 2.20 (4.384)
  Creatinine,Week 8,n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Creatinine,Week 8,n=2,1,1,2,1 | -8.40 (6.930) | -8.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 9.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.45 (5.728) | 0.00 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Creatinine,Week 12,n=2,0,1,1,0: number analyzed (Participants) | 2 | 0 | 1 | 1 | 0
  Creatinine,Week 12,n=2,0,1,1,0 | -11.90 (11.879) |  | 4.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -0.90 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Creatinine,Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Creatinine,Week 14,n=0,0,0,1,0 |  |  |  | 0.80 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Creatinine,Week 16,n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Creatinine,Week 16,n=2,0,0,1,0 | -12.80 (5.657) |  |  | 4.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Creatinine,Week 24,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Creatinine,Week 24,n=2,0,0,0,0 | -9.75 (12.516) |  |  |  |
  Creatinine,Week 36,n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Creatinine,Week 36,n=2,0,0,0,0 | -15.05 (9.970) |  |  |  |
  Creatinine,Week 38,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Creatinine,Week 38,n=1,0,0,0,0 | -19.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |
  Creatinine,Week 40,n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Creatinine,Week 40,n=1,0,0,0,0 | -20.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |  |

65. Secondary Outcome: Part B: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin and Indirect Bilirubin for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: as for outcome 61
Time Frame: Baseline (Week 0) and Weeks 4,8,12,16,24 and 36
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Groups:
- PartBSIR 100 mg SC q2w+6 Month Prednisone: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen in Part A
- PartBSIR 100 mg SC q2w+3 Month Prednisone: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen in Part A
- PartBPlacebo SC q2w + 6 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A
- PartBPlacebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen in Part A
Arm/Group | PartBSIR 100 mg SC q2w+6 Month Prednisone | PartBSIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartBPlacebo SC q2w + 6 Month Prednisone | PartBPlacebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Micromoles per liter
  Bilirubin,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Bilirubin,Week 4,n=3,3,2,1,2 | 0.7 (3.06) | 1.3 (3.06) | -5.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -8.0 (2.83)
  Bilirubin,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Bilirubin,Week 8,n=2,1,2,0,2 | 3.0 (4.24) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (2.83) |  | -6.0 (5.66)
  Bilirubin,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Bilirubin,Week 12,n=1,1,1,1,1 | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -8.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Bilirubin,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Bilirubin,Week 16,n=0,1,1,1,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Bilirubin,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Bilirubin,Week 24,n=0,1,0,0,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Bilirubin,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Bilirubin,Week 36,n=0,1,0,0,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Direct Bilirubin,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Direct Bilirubin,Week 4,n=3,3,2,1,2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (0.00)
  Direct Bilirubin,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Direct Bilirubin,Week 8,n=2,1,2,0,2 | 1.0 (1.41) | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (0.00) |  | -2.0 (0.00)
  Direct Bilirubin,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Direct Bilirubin,Week 12,n=1,1,1,1,1 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Direct Bilirubin,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Direct Bilirubin,Week 16,n=0,1,1,1,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Direct Bilirubin,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Direct Bilirubin,Week 24,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Direct Bilirubin,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Direct Bilirubin,Week 36,n=0,1,0,0,0 |  | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Indirect Bilirubin,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Indirect Bilirubin,Week 4,n=3,3,2,1,2 | 0.7 (3.06) | 1.3 (3.06) | -5.0 (1.41) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (2.83)
  Indirect Bilirubin,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Indirect Bilirubin,Week 8,n=2,1,2,0,2 | 2.0 (2.83) | 0.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (2.83) |  | -4.0 (5.66)
  Indirect Bilirubin,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Indirect Bilirubin,Week 12,n=1,1,1,1,1 | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -6.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Indirect Bilirubin,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Indirect Bilirubin,Week 16,n=0,1,1,1,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Indirect Bilirubin,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Indirect Bilirubin,Week 24,n=0,1,0,0,0 |  | -2.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Indirect Bilirubin,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Indirect Bilirubin,Week 36,n=0,1,0,0,0 |  | -4.0 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Creatinine,Week 4,n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Creatinine,Week 4,n=3,3,2,1,2 | -7.07 (7.887) | -0.63 (4.842) | -1.30 (9.334) | -0.90 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 3.95 (19.445)
  Creatinine,Week 8,n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Creatinine,Week 8,n=2,1,2,0,2 | -8.40 (0.566) | -18.60 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -5.25 (3.748) |  | -5.75 (5.728)
  Creatinine,Week 12,n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Creatinine,Week 12,n=1,1,1,1,1 | -6.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -27.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 9.70 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | -19.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Creatinine,Week 16,n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Creatinine,Week 16,n=0,1,1,1,0 |  | -19.50 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 5.30 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Creatinine,Week 24,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Creatinine,Week 24,n=0,1,0,0,0 |  | -27.40 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |
  Creatinine,Week 36,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Creatinine,Week 36,n=0,1,0,0,0 |  | -21.20 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |  |  |

66. Secondary Outcome: Part B: Cumulative Prednisone Dose Over Time for Participants Who Received at Least One Dose of 100 mg Open-label Sirukumab in Part B
Description: Cumulative prednisone dose is the cumulative doses taken from start of Part B. The cumulative prednisone dose at each visit was calculated based on the number of participants who attended that visit. Data for participants who received at least one dose of 100mg open label Sirukumab was presented.
Time Frame: Weeks 2, 4, 8, 12, 14, 16, 24, 28, 32 and 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Milligrams
  Week 2, n=0,0,0,1,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Week 2, n=0,0,0,1,1 |  |  |  | 561.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 550.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 4,n=0,0,0,2,1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1
  Week 4,n=0,0,0,2,1 |  |  |  | 596.125 (586.7219) | 775.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 8,n=0,0,0,2,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0
  Week 8,n=0,0,0,2,0 |  |  |  | 956.125 (851.8869) |
  Week 12,n=0,0,0,2,1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1
  Week 12,n=0,0,0,2,1 |  |  |  | 1201.125 (1000.3793) | 1600.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 14,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14,n=0,0,0,1,0 |  |  |  | 843.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 16,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 16,n=0,0,0,1,0 |  |  |  | 1233.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 24,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 24,n=0,0,0,1,0 |  |  |  | 1853.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 28,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 28,n=0,0,0,1,0 |  |  |  | 1908.500 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 32,n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 32,n=0,0,0,0,1 |  |  |  |  | 1600.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 38,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 38,n=0,0,0,1,0 |  |  |  | 2153.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |

67. Secondary Outcome: Part B: Cumulative Prednisone Dose Over Time for Participants Who Never Received 100 mg Open Label Sirukumab in Part B
Description: Cumulative prednisone dose is the cumulative doses taken from start of Part B. The cumulative prednisone dose at each visit was calculated based on the number of participants who attended that visit. Data for participants who never received 100 mg open label Sirukumab has been presented.
Time Frame: Weeks 2, 4, 8, 12, 14, 16, 24, 28, 32 and 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | PartBSIR 100 mg SC q2w+6 Month Prednisone | PartBSIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartBPlacebo SC q2w + 6 Month Prednisone | PartBPlacebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Milligrams
  Week 2, n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 4,n=0,0,0,1,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Week 4,n=0,0,0,1,1 |  |  |  | 203.750 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 325.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 8,n=0,0,0,1,1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Week 8,n=0,0,0,1,1 |  |  |  | 357.500 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis | 596.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 12,n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 12,n=0,0,0,0,1 |  |  |  |  | 830.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 14,n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 16,n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 16,n=0,0,0,0,1 |  |  |  |  | 1020.000 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 24,n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 24,n=0,0,0,1,0 |  |  |  | 397.500 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis |
  Week 28,n= 0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 32,n=0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Week 32,n=0,0,0,0,1 |  |  |  |  | 1211.250 (NA) — NA indicates data is not available since standard deviation was not derived because only one participant was available at the time of analysis
  Week 38,n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Part B: Number of Disease Flares Over Time
Description: This summarizes disease flares over time with no adjustment for exposure to study drugs, calculated by taking the last visit before a participant withdrew and then counting the number of participants with at least 1 flare up to that point and summing up the total number of flares experienced by each of these participants. Data for number of disease flares per participant over time for part B were presented.
Time Frame: Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: as for outcome 4
Measure: Number; unit: Disease flares
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 4
Disease flares
  Week 2, n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2, n=1,1,0,1,2 | 0 | 0 |  | 0 | 0
  Week 4, n=5,4,4,3,4: number analyzed (Participants) | 5 | 4 | 4 | 3 | 4
  Week 4, n=5,4,4,3,4 | 0 | 0 | 0 | 0 | 0
  Week 8, n=4,2,3,2,3: number analyzed (Participants) | 4 | 2 | 3 | 2 | 3
  Week 8, n=4,2,3,2,3 | 0 | 0 | 1 | 0 | 0
  Week 12, n=3,2,2,2,1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 1
  Week 12, n=3,2,2,2,1 | 0 | 0 | 1 | 0 | 0
  Week 14, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14, n=0,0,0,1,0 |  |  |  | 1 |
  Week 16, n=2,1,1,2,0: number analyzed (Participants) | 2 | 1 | 1 | 2 | 0
  Week 16, n=2,1,1,2,0 | 0 | 0 | 0 | 1 |
  Week 24, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Week 24, n=2,1,0,0,0 | 0 | 0 |  |  |
  Week 36, n=2,1,0,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Week 36, n=2,1,0,0,0 | 0 | 0 |  |  |
  Week 38, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38, n=1,0,0,0,0 | 2 |  |  |  |
  Week 40, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40, n=1,0,0,0,0 | 2 |  |  |  |

69. Secondary Outcome: Part B: Number of Participants Requiring at Least One Hospitalization for Disease Flare
Description: Number of participants with at least one flare at a given visit was the number of participants with at least one flare between first SC IP intake and the day of the given visit. The hospitalizations for disease flare were planned to be identified through the adjudication of adverse events of special interest, and include events from the category: "Severe Flare including Hospitalizations". Data for participants requiring hospitalizations for disease flare for part B was not available due to early termination of study.
Time Frame: Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: ITT-Part B Population.
Measure: Count of Participants; unit: Participants
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 4
Participants | 0 | 0 | 0 | 0 | 0

70. Secondary Outcome: Part B: Number of Hospitalizations for Disease Flare Over Time
Description: as for outcome 69
Time Frame: Up to Week 104
Population: ITT-Part B Population.
Measure: Number; unit: Number of hospitalizations
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 4
Number of hospitalizations | 0 | 0 | 0 | 0 | 0

71. Secondary Outcome: Part B: Change From Baseline in 36-item SF-36 v2 Acute Score Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: SF-36v2 acute health survey questionnaire was developed as part of the Rand Health Insurance Experiment and consists of the following 8 multi-item scales: 1. Limitations in physical functioning due to health problems, 2. Limitations in usual role activities due to physical health problems, 3. Bodily pain, 4. General mental health (psychological distress and well-being), 5. Limitations in usual role activities due to personal or emotional problems, 6. Limitations in social functioning due to physical or mental health problems. 7. Vitality (energy and fatigue) and 8. General health perception. These 8 scales were scored from 0 to 100, 0 (worst score) to 100 (best score) where higher scores indicates better health. Data for participants (Par) who received at least one dose of 100 mg OL Sirukumab has been presented. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0), Day 85, Day 87, Day 91, Day 113, Day 162, Day 339, Day 344, Week 12 and Week 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 12, Physical Functioning | -10 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Role Physical | -12.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Bodily Pain | -39 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, General Health | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Vitality | -6.25 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Social Functioning | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Role Emotional | -8.33 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Mental Health | 10 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Physical Component Summary | -8.76 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Mental Component Summary | 3.29 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Physical Functioning | -4.99 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Role Physical | -12.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Bodily Pain | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, General Health | -5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Vitality | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Social Functioning | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Role Emotional | -16.67 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Mental Health | 5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Physical Component Summary | -2.09 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Mental Component Summary | -0.76 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Physical Functioning | 9.99 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Role Physical | 37.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Bodily Pain | 23 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, General Health | 5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Vitality | 6.25 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Social Functioning | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Role Emotional | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Mental Health | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Physical Component Summary | 9.98 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Mental Component Summary | -2.78 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Physical Functioning | 4.99 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Role Physical | 50 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Bodily Pain | 49 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, General Health | 10 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Vitality | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Social Functioning | 12.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Mental Health | -10 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Physical Component Summary | 15.7 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Mental Component Summary | -5.84 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Physical Functioning | 24.99 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Role Physical | 50 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Bodily Pain | 33 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, General Health | 5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Vitality | -6.25 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Social Functioning | 12.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Role Emotional | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Mental Health | -20 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Physical Component Summary | 17.37 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Mental Component Summary | -10.18 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Physical Functioning | -5.01 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Role Physical | 37.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Bodily Pain | 11 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, General Health | 10 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Vitality | -6.25 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Social Functioning | 12.5 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Role Emotional | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Mental Health | -15 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Physical Component Summary | 8.12 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Mental Component Summary | -4.89 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.72 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.05 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 15 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 33 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.28 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.59 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -18.75 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -16 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10 | 10
  Par 5, Week 12, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -16.66 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.34 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5.35 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10.01 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -18.75 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -16 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -7 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12.5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -33.33 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Physical Component Summary | 168 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.62 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -8.24 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -15 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 22 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 20 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5.17 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5.95 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 85, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10.01
  Par 7, Day 85, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25
  Par 7, Day 85, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -22
  Par 7, Day 85, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10
  Par 7, Day 85, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12.5
  Par 7, Day 85, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 85, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 85, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5
  Par 7, Day 85, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -4.79
  Par 7, Day 85, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.82
  Par 8, Day 87, Physical Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 8, Day 87, Role Physical | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25
  Par 8, Day 87, Bodily Pain | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 21
  Par 8, Day 87, General Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 8, Day 87, Vitality | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 8, Day 87, Social Functioning | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 12.5
  Par 8, Day 87, Role Emotional | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 16.66
  Par 8, Day 87, Mental Health | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5
  Par 8, Day 87, Physical Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.52
  Par 8, Day 87, Mental Component Summary | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 4.54

72. Secondary Outcome: Part B: Change From Baseline in 36-item SF-36 v2 Acute Score Over Time for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: SF-36v2 acute health survey questionnaire was developed as part of the Rand Health Insurance Experiment and consists of the following 8 multi-item scales: 1. Limitations in physical functioning due to health problems, 2. Limitations in usual role activities due to physical health problems, 3. Bodily pain, 4. General mental health (psychological distress and well-being), 5. Limitations in usual role activities due to personal or emotional problems, 6. Limitations in social functioning due to physical or mental health problems. 7. Vitality (energy and fatigue) and 8. General health perception. These 8 scales were scored from 0 to 100, 0 (worst score) to 100 (best score) where higher scores indicates better health. Data for participants (Par) who never received 100 mg OL Sirukumab has been presented. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Day 23, Day 29, Day 30, Day 57, Day 59, Day 64, Day 65 , Day 85, Day 112, Day 113, Day 163, Day 169, Day 373, Week 8 and Week 12
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 2 | 2
Scores on scale
  Par 1, Day 30, Physical Functioning | -5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Role Physical | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Bodily Pain | -16 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, General health | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Vitality | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Social Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Role emotional | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Mental health | 5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Physical Component Summary | -2.26 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 30, Mental Component Summary | 2.26 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Physical Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Role Physical | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Bodily Pain | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, General health | 8 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Vitality | 6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Social Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Role emotional | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Mental health | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Physical Component Summary | -0.12 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, Mental Component Summary | 3.18 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Physical Functioning | 25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Role Physical | 6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Bodily Pain | 49 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, General health | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Vitality | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Social Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Role emotional | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Mental health | -5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Physical Component Summary | 12.88 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, Mental Component Summary | -5.75 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Physical Functioning | 15 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Role Physical | 18.75 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Bodily Pain | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, General health | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Vitality | 6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Social Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Role emotional | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Mental health | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Physical Component Summary | 4.88 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Mental Component Summary | -1.45 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Physical Functioning | 15 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Role Physical | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Bodily Pain | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, General health | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Vitality | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Social Functioning | -12.5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Role emotional | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Mental health | 25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Physical Component Summary | 0.77 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, Mental Component Summary | 3.61 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Physical Functioning | -5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Role Physical | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Bodily Pain | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, General health | -10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Vitality | -6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Social Functioning | -12.5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Role emotional | 16.67 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Mental health | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Physical Component Summary | -2.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, Mental Component Summary | 1.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Physical Functioning | 5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Role Physical | -6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Bodily Pain | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, General health | -22 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Vitality | -6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Social Functioning | -12.5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Role emotional | 8.33 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Mental health | 10 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Physical Component Summary | -3.17 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, Mental Component Summary | 1.62 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Physical Functioning | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Role Physical | 6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Bodily Pain | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, General health | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Vitality | -6.25 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Social Functioning | 12.5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Role emotional | 8.33 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Mental health | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Physical Component Summary | -0.01 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, Mental Component Summary | 1.88 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 16 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3.33 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2.88 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 15 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 16 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 8 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -15 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 7.95 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -22 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12.5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -15 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3.24 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.02 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 3.22 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3.68 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 12.5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 12.5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.95 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.83 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -29.99 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -18.75 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -13 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -9.37 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.44 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -15.01 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -8 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -37.5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 9 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3.64 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.4 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -6.25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -11 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 6.25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -16.67 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -2.76 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.13 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -12.5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -12.5 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -25 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 2.16 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -7.59 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -5.01 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -18.75 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -32 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 10 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 12.5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -37.5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 15 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -7.54 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 3.62 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 4.99 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 50 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 33 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 6.25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 25 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 50 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 7.93 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 8.48 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Week 12, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5
  Par 16, Week 12, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25
  Par 16, Week 12, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 28
  Par 16, Week 12, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Week 12, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25
  Par 16, Week 12, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Week 12, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Week 12, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Week 12, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5.1
  Par 16, Week 12, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2.52
  Par 16, Day 112, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Day 112, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 12.5
  Par 16, Day 112, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 28
  Par 16, Day 112, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -20
  Par 16, Day 112, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.25
  Par 16, Day 112, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Day 112, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Day 112, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 16, Day 112, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 2.71
  Par 16, Day 112, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2.21
  Par 17, Day 85, Physical Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10
  Par 17, Day 85, Role Physical | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -25
  Par 17, Day 85, Bodily Pain | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10
  Par 17, Day 85, General health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 17, Day 85, Vitality | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6.25
  Par 17, Day 85, Social Functioning | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12.5
  Par 17, Day 85, Role emotional | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0
  Par 17, Day 85, Mental health | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5
  Par 17, Day 85, Physical Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.51
  Par 17, Day 85, Mental Component Summary | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 3.01

73. Secondary Outcome: Part B: Change From Baseline in EQ-5D-5L Index Score Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: EuroQoL-5 Dimensions consist of 2 elements: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprised of following 5 dimensions: 1.Mobility, 2.Self-Care, 3.Usual Activities, 4.Pain/Discomfort and 5.Anxiety/Depression. Each of these 5 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The digits for each of 5 dimensions were combined in a 5-digit number describing the participant's health state: e.g. state 11111 indicates no problem on any of the 5 dimensions. Index score was derived from the 5 dimensions scores using UK tariff. The weights based from the UK population was used for conversion, regardless of the origin country of participant. The score ranged from -0.594 (worst score) to 1.000 (best score). Baseline was last measurement done up to and including Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Day 85, Day 87, Day 91, Day 113, Day 162, Day 339, Day 344, Week 12 and Week24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 12 | -0.127 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Week 24 | -0.098 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Day 339 | -0.070 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 12 | 0.204 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 24 | 0.041 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Day 344 | 0.110 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 3, Day 113 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.000 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 4, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.097 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.028 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Day 162 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.028 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 6, Day 91 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.000 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 7, Day 85 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.000
  Par 8, Day 87 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.012

74. Secondary Outcome: Part B: Change From Baseline in EQ-5D-5L Index Score Over Time for Participants Who Never Received 100mg OL Sirukumab in Part B
Description: as for outcome 73
Time Frame: Baseline (Day 0) and Day 29, 30, 57, 59, 64, 65, 85, 112, 113,163,169 and 373, Week 12
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Scores on scale
  Par 1, Day 30 | -0.248 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29 | 0.000 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 29 | 0.233 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | 0.000 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113 | 0.000 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85 | -0.015 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65 | 0.163 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.163 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.163 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.016 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.212 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.000 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.069 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.042 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.059 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.000 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.000 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Day 169 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.232 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 17,Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.163
  Par 17, Day 112 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.163
  Par 18, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.042

75. Secondary Outcome: Part B: Change From Baseline in FACIT-Fatigue Scores Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: The FACIT-Fatigue is a 13-item questionnaire formatted for self-administration that assesses participant reported fatigue and its impact upon daily activities and function over the past seven days. Participants were asked to answer each question using a 5-point Likert-type scale (4 = Not at all; 3 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 0 = Very Much) where 0 is a bad response and 4 is good response. Each of the 13 items of the FACIT-Fatigue Scale ranges from 0-4, with a range of possible total score from 0-52, 0 (Extreme fatigue) to 52 (No fatigue) where 0 being the worst possible score and 52 the best (i.e. less fatigue). Scores below 30 indicate severe fatigue. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Day 85,87,91,113,162, 344,339,Week 12, 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 12, I Feel Fatigued | -3 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Week 24, I Feel Fatigued | -4 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Day 339, I Feel Fatigued | 3 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 12, I Feel Fatigued | 8 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 24, I Feel Fatigued | 2 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Day 344, I Feel Fatigued | 6 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 3, Day 113, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 2 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 4, Week 12, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Week 12, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Day 162, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -4 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 6, Day 91, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 7, Day 85, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -7
  Par 8, Day 87, I Feel Fatigued | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10

76. Secondary Outcome: Part B: Change From Baseline in FACIT-Fatigue Scores Over Time for Participants Who Never Received 100mg OL Sirukumab in Part B
Description: The FACIT-Fatigue is a 13-item questionnaire formatted for self-administration that assesses participant reported fatigue and its impact upon daily activities and function over the past seven days. Participants were asked to answer each question using a 5-point Likert-type scale (4 = Not at all; 3 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 0 = Very Much) where 0 is a bad response and 4 is good response. Each of the 13 items of the FACIT-Fatigue Scale ranges from 0-4, with a range of possible total score from 0-52, 0 (Extreme fatigue) to 52 (No fatigue) where 0 being the worst possible score and 52 the best (i.e. less fatigue). Scores below 30 indicate severe fatigue. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Participants with post baseline data were reported.
Time Frame: Baseline (Day 0) and Day 85,87,91,113,162 344,339,Week 12, 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Scores on scale
  Par 1, Day 30, I Feel Fatigued | -3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29, I Feel Fatigued | -1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23, I Feel Fatigued | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, I Feel Fatigued | 2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113, I Feel Fatigued | -16 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8, I Feel Fatigued | -1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85, I Feel Fatigued | -3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65, I Feel Fatigued | -1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 13 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 7 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -11 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Day 169, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 17, Week 12, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6
  Par 17, Day112, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 6
  Par 18, Day 85, I Feel Fatigued | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1

77. Secondary Outcome: Part B: Change From Baseline in Pain NRS Scores Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: The assessment of pain severity was made using a single pain severity item on which participants were asked to rate the severity of their average pain now on an 11-point numeric rating scale ranging from 0, "no pain" to 10, "the worst pain imaginable". Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Day 85,87,91,113,162 344,339,Week 12, 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 2 | 4 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 4 | -1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 8 | -1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12 | 4 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24 | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339 | -2 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 4 | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 8 | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12 | 1 | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24 | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 38 | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 40 | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344 | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 14 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 16 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 2 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -1
  Par 7, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 7, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1
  Par 7, Day 85 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 2
  Par 8, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 87 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0

78. Secondary Outcome: Part B: Change From Baseline in Pain NRS Scores Over Time for Participants Who Never Received at Least One Dose of 100mg OL Sirukumab in Part B
Description: The assessment of pain severity was made using a single pain severity item on which participants were asked to rate the severity of their average pain now on an 11-point numeric rating scale ranging from 0, "no pain" to 10, "the worst pain imaginable". Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Participants with post baseline data were reported.
Time Frame: Baseline (Day 0) and Day 85,87,91,113,162 344,339,Week 12, 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Scores on scale
  Par 1, Day 30 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23 | -1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 4 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 8 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85 | 2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 4 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Day 169 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -3 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 17, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2
  Par 17, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2
  Par 17, Day 112 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2
  Par 18, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1
  Par 18, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0

79. Secondary Outcome: Part B: HAQDI Score Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: as for outcome 15
Time Frame: Day 87, 339, 344, Week 12, 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 1
Scores on scale
  Par 1, Week 12, Able to Do Chores | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Stand Up From a Straight | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Dress yourself | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Open a New Milk Carton | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Open Jars Previously Opened | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Turn Faucets On And Off | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Take a Tub Bath | 3 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Bend Down Pick Up Clothing-Floor | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Reach-Get Down 5 Lb Obj Above Head | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Able to Do Chores | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Stand Up From a Straight | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Dress yourself | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Open a New Milk Carton | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Open Jars Previously Opened | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Turn Faucets On And Off | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Take a Tub Bath | 3 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Bend Down Pick Up Clothing-Floor | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Reach-Get Down 5 Lb Obj Above Head | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Able to Do Chores | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Stand Up From a Straight | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Dress yourself | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Open a New Milk Carton | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Open Jars Previously Opened | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Turn Faucets On And Off | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Take a Tub Bath | 3 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Bend Down Pick Up Clothing-Floor | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Reach-Get Down 5 Lb Obj Above Head | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Able to Do Chores | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Stand Up From a Straight | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Dress yourself | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open a New Milk Carton | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open Jars Previously Opened | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Turn Faucets On And Off | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Take a Tub Bath | 3 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Bend Down Pick Up Clothing-Floor | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Reach-Get Down 5 Lb Obj Above Head | 2 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Able to Do Chores | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Stand Up From a Straight | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Dress yourself | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Open a New Milk Carton | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Open Jars Previously Opened | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Turn Faucets On And Off | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Take a Tub Bath | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Bend Down Pick Up Clothing-Floor | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Reach-Get Down 5 Lb Obj Above Head | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Able to Do Chores | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Get In and Out of a car | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Run Errands and Shop | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Get In and Out of Bed | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Stand Up From a Straight | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Dress yourself | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Shampoo your hair | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Cut your meat | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Lift a Full Cup/Glass to mouth | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Open a New Milk Carton | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Open car doors | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344,Open Jars Previously Opened | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Turn Faucets On And Off | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Get On and Off The Toilet | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Take a Tub Bath | 3 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Wash and Dry Your Body | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Bend Down Pick Up Clothing-Floor | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Reach-Get Down 5 Lb Obj Above Head | 1 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Climb Up Five Steps | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344, Walk Outdoors on Flat Ground | 0 |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Able to Do Chores | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Get In and Out of a car | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Run Errands and Shop | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Get In and Out of Bed | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Stand Up From a Straight | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Dress yourself | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Shampoo your hair | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Cut your meat | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Lift a Full Cup/Glass to mouth | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Open a New Milk Carton | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Open car doors | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Open Jars Previously Opened | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Turn Faucets On And Off | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Get On and Off The Toilet | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Take a Tub Bath | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Wash and Dry Your Body | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Bend Down Pick Up Clothing-Floor | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Reach-Get Down 5 Lb Obj Above Head | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Climb Up Five Steps | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12, Walk Outdoors on Flat Ground | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | 0 |  | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 87, Able to Do Chores | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 1
  Par 4, Day 87, Get In and Out of a car | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Run Errands and Shop | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Get In and Out of Bed | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Stand Up From a Straight | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Dress yourself | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Shampoo your hair | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Cut your meat | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Lift a Full Cup/Glass to mouth | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Open a New Milk Carton | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Open Jars Previously Opened | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Turn Faucets On And Off | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Get On and Off The Toilet | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Take a Tub Bath | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Wash and Dry Your Body | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 1
  Par 4, Day 87, Bend Down Pick Up Clothing-Floor | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Reach-Get Down 5 Lb Obj Above Head | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 1
  Par 4, Day 87, Climb Up Five Steps | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0
  Par 4, Day 87, Walk Outdoors on Flat Ground | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. |  | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikum |  | 0

80. Secondary Outcome: Part B: HAQDI Score Over Time for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: as for outcome 15
Time Frame: Day 29, 64, 65, 85, 112, 113, 169, 373 and Week 12
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 3 | 2 | 1 | 1 | 1
Scores on scale
  Par 1, Day 29, Able to Do Chores | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Get In and Out of a car | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Run Errands and Shop | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Get In and Out of Bed | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Stand Up From a Straight Chair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Dress yourself | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Shampoo your hair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Cut your meat | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Lift a Full Cup or Glass to Mouth | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Open a New Milk Carton | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Open car doors | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Open Jars Previously Opened | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Turn Faucets On And Off | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Get On and Off The Toilet | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Take a Tub Bath | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Wash and Dry Your Body | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Bend Down Pick Up Clothing- Floor | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Reach-Get Down 5 Lb Obj Above Head | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Climb Up Five Steps | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 29, Walk Outdoors on Flat Ground | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Able to Do Chores | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get In and Out of a car | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Run Errands and Shop | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get In and Out of Bed | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Stand Up From a Straight Chair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Dress yourself | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Shampoo your hair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Cut your meat | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Lift a Full Cup or Glass to Mouth | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open a New Milk Carton | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open r car doors | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Open Jars Previously Opened | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Turn Faucets On And Off | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Get On and Off The Toilet | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Take a Tub Bath | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Wash and Dry Your Body | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Bend Down Pick Up Clothing- Floor | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Reach-Get Down 5 Lb Obj Above Head | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Climb Up Five Steps | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12, Walk Outdoors on Flat Ground | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Able to Do Chores | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Get In and Out of a car | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Run Errands and Shop | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Get In and Out of Bed | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Stand Up From a Straight Chair | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Dress yourself | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Shampoo your hair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Cut your meat | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Lift a Full Cup or Glass to Mouth | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Open a New Milk Carton | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Open car doors | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Open Jars Previously Opened | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Turn Faucets On And Off | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Get On and Off The Toilet | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Take a Tub Bath | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Wash and Dry Your Body | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Bend Down Pick Up Clothing- Floor | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Reach-Get Down 5 Lb Obj Above Head | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Climb Up Five Steps | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 113, Walk Outdoors on Flat Ground | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Able to Do Chores | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Get In and Out of a car | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Run Errands and Shop | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Get In and Out of Bed | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Stand Up From a Straight Chair | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Dress yourself | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Shampoo your hair | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Cut your meat | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Lift a Full Cup or Glass to Mouth | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Open a New Milk Carton | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Open car doors | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Open Jars Previously Opened | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Turn Faucets On And Off | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Get On and Off The Toilet | 0 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Take a Tub Bath | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Wash and Dry Your Body | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Bend Down Pick Up Clothing- Floor | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Reach-Get Down 5 Lb Obj Above Head | 1 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Climb Up Five Steps | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 65, Walk Outdoors on Flat Ground | 0 | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 373, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 64, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85 Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85,Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 85, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169,Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 169, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0 | NA — Only 1 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Week 12, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12,Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Lift a Full Cup or Glass to Mouth | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12,Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12 Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Week 12, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Able to Do Chores | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Get In and Out of a car | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Run Errands and Shop | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Get In and Out of Bed | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Stand Up From a Straight Chair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Dress yourself | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Shampoo your hair | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Cut your meat | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Lift a Full Cup or Glass to Mout | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Open a New Milk Carton | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Open car doors | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Open Jars Previously Opened | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Turn Faucets On And Off | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Get On and Off The Toilet | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Take a Tub Bath | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Wash and Dry Your Body | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Bend Down Pick Up Clothing- Floor | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Reach-Get Down 5 Lb Obj Above Head | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Climb Up Five Steps | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0
  Par 8, Day 112, Walk Outdoors on Flat Ground | NA — Only 3 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0

81. Secondary Outcome: Part B: Change From Baseline in PtGA Score for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: The Patient's Global Assessments of Disease Activity was recorded on a Visual analog scale (VAS). of 10 centimeter (cm) ranging from 0 ("very well) to 10 ("very poor"). Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38, 40; Days 85, 87, 91, , 113, 162, 339, and 344
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 2 | 4.3 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 4 | 2.3 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 8 | -0.2 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12 | 4.0 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 16 | 4.7 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24 | 2.2 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 36 | 0.4 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339 | -0.7 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 4 | -1.0 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 8 | -0.3 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12 | -0.6 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 16 | -0.7 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24 | 0.5 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 36 | -0.6 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 38 | 0.9 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 40 | -0.3 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344 | -0.7 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3,Par 3,, Day 113 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 2.1 | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 4.9 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.4 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 2.0 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.4
  Par 5, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.2 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 14 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1.0 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 16 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1.0 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 162 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.8 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -3.1 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -3.2 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 91 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -3.5 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.7
  Par 7, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.7
  Par 7, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.8
  Par 7, Day 85 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.4
  Par 8, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.1
  Par 8, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -3.7
  Par 8, Day 87 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -3.1
  Par 6, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.1 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.

82. Secondary Outcome: Part B: Change From Baseline in PtGA Score for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: The Patient's Global Assessments of Disease Activity was recorded on a Visual analog scale (VAS). of 10 centimeter (cm) ranging from 0 ("very well) to 10 ("very poor"). Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Participants with post baseline data were reported.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12, 16, 36; Days 23, 29, 30, 57, 59, 64, 65, 85,112, 113, 115, 163, 169 and 373
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 2 | 2
Scores on scale
  Par 1, Day 30 | 0.2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29 | -0.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 4 | -0.2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 8 | 0.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | 0.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8 | 0.4 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85 | 2.3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 4 | -1.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65 | 0.5 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 16 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 36 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.9 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.4 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.3 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 16 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.3 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.8 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.7 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.9 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.7 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.0 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.4 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.9 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.3
  Par 16, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.3
  Par 16, Day 112 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.1
  Par 17, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 0.2
  Par 17, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.1

83. Secondary Outcome: Part B: Change From Baseline in PhGA Score for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: In PhGA was based on "What is physician's assessment of the participant's current disease activity". PhGA used a 10 cm VAS ranging from 0 ("none") to 10 ("extremely active"). Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Day 85, Day 113, Day 162, Day 203, Day 339, Day 344, Week 2, Week 4, Week 8, Week 12, Week 14, Week 16, Week 24, Week 36, Week 38, Week 40
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 2 | 0.0 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 4 | -0.5 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 8 | -1.2 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 12 | -0.6 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 16 | -0.9 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 24 | -0.6 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Week 36 | -1.1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 1, Day 339 | -1.2 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 4 | 0.0 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 8 | 0.1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 12 | 0.4 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 16 | 0.1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 24 | 0.0 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 36 | 0.1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 38 | 0.7 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Week 40 | 0.4 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 344 | 0.2 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 113 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.2 | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.2 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.8 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1.1 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.7 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 14 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1.5 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 16 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -1.1 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Day 162 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -0.4 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 6, Day 203 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 7.6 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 7, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0
  Par 7, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1
  Par 7, Week 8 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0
  Par 7, Day 85 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0
  Par 8, Week 2 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.0
  Par 8, Week 4 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -6.3

84. Secondary Outcome: Part B: Change From Baseline in PhGA Score for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: In PhGA was based on "What is physician's assessment of the participant's current disease activity". PhGA used a 10 cm VAS ranging from 0 ("none") to 10 ("extremely active"). Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value. Participants with post baseline data were reported.
Time Frame: Baseline (Day 0), Weeks 4, 8, 12, 16, 36; Days 23, 29, 30, 57, 59, 64, 65, 85, 112, 113, 163, 169 and 373
Population: ITT-Part B Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 2 | 2
Scores on scale
  Par 1, Day 30 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29 | 0.1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Week 12 | 0.7 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113 | 0.0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Week 4 | -0.3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85 | 0.3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Week 4 | -0.2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65 | -0.3 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 16 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.4 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 36 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.4 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.9 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 16 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.9 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.4 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.6 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.3 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.3 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.3 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 169 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.5 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Week 4 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -0.1
  Par 16, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.0
  Par 16, Day 112 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.4
  Par 17, Week 8 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.1
  Par 17, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 0.2

85. Secondary Outcome: Part B: Number of Participants With PGIC Score Over Time Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: as for outcome 16
Time Frame: Baseline (Day 1), Days 103 and 271
Population: ITT-Part B Population
Measure: Number; unit: Participants
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Participants
  Par 1, Day 1: Much Better | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Day 1: Much Better | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Day 271: Worse | 1 | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 3, Day 1: Much Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1 | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 4, Day 1: Much Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5,Day 1: Slightly Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Day 103: No change | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 6, Day 1: Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 7, Day 1: Much Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1
  Par 8, Day 1: Slightly Better | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 1 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1

86. Secondary Outcome: Part B: Number of Participants With PGIC Score Over Time Who Never Received 100 mg OL Sirukumab in Part B
Description: as for outcome 16
Time Frame: Baseline (Day 1)
Population: ITT-Part B Population
Measure: Number; unit: Participants
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Participants
  Par 1, Day 1: No change | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 1: Much Better | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 1: Much Better | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 1: Much Better | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 1: Better | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 1: Much Better | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 1: Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 1: Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 1: Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 1: Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 15, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 2 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 17, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1
  Par 18, Day 1: Much Better | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 3 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 1

87. Secondary Outcome: Part B: Change From Baseline in CRP Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: Blood samples were collected for analysis of CRP. Data for Change from Baseline in serum CRP over time for part B was reported. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: ITT-Part B Population
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Milligram per liter (mg/L)
  Week 2, n=1,1,0,1,2: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2
  Week 2, n=1,1,0,1,2 | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -0.20 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |  | -3.70 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -4.20 (2.970)
  Week 4, n=2,1,1,2,2 | 0.10 (0.000) | 0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -2.35 (1.909) | -4.20 (2.828)
  Week 8, n=2,1,1,2,1: number analyzed (Participants) | 2 | 1 | 1 | 2 | 1
  Week 8, n=2,1,1,2,1 | 0.10 (0.000) | -0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.30 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.55 (6.010) | -2.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant
  Week 12, n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12, n=2,1,1,1,0 | 0.10 (0.000) | -0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 3.90 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |
  Week 14, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14, n=0,0,0,1,0 |  |  |  | -30.20 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |
  Week 16, n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16, n=2,0,0,1,0 | 0.40 (0.424) |  |  | -30.70 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |
  Week 24, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24, n=2,0,0,0,0 | 1.90 (2.546) |  |  |  |
  Week 36, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36, n=2,0,0,0,0 | 0.80 (0.849) |  |  |  |
  Week 38, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38, n=1,0,0,0,0 | -0.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |  |  |  |
  Week 40, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40, n=1,0,0,0,0 | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |  |  |  |

88. Secondary Outcome: Part B: Change From Baseline in CRP Over Time for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: as for outcome 87
Time Frame: Baseline (Day 0), Weeks 4, 8, 12, 16, 24 and 36
Population: ITT-Part B Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
mg/L
  Week 4, n=3,3,2,1,2: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2
  Week 4, n=3,3,2,1,2 | -0.30 (0.361) | -0.23 (0.252) | 0.05 (0.071) | 6.10 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -0.55 (1.202)
  Week 8, n=2,1,2,0,2: number analyzed (Participants) | 2 | 1 | 2 | 0 | 2
  Week 8, n=2,1,2,0,2 | -0.05 (0.778) | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.00 (0.000) |  | 0.95 (0.636)
  Week 12, n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12, n=1,1,1,1,1 | -0.90 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -0.80 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.70 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant
  Week 16, n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16, n=0,1,1,1,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant | -0.70 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |
  Week 24, n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24, n=0,1,0,0,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |  |  |
  Week 36, n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36, n=0,1,0,0,0 |  | 0.00 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant |  |  |

89. Secondary Outcome: Part B: Change From Baseline in ESR Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: Blood samples were collected for analysis of ESR. Data for Change from Baseline in ESR over time for part A was reported. Baseline was the last measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12, 14, 16, 24, 36, 38 and 40
Population: Safety-Part B Population
Measure: Mean (Standard Deviation); unit: Millimeter per hour (mm/h)
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Millimeter per hour (mm/h)
  Week 2, n=1,1,0,1,1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Week 2, n=1,1,0,1,1 | -1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 4.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. |  | -14.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -7.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.
  Week 4, n=2,1,1,2,2 | 0.5 (2.12) | 4.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 4.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -5.0 (16.97) | -29.5 (31.82)
  Week 8, n=2,1,0,2,1: number analyzed (Participants) | 2 | 1 | 0 | 2 | 1
  Week 8, n=2,1,0,2,1 | 3.0 (7.07) | 2.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. |  | -6.0 (15.56) | -7.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.
  Week 12, n=2,1,1,1,0: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0
  Week 12, n=2,1,1,1,0 | 0.0 (1.41) | 2.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 4.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 10.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.. |
  Week 14, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Week 14, n=0,0,0,1,0 |  |  |  | -19.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.. |
  Week 16, n=2,0,0,1,0: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0
  Week 16, n=2,0,0,1,0 | -0.5 (2.12) |  |  | -18.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.. |
  Week 24, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 24, n=2,0,0,0,0 | -1.5 (0.71) |  |  |  |
  Week 36, n=2,0,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Week 36, n=2,0,0,0,0 | 6.0 (11.31) |  |  |  |
  Week 38, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 38, n=1,0,0,0,0 | -1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.. |  |  |  |
  Week 40, n=1,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Week 40, n=1,0,0,0,0 | 1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.. |  |  |  |

90. Secondary Outcome: Part B: Change From Baseline in ESR Over Time for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: as for outcome 89
Time Frame: Baseline (Day 0), Weeks 4, 8, 12, 16, 24 and 36
Population: Safety-Part B Population
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
mm/h
  Week 4, n=3,3,3,1,2: number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  Week 4, n=3,3,3,1,2 | -1.7 (5.03) | 1.3 (1.53) | -1.0 (1.00) | 8.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -2.0 (5.66)
  Week 8, n=2,1,3,0,2: number analyzed (Participants) | 2 | 1 | 3 | 0 | 2
  Week 8, n=2,1,3,0,2 | -1.0 (7.07) | 2.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -2.0 (0.00) |  | 0.0 (2.83)
  Week 12, n=1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 12, n=1,1,1,1,1 | -6.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 0.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -6.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 12.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant.
  Week 16, n=0,1,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Week 16, n=0,1,1,1,0 |  | 3.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | 1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. | -4.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. |
  Week 24, n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 24, n=0,1,0,0,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. |  |  |
  Week 36, n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Week 36, n=0,1,0,0,0 |  | 1.0 (NA) — NA indicates data is not available since standard deviation could not be calculated for single participant. |  |  |

91. Secondary Outcome: Part B: Change From Baseline in EQ-5D-5L VAS Over Time for Participants Who Received at Least One Dose of 100 mg OL Sirukumab in Part B
Description: EQ-5D essentially consists of 2 elements: the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system comprised of the following 6 dimensions: 1.Mobility, 2.Self, 3.Usual Activities, 4.Pain/Discomfort, 5.Anxiety/Depression; 6.How good or or bad your health is today. Each of these 6 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The EQ VAS records the respondent's self-rated health on a vertical line, VAS where the endpoints are 'Best imaginable health state' and 'Worst imaginable health state'. Answers to 'How good or bad your health is today' were measured on a 100 point VAS scale. Baseline for Part B is the last non-missing measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Days 85, 87, 91, 113, 162, 339 and 344 and Weeks 12 and 24
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 2
Scores on scale
  Par 1, Week 12 | -12 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Week 24 | 1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 1, Day 339 | 8 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 12 | 3 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Week 24 | 14 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 2, Day 344 | -1 | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 3, Day 113 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 1 | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 4, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.v | -4 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Week 12 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 9 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 5, Day 162 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | -15 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 6, Day 91 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | 20 | NA — Only 2 participant in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab
  Par 7, Day 85 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 4
  Par 8, Day 87 | NA — Only 2 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participant in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 21

92. Secondary Outcome: Part B: Change From Baseline in EQ-5D-5L VAS Over Time for Participants Who Never Received 100 mg OL Sirukumab in Part B
Description: EQ-5D essentially consists of 2 elements: the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system comprised of the following 6 dimensions: 1.Mobility, 2.Self, 3.Usual Activities, 4.Pain/Discomfort, 5.Anxiety/Depression; 6.How good or or bad your health is today. Each of these 6 dimensions has 5 levels: 1: no problems; 2: slight problems; 3: moderate problems; 4: severe problems; 5: Unable to do. The EQ VAS records the respondent's self-rated health on a vertical line, VAS where the endpoints are 100 (Best imaginable health state) and 0 (Worst imaginable health state). Answers to 'How good or bad your health is today' were measured on a 100 point VAS scale. Baseline for Part B is the last non-missing measurement done up to and including the Week 52 visit date of Part A. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline (Day 0) and Days 23, 29, 30, 57, 59, 64, 65, 85, 112, 113, 163, 169, 344 and 373 and Week 12
Population: ITT-Part B Population
Measure: Number; unit: Scores on scale
Arm/Group | PartB:SIR 100 mg SC q2w+6 Month Prednisone | PartB:SIR 100 mg SC q2w+3 Month Prednisone | PartB:SIR 50 mg SC q4w+6 Month Prednisone | PartB:Placebo SC q2w + 6 Month Prednisone | PartB:Placebo SC q2w + 12 Month Prednisone
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 2
Scores on scale
  Par 1, Day 30 | 2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 2, Day 29 | 0 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 3, Day 23 | 1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Week 12 | -2 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 4, Day 113 | -47 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 5, Day 85 | -1 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 6, Day 65 | 20 | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 4 | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 7, Day 373 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 8 | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 8, Day 64 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -2 | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 9, Day 29 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -1 | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 10, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 5 | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -10 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 11, Day 163 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -12 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 12, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -8 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 13, Day 59 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 10 | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 14, Day 57 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -42 | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 16, Day 169 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 62 | NA — Only 1 participants in Arm5 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab.
  Par 17, Week 12 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 9
  Par 17, Day 112 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | 7
  Par 18, Day 85 | NA — Only 6 participants in Arm1 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 4 participants in Arm2 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm3 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | NA — Only 2 participants in Arm4 completed Part A of the study, entered Part B and received at least one dose of 100mg OL Sirikumab. | -4

ADVERSE EVENTS:
Time Frame: On-treatment serious Adverse events (SAEs) and non-serious Adverse Events (nSAEs) were collected from the start of study treatment up to Week 52 in Part A and up to Week 120 in Part B.
Description: Safety Set was used. Safety Population comprised of all randomized participants who received at least 1 dose of SC Investigational Product.
Groups:
- Part A: SIR 50 mg SC q4w+6 Month Prednisone: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen
- Part A:Placebo SC q2w + 12 Month Prednisone: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen
- Part B:SIR 100 mg SC q2w+6 Month Prednisone+100mg OL SIR: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen in Part A. Participants received at least one dose of 100mg OL SIR in Part B.
- Part B:SIR 100 mg SC q2w+3 Month Prednisone+100mg OL SIR: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen in Part A. Participants received at least one dose of 100mg OL SIR in Part B.
- Part B:SIR 50 mg SC q4w+6 Month Prednisone+100mg OL SIR: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A. Participants received at least one dose of 100mg OL SIR in Part B.
- Part B:Placebo SC q2w + 6 Month Prednisone+100mg OL SIR: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen in Part A. Participants received at least one dose of 100mg OL SIR in Part B.
- Part B:Placebo SC q2w + 12 Month Prednisone+100mg OL SIR: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen in Part A. Participants received at least one dose of 100mg OL SIR in Part B.
- Part B:SIR 100 mg SC q2w+6 Month Prednisone/ No 100mg OL SIR: Participants received SIR 100 milligram (mg) subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a pre-specified maximum of 6-months prednisone taper regimen in Part A. Participants never received 100mg OL SIR in Part B.
- Part B:SIR 100 mg SC q2w+3 Month Prednisone/ No 100mg OL SIR: Participants received SIR 100 mg SC q2w for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen. Participants never received 100mg OL SIR in Part B.
- Part B:SIR 50 mg SC q4w+6 Month Prednisone/ No 100mg OL SIR: Participants received SIR 50 mg SC every 4 weeks (q4w) for 52 weeks plus a pre-specified maximum of 3-month prednisone taper regimen. Participants never received 100mg OL SIR in Part B.
- Part B:Placebo SC q2w + 6 Month Prednisone/ No 100mg OL SIR: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 6-month prednisone taper regimen. Participants never received 100mg OL SIR in Part B.
- Part B:Placebo SC q2w + 12 Month Prednisone/ No 100mg OL SIR: Participants received placebo SC q2w for 52 weeks plus a pre-specified maximum of 12-month prednisone taper regimen. Participants never received 100mg OL SIR in Part B.
Arm/Group | Part A:SIR 100 mg SC q2w+6 Month Prednisone | Part A:SIR 100 mg SC q2w+3 Month Prednisone | Part A: SIR 50 mg SC q4w+6 Month Prednisone | Part A:Placebo SC q2w + 6 Month Prednisone | Part A:Placebo SC q2w + 12 Month Prednisone | Part B:SIR 100 mg SC q2w+6 Month Prednisone+100mg OL SIR | Part B:SIR 100 mg SC q2w+3 Month Prednisone+100mg OL SIR | Part B:SIR 50 mg SC q4w+6 Month Prednisone+100mg OL SIR | Part B:Placebo SC q2w + 6 Month Prednisone+100mg OL SIR | Part B:Placebo SC q2w + 12 Month Prednisone+100mg OL SIR | Part B:SIR 100 mg SC q2w+6 Month Prednisone/ No 100mg OL SIR | Part B:SIR 100 mg SC q2w+3 Month Prednisone/ No 100mg OL SIR | Part B:SIR 50 mg SC q4w+6 Month Prednisone/ No 100mg OL SIR | Part B:Placebo SC q2w + 6 Month Prednisone/ No 100mg OL SIR | Part B:Placebo SC q2w + 12 Month Prednisone/ No 100mg OL SIR
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39 | 0/26 | 0/27 | 0/27 | 0/2 | 0/1 | 0/1 | 0/2 | 0/2 | 0/6 | 0/4 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 8/42 | 6/39 | 6/26 | 5/27 | 6/27 | 0/2 | 0/1 | 0/1 | 0/2 | 0/2 | 0/6 | 0/4 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 41/42 | 36/39 | 25/26 | 26/27 | 24/27 | 2/2 | 1/1 | 1/1 | 2/2 | 2/2 | 4/6 | 3/4 | 2/3 | 1/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A:SIR 100 mg SC q2w+6 Month Prednisone (N=42) | Part A:SIR 100 mg SC q2w+3 Month Prednisone (N=39) | Part A: SIR 50 mg SC q4w+6 Month Prednisone (N=26) | Part A:Placebo SC q2w + 6 Month Prednisone (N=27) | Part A:Placebo SC q2w + 12 Month Prednisone (N=27) | Part B:SIR 100 mg SC q2w+6 Month Prednisone+100mg OL SIR (N=2) | Part B:SIR 100 mg SC q2w+3 Month Prednisone+100mg OL SIR (N=1) | Part B:SIR 50 mg SC q4w+6 Month Prednisone+100mg OL SIR (N=1) | Part B:Placebo SC q2w + 6 Month Prednisone+100mg OL SIR (N=2) | Part B:Placebo SC q2w + 12 Month Prednisone+100mg OL SIR (N=2) | Part B:SIR 100 mg SC q2w+6 Month Prednisone/ No 100mg OL SIR (N=6) | Part B:SIR 100 mg SC q2w+3 Month Prednisone/ No 100mg OL SIR (N=4) | Part B:SIR 50 mg SC q4w+6 Month Prednisone/ No 100mg OL SIR (N=3) | Part B:Placebo SC q2w + 6 Month Prednisone/ No 100mg OL SIR (N=3) | Part B:Placebo SC q2w + 12 Month Prednisone/ No 100mg OL SIR (N=2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/36 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A:SIR 100 mg SC q2w+6 Month Prednisone (N=42) | Part A:SIR 100 mg SC q2w+3 Month Prednisone (N=39) | Part A: SIR 50 mg SC q4w+6 Month Prednisone (N=26) | Part A:Placebo SC q2w + 6 Month Prednisone (N=27) | Part A:Placebo SC q2w + 12 Month Prednisone (N=27) | Part B:SIR 100 mg SC q2w+6 Month Prednisone+100mg OL SIR (N=2) | Part B:SIR 100 mg SC q2w+3 Month Prednisone+100mg OL SIR (N=1) | Part B:SIR 50 mg SC q4w+6 Month Prednisone+100mg OL SIR (N=1) | Part B:Placebo SC q2w + 6 Month Prednisone+100mg OL SIR (N=2) | Part B:Placebo SC q2w + 12 Month Prednisone+100mg OL SIR (N=2) | Part B:SIR 100 mg SC q2w+6 Month Prednisone/ No 100mg OL SIR (N=6) | Part B:SIR 100 mg SC q2w+3 Month Prednisone/ No 100mg OL SIR (N=4) | Part B:SIR 50 mg SC q4w+6 Month Prednisone/ No 100mg OL SIR (N=3) | Part B:Placebo SC q2w + 6 Month Prednisone/ No 100mg OL SIR (N=3) | Part B:Placebo SC q2w + 12 Month Prednisone/ No 100mg OL SIR (N=2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (36) | 5 (6) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (9) | 3 (5) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (6) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (7) | 1 (2) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (6) | 3 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 8 (8) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2) | 2 (2) | 2 (2) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (5) | 2 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (20) | 7 (14) | 8 (16) | 7 (7) | 8 (13) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (41) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 9 (29) | 4 (4) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 3 (3) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 3 (19) | 4 (7) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 6 (9) | 2 (6) | 4 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 4 (6) | 4 (4) | 2 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 8 (14) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 5 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (3) | 2 (2) | 2 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (8) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1/2 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (8) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 2 (3) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT02531633/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02531633/SAP_001.pdf